CLINICAL TRIAL: NCT00975130
Title: An Open-Label Study Assessing the Addition of Subcutaneous Golimumab (GLM) to Conventional Disease-Modifying Antirheumatic Drug (DMARD) Therapy in Biologic-Naïve Subjects With Rheumatoid Arthritis (Part 1), Followed by a Randomized Study Assessing the Value of Combined Intravenous and Subcutaneous GLM Administration Aimed at Inducing and Maintaining Remission (Part 2)
Brief Title: Subcutaneous Golimumab (GLM) Plus DMARDs for Rheumatoid Arthritis, Followed by Intravenous/Subcutaneous GLM Strategy (P06129 AM2)
Acronym: GO-MORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P06129; 2009-011137-26 (EudraCT Number); CTRI/2009/091/000883 (Registry Identifier: CTRI)
Record Dates: First submitted 2009-08-20; First posted 2009-09-11 (Estimated); Results first posted 2012-12-07 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Injections, Subcutaneous; golimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SC-GLM50 (Experimental): In Part 1 of the study, participants received subcutaneous golimumab treatment at a dose of 50 mg once monthly for 6 months in combination with background DMARD treatment.
  Interventions: Biological: SC golimumab
- IV GLM 2 mg/kg + GLM50-SC (Experimental): After 6 months of treatment in study Part 1, participants with good or moderate response but not in remission will receive intravenous (IV) golimumab at a dose of 2 mg/kg once monthly for a period of 6 months or until remission is achieved. Participants will receive IV GLM at a dose of 2 mg/kg at the start of Month 7, and then at the start of Month 8 and Month 10 if the subject has not achieved remission at any of these IV administration visits. If remission is achieved, participants were switched to subcutaneous golimumab at a dose of 50 mg once monthly until study end, in combination with background DMARD treatment.
  Interventions: Biological: SC golimumab; Biological: IV golimumab
- GLM50-SC (Experimental): After 6 months of treatment in study Part 1, participants with good or moderate response but not in remission will receive subcutaneous golimumab at a dose of 50 mg once monthly for a period of 6 months, in combination with background DMARD treatment.
  Interventions: Biological: SC golimumab

INTERVENTIONS:
Biological: SC golimumab — Subcutaneous golimumab at a dose of 50 mg administered once monthly.
  Other Names: SCH 900259, subcutaneous
Biological: IV golimumab — Intravenous golimumab administered up to 3 times (month 7, 8, 10) during a period of 6 months at a dose of 2 mg/kg of body weight.
  Other Names: SCH 900259, intravenous
  Arms: IV GLM 2 mg/kg + GLM50-SC

SUMMARY:
Part 1 of this trial will assess the safety and effectiveness of subcutaneous (SC) golimumab administered by autoinjector once monthly, when combined with different disease-modifying antirheumatic drug (DMARD) regimens used in daily rheumatology practice. Subsequently, Part 2 will study if a strategy of intravenous (IV) golimumab to induce remission followed by SC golimumab to retain remission is superior to continuing a SC regimen.

DETAILED DESCRIPTION:
Participants who had a good or moderate European League Against Rheumatism (EULAR) response but not achieve remission at the end of Part 1 were invited to participate in Part 2 and were randomized to either intravenous golimumab (IV GLM) + subcutaneous golimumab (SC GLM) or SC GLM alone.

ELIGIBILITY:
Inclusion Criteria:

For Part 1:

* Age >=18 years, either sex, any race.
* Diagnosis of RA according to the 1987 revised American College of Rheumatology (ACR) criteria.
* Active disease despite DMARD treatment
* Subject must be taking at least one of the allowed DMARDs, and must be able to continue with it during the trial.
* Eligibility for anti tumor necrosis factor (TNF) use according to the following criteria:

  * Participant must have failed conventional treatment according to the investigator's opinion OR local guidelines.
  * Local guidelines regarding safety screening of anti TNF candidates (ie, tuberculosis [TB] screening and other safety screening such as vaccination, if applicable) must be met. Chest X-ray and either a PPD skin test or QuantiFERON®-TB Gold test are also required.
  * Anamnesis and physical examination must make the participant eligible for anti TNF use and trial participation according to the investigator's judgment.

For Part 2:

* Participant must have completed Part 1 of this trial.
* Participant must have:

  * good or moderate response to SC golimumab at the end of Month 6 compared to Baseline, AND.
  * no DAS28 ESR remission.
* Both the investigator and the subject must agree to switch the participant's treatment to IV administration as may be required in Part 2 of this trial.
* The investigator must judge that no safety events (eg, serious adverse events [SAEs], serious infections, marked injection-site reactions or intolerance to drug) have occurred that could reoccur or aggravate with increased drug exposure.

Exclusion Criteria:

* History of biologic drug use for RA.
* Evidence of active TB. or latent TB that is untreated.
* Moderate to severe heart failure
* Certain inflammatory rheumatic disease other than RA or certain systemic inflammatory condition
* Allergy to latex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3366 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2012-02 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Combe B, Dasgupta B, Louw I, Pal S, Wollenhaupt J, Zerbini CA, Beaulieu AD, Schulze-Koops H, Durez P, Yao R, Vastesaeger N, Weng HH; GO-MORE Investigators. Efficacy and safety of golimumab as add-on therapy to disease-modifying antirheumatic drugs: results of the GO-MORE study. Ann Rheum Dis. 2014 Aug;73(8):1477-86. doi: 10.1136/annrheumdis-2013-203229. Epub 2013 Jun 5. PMID 23740226
- [Derived] Durez P, Vanthuyne M, Soyfoo MS, Hoffman I, Malaise M, Geusens P. Efficacy of golimumab in Belgian patients with active rheumatoid arthritis despite treatment with non-biologic disease-modifying anti-rheumatic drugs: sub-analysis of the GO-MORE study. Acta Clin Belg. 2017 Dec;72(6):424-428. doi: 10.1080/17843286.2017.1314079. Epub 2017 Apr 21. PMID 28431485
- [Derived] Schulze-Koops H, Giacomelli R, Samborski W, Rednic S, Herold M, Yao R, Govoni M, Vastesaeger N, Weng HH. Factors influencing the patient evaluation of injection experience with the SmartJect autoinjector in rheumatoid arthritis. Clin Exp Rheumatol. 2015 Mar-Apr;33(2):201-8. Epub 2015 Jan 29. PMID 25664404
- [Derived] Dasgupta B, Combe B, Louw I, Wollenhaupt J, Zerbini CA, Beaulieu A, Schulze-Koops H, Durez P, Wolff V, Yao R, Weng HH, Govoni M, Vastesaeger N. Patient and physician expectations of add-on treatment with golimumab for rheumatoid arthritis: relationships between expectations and clinical and quality of life outcomes. Arthritis Care Res (Hoboken). 2014 Dec;66(12):1799-807. doi: 10.1002/acr.22371. PMID 24839031

RESULTS

PARTICIPANT FLOW:
Groups:
- Golimumab 50 mg Subcutaneous (GLM50-SC): Participants received GLM50-SC once monthly for a period of 6 months in Study Part 1.
- Intravenous GLM (IV-GLM) 2 mg/kg + SC GLM 50 mg: Participants achieving good or moderate response but not in remission at the conclusion of Study Part 1 received IV-GLM at a dose of 2 mg/kg at the start of Month 7, start of Month 8, and start of Month 10 if remission was not achieved at any of these IV administration visits. If remission was achieved, participants were switched subcutaneous golimumab at a dose of 50 mg once monthly.
- SC-GLM50: Participants achieving good or moderate response but not in remission at the end of Study Part 1, received subcutaneous golimumab at a dose of 50 mg once monthly for a period of 6 months in Part 2 of the study.
Period: Study Part 1
Arm/Group | Golimumab 50 mg Subcutaneous (GLM50-SC) | Intravenous GLM (IV-GLM) 2 mg/kg + SC GLM 50 mg | SC-GLM50
Started | 3366 | 0 | 0
Completed | 3086 | 0 | 0
Not Completed | 280 | 0 | 0
Not completed — Adverse Event | 150 | 0 | 0
Not completed — Lost to Follow-up | 19 | 0 | 0
Not completed — Withdrawal by Subject | 61 | 0 | 0
Not completed — Protocol Violation | 13 | 0 | 0
Not completed — Did Not Meet Protocol Eligibility | 9 | 0 | 0
Not completed — Administrative | 4 | 0 | 0
Not completed — Withdrew Consent | 24 | 0 | 0
Period: Study Part 2
Arm/Group | Golimumab 50 mg Subcutaneous (GLM50-SC) | Intravenous GLM (IV-GLM) 2 mg/kg + SC GLM 50 mg | SC-GLM50
Started | 0 | 250 (Good/moderate responders without remission at the end of Part 1 were invited to enroll in Part 2.) | 255 (Good/moderate responders without remission at the end of Part 1 were invited to enroll in Part 2.)
Completed | 0 | 212 | 238
Not Completed | 0 | 38 | 17
Not completed — Adverse Event | 0 | 14 | 7
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 13 | 5
Not completed — Withdrew Consent | 0 | 6 | 2
Not completed — Did Not Meet Protocol Eligibility | 0 | 4 | 1
Not completed — Administrative | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- GLM50-SC: Participants received 50 mg of golimumab subcutaneously once monthly for a period of 6 months. 3280 enrolled participants were included in the Efficacy-Evaluable population; baseline characteristics are presented for this population.
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Age, Continuous [Median (Full Range); unit: Years] | 53 [18 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2716
  Male | 564

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving a Good or Moderate European League Against Rheumatism (EULAR) Response at Month 6
Description: EULAR response was assessed at the end of Month 6 by the Disease Activity Score using the 28 tender and swollen joint count calculated with erythrocyte sedimentation rate values (DAS28-ESR). A good response was defined as a decrease >1.2 units and a final DAS28-ESR < 3.2 units, while a moderate response was defined as a decrease > 1.2 units and final DAS28-ESR >= 3.2 units, OR a decrease of 0.6 to 1.2 units AND final DAS28-ESR <= 5.1 units
Time Frame: Month 6
Population: The Efficacy Evaluable population in Part 1 of the study excluded participants without a DAS28-ESR at baseline and at least 1 post-line value DAS28-ESR or those that had very poor data quality due to incomplete documentation.
Measure: Number; unit: Participants
Groups:
- GLM50-SC: Participants received subcutaneous golimumab 50 mg once monthly.
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Participants | 2692

2. Primary Outcome: Number of Participants Experiencing Disease Activity Score 28-Erythrocyte Sedimentation Rate (DAS28-ESR) Remission at the Start of Month 11 and End of Month 12
Description: The number of participants experiencing DAS28-ESR remission was evaluated at the start of study Month 11 and the end of study Month 12. The DAS28-ESR is expressed on a unit on a scale with the minimum score=0 (best) to maximum score=10 (worst). Remission was defined as DAS28-ESR <2.6.
Time Frame: Start of Month 11, End of Month 12
Population: The efficacy evaluable population comprised all participants with a baseline DAS28-ESR and at least one post-baseline measurement of DAS28-ESR.
Measure: Number; unit: Participants
Groups:
- IV-GLM2/SC-GLM50: Intravenous golimumab 2 mg/kg followed by subcutaneous golimumab 50 mg once monthly.
- SC-GLM50: Subcutaneous golimumab 50 mg administered once monthly for for 6 months (study Months 6-12).
Arm/Group | IV-GLM2/SC-GLM50 | SC-GLM50
Number analyzed (Participants) | 242 | 248
Participants
  Start of Month 11 | 58 | 64
  End of Month 12 | 59 | 67

3. Secondary Outcome: Mean Change From Baseline in the Number of Swollen Joints by Concomitant Methotrexate (MTX) Dose at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the mean number of swollen joints was calculated at study Month 2, Month 4, and Month 6 by concomitant MTX dose (low < 10mg/wk, medium >= 10 to < 15 mg/week, and high >=15 mg/week). A total of 28 joints were evaluated.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: The efficacy evaluable population comprised all participants with a baseline DAS28-ESR and at least one post-baseline measurement of DAS28-ESR. n values represent the number of participants at baseline.
Measure: Mean (Standard Deviation); unit: Swollen Joints
Groups:
- GLM50-SC: Participants received subcutaneous golimumab 50 mg once monthly for 6 months (study Month 1 to Month 6).
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Swollen Joints
  Low MTX Dose - Month 2 (n =142) | -4.7 (4.46)
  Low MTX Dose - Month 4 (n=142) | -6.3 (5.37)
  Low MTX Dose - Month 6 (n=142) | -7.7 (5.59)
  Medium MTX Dose - Month 2 (n=526) | -4.6 (4.45)
  Medium MTX Dose - Month 4 (n=526) | -6.2 (4.98)
  Medium MTX Dose - Month 6 (n=526) | -7.1 (5.37)
  High MTX Dose - Month 2 (n=1995) | -4.5 (4.67)
  High MTX Dose - Month 4 (n=1995) | -6.2 (5.07)
  High MTX Dose - Month 6 (n=1995) | -6.9 (5.30)

4. Secondary Outcome: Mean Change From Baseline in the Number of Swollen Joints by Disease Modifying Antirheumatic Drug (DMARD) Background Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of swollen joints was calculated by participant baseline background DMARD treatment regimen at study Month 2, Month 4, and Month 6. A total of 28 joints were evaluated. DMARD Combination 1 = MTX + hydrochloroquine, chloroquine, chloroquine phosphate; Combination 2 = MTX + leflunomide; Combination 3 = MTX + sulfasalazine; Combination 4 = MTX + hydrochloroquine, chloroquine, chloroquine phosphate + sulfasalazine; Combination 5 = leflunomide only.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Swollen Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Swollen Joints
  DMARD Combination 1 - Month 2 (n=1681) | -4.5 (4.61)
  DMARD Combination 1 - Month 4 (n=1681) | -6.1 (5.07)
  DMARD Combination 1 - Month 6 (n=1681) | -6.9 (5.31)
  DMARD Combination 2 - Month 2 (n=433) | -4.5 (4.91)
  DMARD Combination 2 - Month 4 (n=433) | -6.5 (5.17)
  DMARD Combination 2 - Month 6 (n=433) | -7.3 (5.35)
  DMARD Combination 3 - Month 2 (n=216) | -4.6 (4.68)
  DMARD Combination 3 - Month 4 (n=216) | -6.0 (5.11)
  DMARD Combination 3 - Month 6 (n=216) | -6.7 (5.54)
  DMARD Combination 4 - Month 2 (n=150) | -3.8 (4.58)
  DMARD Combination 4 -Month 4 (n=150) | -5.9 (5.40)
  DMARD Combination 4 - Month 6 (n=150) | -6.7 (6.10)
  DMARD Combination 5 - Month 2 (n=106) | -4.8 (3.89)
  DMARD Combination 5 - Month 4 (n=106) | -6.0 (4.96)
  DMARD Combination 5 - Month 6 (n=106) | -6.2 (4.86)
  DMARD Combination 6 - Month 2 (n=303) | -3.9 (4.27)
  DMARD Combination 6 - Month 4 (n=303) | -5.6 (4.51)
  DMARD Combination 6 - Month 6 (n=303) | -6.2 (4.90)

5. Secondary Outcome: Mean Change From Baseline in the Number of Swollen Joints by Concomitant Corticosteroid Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of swollen joints by participant baseline concomitant corticosteroid treatment was calculated at study Month 2, Month 4, and Month 6 . A total of 28 joints were evaluated.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Swollen Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Swollen Joints
  Did Not Receive Corticosteroids - Month 2 (n=1202) | -4.5 (4.43)
  Did Not Receive Corticosteroids - Month 4 (n=1202) | -6.1 (4.88)
  Did Not Receive Corticosteroids - Month 6 (n=1202) | -6.8 (5.24)
  Received Corticosteroids - Month 2 (n=2078) | -4.3 (4.66)
  Received Corticosteroids - Month 4 (n=2078) | -6.1 (5.10)
  Received Corticosteroids - Month 6 (n=2078) | -6.9 (5.33)

6. Secondary Outcome: Mean Change From Baseline in the Number of Swollen Joints by the Number of DMARD Failures at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the mean number of swollen joints by the number of baseline participant DMARD failures was calculated at study Month 2, Month 4, and Month 6. A total of 28 joints were evaluated.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Swollen Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Swollen Joints
  Failed 1 DMARD - Month 2 (n=1129) | -4.7 (4.81)
  Failed 1 DMARD - Month 4 (n=1129) | -6.3 (5.35)
  Failed 1 DMARD - Month 6 (n=1129) | -7.2 (5.50)
  Failed 2 DMARDs - Month 2 (n=1176) | -4.4 (4.54)
  Failed 2 DMARDs - Month 4 (n=1176) | -6.0 (4.84)
  Failed 2 DMARDs - Month 6 (n=1176) | -6.7 (5.24)
  Failed >=3 DMARDs - Month 2 (n=974) | -4.1 (4.34)
  Failed >=3 DMARDs - Month 4 (n=974) | -5.8 (4.83)
  Failed >=3 DMARDs - Month 6 (n=974) | -6.6 (5.10)

7. Secondary Outcome: Mean Change From Baseline in the Number of Swollen Joints by Duration of Disease at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the mean number of swollen joints was calculated by the participant duration of disease at study Month 2, Month 4, and Month 6. The participant duration of disease is defined as the time since the diagnosis of rheumatoid arthritis. A total of 28 joints were evaluated.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Swollen Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Swollen Joints
  Duration < 2 years - Month 2 (n=899) | -4.4 (4.74)
  Duration < 2 years - Month 4 (n= 899) | -5.9 (5.08)
  Duration < 2 years - Month 6 (n=899) | -6.5 (5.26)
  Duration 2 to <5 years - Month 2 (n=764) | -4.3 (4.63)
  Duration 2 to <5 years - Month 4 (n=764) | -6.0 (5.04)
  Duration 2 to <5 years - Month 6 (n=764) | -6.8 (5.41)
  Duration 5 to 10 years - Month 2 (n=692) | -4.3 (4.49)
  Duration 5 to 10 years - Month 4 (n=692) | -6.1 (4.96)
  Duration 5 to 10 years - Month 6 (n=692) | -6.7 (5.40)
  Duration > 10 years - Month 2 (n=924) | -4.6 (4.45)
  Duration > 10 years - Month 4 (n=924) | -6.2 (4.99)
  Duration > 10 years - Month 6 (n=924) | -7.2 (5.13)

8. Secondary Outcome: Mean Change From Baseline in the Number of Swollen Joints by Baseline Level of Disease Activity at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of swollen joints by participant baseline level of disease activity was calculated at study Month 2, Month 4, and Month 6 by the participant's level of baseline disease activity, as measured by DAS28-ESR. A total of 28 joints were evaluated. DAS28-ESR > 5.1 = high disease activity, DAS28-ESR < 3.2 to < =5.1 = low disease activity, and DAS28-ESR <2.6 = remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Swollen Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Swollen Joints
  DAS28 > 3.2 to <=5.1 - Month 2 (n=698) | -2.4 (3.33)
  DAS28 > 3.2 to <=5.1 - Month 4 (n=698) | -3.4 (3.43)
  DAS28 > 3.2 to <=5.1 - Month 6 (n=698) | -3.8 (3.60)
  DAS28 > 5.1 - Month 2 (n=2572) | -4.9 (4.73)
  DAS28 > 5.1 - Month 4 (n=2572) | -6.8 (5.13)
  DAS28 > 5.1 - Month 6 (n=2572) | -7.7 (5.39)

9. Secondary Outcome: Mean Change From Baseline in the Number of Swollen Joints by Baseline Rheumatoid Factor (RF) Level at Month 2, Month 4, and Month 6
Description: The change from baseline in the mean number of swollen joints was calculated by the participant baseline level of RF at study Month 2, Month 4, and Month 6. A total of 28 joints were evaluated.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Swollen Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Swollen Joints
  RF <=22 IU/mL - Month 2 (n=1026) | -3.9 (4.36)
  RF <=22 IU/mL - Month 4 (n=1026) | -5.5 (4.85)
  RF <=22 IU/mL - Month 6 (n=1026) | -6.2 (5.07)
  RF >22 to <=146 IU/mL - Month 2 (n=1081) | -4.2 (4.47)
  RF >22 to <=146 IU/mL - Month 4 (n=1081) | -5.8 (4.89)
  RF >22 to <=146 IU/mL - Month 6 (n=1081) | -6.4 (5.08)
  RF >146 IU/mL - Month 2 (n=1127) | -5.0 (4.83)
  RF >146 IU/mL - Month 4 (n=1127) | -6.8 (5.25)
  RF >146 IU/mL - Month 6 (n=1127) | -7.8 (5.56)

10. Secondary Outcome: Mean Change From Baseline in the Number of Swollen Joints by Baseline Anti-Cyclic Citrullinated Antibody (Anti-CCP) Level at Month 2, Month 4, and Month 6
Description: The change from baseline in the mean number of swollen joints was calculated by the participant baseline level of anti-CCP at study Month 2, Month 4, and Month 6. A total of 28 joints were evaluated.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Swollen Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Swollen Joints
  Anti-CCP <=40 U/mL - Month 2 (n=1038) | -4.0 (4.44)
  Anti-CCP <=40 U/mL - Month 4 (n=1038) | -5.7 (4.89)
  Anti-CCP <=40 U/mL - Month 6 (n=1038) | -6.5 (5.16)
  Anti-CCP >40 to <=380 U/mL - Month 2 (n=1112) | -4.4 (4.41)
  Anti-CCP >40 to <=380 U/mL - Month 4 (n=1112) | -6.1 (4.92)
  Anti-CCP >40 to <=380 U/mL - Month 6 (n=1112) | -6.7 (5.23)
  Anti-CCP >380 U/mL - Month 2 (n=1075) | -4.8 (4.86)
  Anti-CCP >380 U/mL - Month 4 (n=1075) | -6.3 (5.30)
  Anti-CCP >380 U/mL - Month 6 (n=1075) | -7.3 (5.51)

11. Secondary Outcome: Mean Change From Baseline in the Number of Swollen Joints by Smoking History at Month 2, Month 4, and Month 6
Description: The change from baseline in the mean number of swollen joints was calculated by the baseline participant smoking status at study Month 2, Month 4, and Month 6. A total of 28 joints were evaluated. Pack years smoked is defined as the total number of packs smoked per day multiplied by the number of years the participant smoked.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Swollen Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Swollen Joints
  Non-Smoker - Month 2 (n=1963) | -4.7 (4.66)
  Non-Smoker - Month 4 (n=1963) | -6.5 (5.05)
  Non-Smoker - Month 6 (n=1963) | -7.3 (5.35)
  Smoking history >=20 years - Month 2 (n=324) | -4.4 (4.43)
  Smoking history >=20 years - Month 4 (n=324) | -5.5 (5.22)
  Smoking history >=20 years - Month 6 (n=324) | -6.5 (5.35)
  Smoking history <20 years - Month 2 (n=314) | -4.0 (4.32)
  Smoking history <20 years - Month 4 (n=314) | -5.4 (4.64)
  Smoking history <20 years - Month 6 (n=314) | -6.1 (4.85)
  Currently smokes <0.5 packs/day - Month 2 (n=223) | -4.0 (4.71)
  Currently smokes <0.5 packs/day - Month 4 (n=223) | -6.1 (4.87)
  Currently smokes <0.5 pack/day - Month 6 (n=223) | -6.6 (5.26)
  Currently smokes 0.5-1 pack/day - Month 2 (n=397) | -3.6 (4.11)
  Currently smokes 0.5-1 pack/day - Month 4 (n=397) | -5.0 (4.59)
  Currently smokes 0.5-1 pack/day - Month 6 (n=397) | -5.5 (4.95)
  Currently smokes >1 packs/day - Month 2 (n=59) | -4.0 (5.6)
  Currently smokes >1 packs/day - Month 4 (n=59) | -4.8 (6.25)
  Currently smokes >1 packs/day - Month 6 (n=59) | -5.0 (5.46)
  Pack years <7.5 - Month 2 (n=423) | -4.2 (4.68)
  Pack years <7.5 - Month 4 (n=423) | -6.0 (5.04)
  Pack years <7.5 - Month 6 (n=423) | -6.5 (5.21)
  Pack years 7.5 to 20.5 - Month 2 (n=454) | -3.8 (4.12)
  Pack years 7.5 to 20.5 - Month 4 (n=454) | -5.3 (4.84)
  Pack years 7.5 to 20.5 - Month 6 (n=454) | -5.9 (5.17)
  Pack years >20.5 - Month 2 (n=418) | -3.9 (4.35)
  Pack years >20.5 - Month 4 (n=418) | -5.0 (4.77)
  Pack years >20.5 - Month 6 (n=418) | -5.8 (5.01)

12. Secondary Outcome: Mean Change From Baseline in the Number of Swollen Joints by Eligibility for Anti-Tumor Necrosis Factor (Anti-TNF) Treatment at Month 2, Month 4, and Month 6
Description: The change from baseline in the mean number of swollen joints was calculated by the baseline participant eligibility for anti-TNF treatment at study Month 2, Month 4, and Month 6. A total of 28 joints were evaluated.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Swollen Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Swollen Joints
  Anti-TNF treatment Ineligible - Month 2 (n=106) | -3.1 (3.34)
  Anti-TNF treatment Ineligible - Month 4 (n=106) | -4.4 (3.82)
  Anti-TNF treatment Ineligible - Month 6 (n=106) | -4.5 (3.81)
  Anti-TNF treatment Eligible - Month 2 (n=3174) | -4.4 (4.61)
  Anti-TNF treatment Eligible - Month 4 (n=3174) | -6.1 (5.05)
  Anti-TNF treatment Eligible - Month 6 (n=3174) | -6.9 (5.32)

13. Secondary Outcome: Mean Change From Baseline in the Number of Swollen Joints by Participant Baseline Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of swollen joints was calculated by the participant baseline expectation of treatment outcome at study Month 2, Month 4, Month 6. A total of 28 joints were evaluated. The participant expectation scale was evaluated by questionnaire for a categorical score of 1 (best) to 5 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: The efficacy evaluable population comprised all participants with a baseline DAS28-ESR and at least one post-baseline measurement of DAS28-ESR. n values represent the number of participants at baseline. Participants were grouped by participant expectation score into 3 groups: <=1.5, >1.5 to <1.86, and >=1.86.
Measure: Mean (Standard Deviation); unit: Swollen Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Swollen Joints
  <=1.5 - Month 2 (n=1212) | -4.8 (4.68)
  <=1.5 - Month 4 (n=1212) | -6.4 (5.14)
  <=1.5 - Month 6 (n=1212) | -7.3 (5.40)
  >1.5 to 1.86 - Month 2 (n=1009) | -4.4 (4.54)
  >1.5 to 1.86 - Month 4 (n=1009) | -6.2 (5.09)
  >1.5 to 1.86 - Month 6 (n=1009) | -6.9 (5.28)
  >=1.86 - Month 2 (n=1054) | -3.9 (4.46)
  >=1.86 - Month 4 (n=1054) | -5.5 (4.77)
  >=1.86 - Month 6 (n=1054) | -6.3 (5.13)

14. Secondary Outcome: Mean Change From Baseline in the Number of Swollen Joints by Physician Experience Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of swollen joints was calculated by the physician experience level at study Month 2, Month 4, Month 6. A total of 28 joints were evaluated. Physician experience is defined as the number of years the treating physician has experience managing rheumatoid arthritis.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Swollen Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Swollen Joints
  <=10 years - Month 2 (n=1305) | -4.2 (4.49)
  <=10 years - Month 4 (n=1305) | -5.8 (4.88)
  <=10 years - Month 6 (n =1305) | -6.5 (5.13)
  >10 to 20 years - Month 2 (n=1105) | -4.7 (4.83)
  >10 to 20 years - Month 4 (n=1105) | -6.4 (5.35)
  >10 to 20 years - Month 6 (n=1105) | -7.2 (5.42)
  >20 years - Month 2 (n=850) | -4.3 (4.35)
  >20 years - Month 4 (n=850) | -6.0 (4.77)
  >20 years - Month 6 (n=850) | -6.8 (5.32)

15. Secondary Outcome: Mean Change From Baseline in the Number of Swollen Joints by Physician Experience Level With Biologics at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of swollen joints was calculated by the physician experience level with biologics at study Month 2, Month 4, and Month 6. A total of 28 joints were evaluated. Physician experience is defined as the number of years the treating physician has experience managing rheumatoid arthritis with biologics.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Swollen Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Swollen Joints
  0 to 6 years - Month 2 (n=1160) | -4.2 (4.52)
  0 to 6 years - Month 4 (n=1160) | -5.9 (5.09)
  0 to 6 years - Month 6 (n=1160) | -6.9 (5.35)
  6 to 10 years - Month 2 (n=1745) | -4.5 (4.63)
  6 to 10 years - Month 4 (n=1745) | -6.2 (4.98)
  6 to 10 years - Month 6 (n=1745) | -6.8 (5.26)
  >10 years - Month 2 (n=355) | -4.3 (4.49)
  >10 years - Month 4 (n=355) | -5.9 (4.98)
  >10 years - Month 6 (n=355) | -6.6 (5.18)

16. Secondary Outcome: Mean Change From Baseline in the Number of Swollen Joints by the Number of Patients Treated by the Physician With Biologics at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of swollen joints was calculated by the baseline number of patients the physician treats with biologics at study Month 2, Month 4, and Month 6. A total of 28 joints were evaluated. The number of patients treated with biologics is defined as the number of patients treated by the physician in the last month with biologics for rheumatoid arthritis.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Swollen Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Swollen Joints
  1-17 patients in prior month - Month 2 (n=1056) | -4.3 (4.59)
  1-17 patients in prior month - Month 4 (n=1056) | -6.2 (5.00)
  1-17 patients in prior month - Month 6 (n=1056) | -7.4 (5.40)
  18-34 patients in prior month - Month 2 (n=1061) | -4.5 (4.52)
  18-34 patients in prior month - Month 4 (n=1061) | -6.1 (4.98)
  18-34 patients in prior month - Month 6 (n=1061) | -6.8 (5.02)
  >=35 patients in prior month - Month 2 (n=1097) | -4.5 (4.60)
  >=35 patients in prior month - Month 4 (n=1097) | -6.1 (4.98)
  >=35 patients in prior month - Month 6 (n=1097) | -6.8 (5.02)

17. Secondary Outcome: Mean Change From Baseline in the Number of Swollen Joints by the the Physician Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of swollen joints was calculated by the physician's expectation of treatment outcome at study Month 2, Month 4, and Month 6. A total of 28 joints were evaluated. The physician's expectation of treatment outcomes was assessed at the start of Month 4 at which time physicians were asked to rate their expectations of treatment outcome in each participant as: high disease activity, moderate disease activity, low disease activity, or remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Swollen Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Swollen Joints
  High disease activity - Month 2 (n=40) | -5.5 (4.74)
  High disease activity - Month 4 (n=40) | -7.1 (4.21)
  High disease activity - Month 6 (n=40) | -8.2 (4.77)
  Moderate disease activity - Month 2 (n=325) | -4.9 (4.98)
  Moderate disease activity - Month 4 (n=325) | -6.3 (4.94)
  Moderate disease activity - Month 6 (n=325) | -7.2 (5.75)
  Low disease activity - Month 2 (n=1932) | -4.2 (4.53)
  Low disease activity - Month 4 (n=1932) | -6.0 (5.12)
  Low disease activity - Month 6 (n=1932) | -6.9 (5.23)
  Remission - Month 2 (n=966) | -4.6 (4.50)
  Remission - Month 4 (n=966) | -6.0 (4.84)
  Remission - Month 6 (n=966) | -6.5 (5.24)

18. Secondary Outcome: Mean Change From Baseline in the Number of Tender Joints by Concomitant MTX Dose at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of tender joints was calculated by participant concomitant MTX dose (low < 10mg/wk, medium >= 10 to < 15 mg/week, and high >=15 mg/week) at study Month 2, Month 4, and Month 6. A total of 28 joints were evaluated.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Tender Joints
  Low MTX Dose - Month 2 (n=142) | -5.5 (5.82)
  Low MTX Dose - Month 4 (n=142) | -7.9 (6.67)
  Low MTX Dose - Month 6 (n=142) | -9.0 (6.82)
  Medium MTX Dose - Month 2 (n=526) | -5.6 (5.76)
  Medium MTX Dose - Month 4 (n=526) | -8.0 (6.52)
  Medium MTX Dose - Month 6 (n=526) | -9.1 (6.57)
  High MTX Dose - Month 2 (n=1995) | -5.5 (5.91)
  High MTX Dose - Month 4 (n=1995) | -7.8 (6.48)
  High MTX Dose - Month 6 (n=1995) | -8.7 (6.72)

19. Secondary Outcome: Mean Change From Baseline in the Number of Tender Joints by Concomitant DMARD Background Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of tender joints was calculated by participant background DMARD treatment at study Month 2, Month 4, and Month 6. A total of 28 joints were evaluated. DMARD Combination 1 = MTX + hydrochloroquine, chloroquine, chloroquine phosphate; Combination 2 = MTX + leflunomide; Combination 3 = MTX + sulfasalazine; Combination 4 = MTX + hydrochloroquine, chloroquine, chloroquine phosphate + sulfasalazine; Combination 5 = leflunomide only.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Tender Joints
  DMARD Combination 1 - Month 2 (n=1681) | -5.5 (5.56)
  DMARD Combination 1 - Month 4 (n=1681) | -7.8 (6.39)
  DMARD Combination 1 - Month 6 (n=1681) | -8.7 (6.58)
  DMARD Combination 2 - Month 2 (n=433) | -5.7 (6.37)
  DMARD Combination 2 - Month 4 (n=433) | -8.0 (6.81)
  DMARD Combination 2 - Month 6 (n=433) | -9.2 (6.46)
  DMARD Combination 3 - Month 2 (n=216) | -5.6 (6.86)
  DMARD Combination 3 - Month 4 (n=216) | -7.6 (6.87)
  DMARD Combination 3 - Month 6 (n=216) | -8.2 (7.52)
  DMARD Combination 4 - Month 2 (n=150) | -5.5 (6.11)
  DMARD Combination 4 -Month 4 (n=150) | -8.0 (6.92)
  DMARD Combination 4 - Month 6 (n=150) | -9.2 (7.44)
  DMARD Combination 5 - Month 2 (n=106) | -5.4 (5.72)
  DMARD Combination 5 - Month 4 (n=106) | -8.3 (5.81)
  DMARD Combination 5 - Month 6 (n=106) | -8.4 (7.07)
  DMARD Combination 6 - Month 2 (n=303) | -5.1 (5.77)
  DMARD Combination 6 - Month 4 (n=303) | -7.5 (6.37)
  DMARD Combination 6 - Month 6 (n=303) | -8.0 (6.68)

20. Secondary Outcome: Mean Change From Baseline in the Number of Tender Joints by Concomitant Corticosteroid Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of tender joints was calculated by participant baseline concomitant steroid treatment at study Month 2, Month 4, and Month 6. A total 28 joints were evaluated.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Tender Joints
  Did Not Receive Corticosteroids - Month 2 (n=1202) | -5.4 (5.54)
  Did Not Receive Corticosteroids - Month 4 (n=1202) | -7.6 (6.31)
  Did Not Receive Corticosteroids - Month 6 (n=1202) | -8.6 (6.44)
  Received Corticosteroids - Month 2 (n=2078) | -5.6 (5.99)
  Received Corticosteroids - Month 4 (n=2078) | -7.8 (6.61)
  Received Corticosteroids - Month 6 (n=2078) | -8.7 (6.85)

21. Secondary Outcome: Mean Change From Baseline in the Number of Tender Joints by the Number of DMARD Failures at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of tender joints was calculated by the number of participant DMARD failures at baseline at study Month 2, Month 4, Month 6. A total of 28 joints were evaluated.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Tender Joints
  Failed 1 DMARD - Month 2 (n=1129) | -5.8 (5.74)
  Failed 1 DMARD - Month 4 (n=1129) | -7.8 (6.65)
  Failed 1 DMARD - Month 6 (n=1129) | -8.8 (6.94)
  Failed 2 DMARDs - Month 2 (n=1176) | -5.5 (6.02)
  Failed 2 DMARDs - Month 4 (n=1176) | -7.7 (6.64)
  Failed 2 DMARDs - Month 6 (n=1176) | -8.7 (6.64)
  Failed >=3 DMARDs - Month 2 (n=974) | -5.1 (5.68)
  Failed >=3 DMARDs - Month 4 (n=974) | -7.6 (6.15)
  Failed >=3 DMARDs - Month 6 (n=974) | -8.4 (6.48)

22. Secondary Outcome: Mean Change From Baseline in the Number of Tender Joints by Duration of Disease at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of tender joints was calculated by the participant duration of disease at study Month 2, Month 4, and Month 6. Duration of disease is defined as the time since the diagnosis of rheumatoid arthritis. A total of 28 joints were evaluated.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Tender Joints
  Duration < 2 years - Month 2 (n=899) | -5.4 (6.03)
  Duration < 2 years - Month 4 (n=899) | -7.4 (6.78)
  Duration < 2 years - Month 6 (n=899) | -8.3 (6.59)
  Duration 2 to <5 years - Month 2 (n=764) | -5.9 (5.95)
  Duration 2 to <5 years - Month 4 (n=764) | -8.2 (6.43)
  Duration 2 to <5 years - Month 6 (n=764) | -8.9 (6.86)
  Duration 5 to 10 years - Month 2 (n=692) | -5.3 (5.52)
  Duration 5 to 10 years - Month 4 (n=692) | -7.7 (6.27)
  Duration 5 to 10 years - Month 6 (n=692) | -8.6 (6.66)
  Duration > 10 years - Month 2 (n=924) | -5.4 (5.74)
  Duration > 10 years - Month 4 (n=924) | -7.6 (6.45)
  Duration > 10 years - Month 6 (n=924) | -8.7 (6.67)

23. Secondary Outcome: Mean Change From Baseline in the Number of Tender Joints by Baseline Level of Disease Activity at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of tender joints was calculated by the participant baseline level of disease activity, as measured by DAS28, at study Month 2, Month 4, and Month 6. A total of 28 joints were evaluated. DAS28-ESR > 5.1 = high disease activity, DAS28-ESR < 3.2 to < =5.1 = low disease activity, and DAS28-ESR <2.6 = remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Tender Joints
  DAS28 > 3.2 to <=5.1 - Month 2 (n=698) | -2.9 (4.10)
  DAS28 > 3.2 to <=5.1 - Month 4 (n=698) | -3.8 (4.42)
  DAS28 > 3.2 to <=5.1 - Month 6 (n=698) | -4.0 (4.59)
  DAS28 > 5.1 - Month 2 (n=2572) | -6.2 (6.00)
  DAS28 > 5.1 - Month 4 (n=2572) | -8.8 (6.55)
  DAS28 > 5.1 - Month 6 (n=2572) | -9.9 (6.62)

24. Secondary Outcome: Mean Change From Baseline in the Number of Tender Joints by Baseline RF Level at Month 2, Month 4, and Month 6
Description: The change from baseline in the mean number of tender joints was calculated by the participant baseline level of RF at study Month 2, Month 4, and Month 6. A total of 28 joints were evaluated.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Tender Joints
  RF <=22 IU/mL - Month 2 (n=1026) | -5.0 (5.82)
  RF <=22 IU/mL - Month 4 (n=1026) | -7.2 (6.60)
  RF <=22 IU/mL - Month 6 (n=1026) | -8.1 (6.76)
  RF >22 to <=146 IU/mL - Month 2 (n=1081) | -5.4 (5.46)
  RF >22 to <=146 IU/mL - Month 4 (n=1081) | -7.6 (6.20)
  RF >22 to <=146 IU/mL - Month 6 (n=1081) | -8.5 (6.36)
  RF >146 IU/mL - Month 2 (n=1127) | -6.1 (6.16)
  RF >146 IU/mL - Month 4 (n=1127) | -8.3 (6.69)
  RF >146 IU/mL - Month 6 (n=1127) | -9.3 (6.97)

25. Secondary Outcome: Mean Change From Baseline in the Number of Tender Joints by Baseline Anti-CCP Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of tender joints was calculated by the participant baseline level of anti-CCP at study Month 2, Month 4, and Month 6. A total of 28 joints were evaluated.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Tender Joints
  Anti-CCP <=40 U/mL - Month 2 (n=1038) | -5.0 (5.78)
  Anti-CCP <=40 U/mL - Month 4 (n=1038) | -7.2 (6.64)
  Anti-CCP <=40 U/mL - Month 6 (n=1038) | -8.1 (6.73)
  Anti-CCP >40 to <=380 U/mL - Month 2 (n=1112) | -5.7 (5.73)
  Anti-CCP >40 to <=380 U/mL - Month 4 (n=1112) | -8.0 (6.39)
  Anti-CCP >40 to <=380 U/mL - Month 6 (n=1112) | -8.8 (6.72)
  Anti-CCP >380 U/mL - Month 2 (n=1075) | -5.8 (5.95)
  Anti-CCP >380 U/mL - Month 4 (n=1075) | -7.9 (6.49)
  Anti-CCP >380 U/mL - Month 6 (n=1075) | -9.0 (6.65)

26. Secondary Outcome: Mean Change From Baseline in the Number of Tender Joints by Smoking History at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of tender joints was calculated by the baseline participant smoking status at study Month 2, Month 4, and Month 6. A total of 28 joints were evaluated. Pack years smoked is defined as the total number of packs smoked per day multiplied by the number of years the participant smoked.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Tender Joints
  Non-Smoker - Month 2 (n=1963) | -5.8 (5.86)
  Non-Smoker - Month 4 (n=1963) | -8.2 (6.49)
  Non-Smoker - Month 6 (n=1963) | -9.2 (6.59)
  Smoking history >=20 years - Month 2 (n=324) | -5.5 (5.97)
  Smoking history >=20 years - Month 4 (n=324) | -7.4 (6.73)
  Smoking history >=20 years - Month 6 (n=324) | -8.7 (6.77)
  Smoking history <20 years - Month 2 (n=314) | -5.7 (5.74)
  Smoking history <20 years - Month 4 (n=314) | -7.5 (6.12)
  Smoking history <20 years - Month 6 (n=314) | -8.4 (6.51)
  Currently smokes <0.5 packs/day - Month 2 (n=223) | -4.6 (5.11)
  Currently smokes <0.5 packs/day - Month 4 (n=223) | -7.2 (6.67)
  Currently smokes <0.5 pack/day - Month 6 (n=223) | -8.2 (6.84)
  Currently smokes 0.5-1 pack/day - Month 2 (n=397) | -4.4 (5.67)
  Currently smokes 0.5-1 pack/day - Month 4 (n=397) | -6.4 (6.36)
  Currently smokes 0.5-1 pack/day - Month 6 (n=397) | -6.7 (6.70)
  Currently smokes >1 packs/day - Month 2 (n=59) | -5.2 (6.83)
  Currently smokes >1 packs/day - Month 4 (n=59) | -6.9 (6.49)
  Currently smokes >1 packs/day - Month 6 (n=59) | -7.5 (7.64)
  Pack years <7.5 - Month 2 (n=423) | -5.4 (5.51)
  Pack years <7.5 - Month 4 (n=423) | -7.5 (6.37)
  Pack years <7.5 - Month 6 (n=423) | -8.4 (6.77)
  Pack years 7.5 to 20.5 - Month 2 (n=454) | -5.2 (5.67)
  Pack years 7.5 to 20.5 - Month 4 (n=454) | -7.6 (6.37)
  Pack years 7.5 to 20.5 - Month 6 (n=454) | -8.1 (6.80)
  Pack years >20.5 - Month 2 (n=418) | -4.5 (5.76)
  Pack years >20.5 - Month 4 (n=418) | -6.1 (6.29)
  Pack years >20.5 - Month 6 (n=418) | -7.1 (6.61)

27. Secondary Outcome: Mean Change From Baseline in the Number of Tender Joints by Eligibility for Anti-TNF Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of tender joints was calculated by the baseline participant eligibility for anti-TNF treatment at study Month 2, Month 4, and Month 6. A total of 28 joints were evaluated.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Tender Joints
  Anti-TNF treatment Ineligible - Month 2 (n=106) | -4.6 (4.75)
  Anti-TNF treatment Ineligible - Month 4 (n=106) | -7.0 (5.68)
  Anti-TNF treatment Ineligible - Month 6 (n=106) | -7.0 (5.70)
  Anti-TNF treatment Eligible - Month 2 (n=3174) | -5.5 (5.86)
  Anti-TNF treatment Eligible - Month 4 (n=3174) | -7.7 (6.53)
  Anti-TNF treatment Eligible - Month 6 (n=3174) | -8.7 (6.72)

28. Secondary Outcome: Mean Change From Baseline in the Number of Tender Joints by Participant Baseline Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of tender joints was calculated by the participant baseline expectation of treatment outcome at study Month 2, Month 4, Month 6. A total of 28 joints were evaluated. The participant expectation scale was evaluated by questionnaire for a categorical score of 1 (best) to 5 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Tender Joints
  <=1.5 - Month 2 (n=1212) | -6.1 (5.97)
  <=1.5 - Month 4 (n=1212) | -8.2 (6.40)
  <=1.5 - Month 6 (n=1212) | -9.2 (6.69)
  >1.5 to 1.86 - Month 2 (n=1009) | -5.5 (5.73)
  >1.5 to 1.86 - Month 4 (n=1009) | -7.9 (6.67)
  >1.5 to 1.86 - Month 6 (n=1009) | -8.8 (6.77)
  >=1.86 - Month 2 (n=1054) | -4.8 (5.67)
  >=1.86 - Month 4 (n=1054) | -6.9 (6.39)
  >=1.86 - Month 6 (n=1054) | -7.8 (6.58)

29. Secondary Outcome: Mean Change From Baseline in the Number of Tender Joints by Physician Experience Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of tender joints was calculated by the physician experience level at study Month 2, Month 4, Month 6. A total of 28 joints were evaluated. Physician experience is defined as the number of years the treating physician has experience managing rheumatoid arthritis.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Tender Joints
  <=10 years - Month 2 (n=1305) | -5.3 (5.80)
  <=10 years - Month 4 (n=1305) | -7.9 (6.41)
  <=10 years - Month 6 (n=1305) | -8.7 (6.58)
  >10 to 20 years - Month 2 (n=1105) | -5.6 (5.80)
  >10 to 20 years - Month 4 (n=1105) | -7.7 (6.48)
  >10 to 20 years - Month 6 (n=1105) | -8.8 (6.59)
  >20 years - Month 2 (n=850) | -5.5 (5.89)
  >20 years - Month 4 (n=850) | -7.6 (6.69)
  >20 years - Month 6 (n=850) | -8.4 (7.01)

30. Secondary Outcome: Mean Change From Baseline in the Number of Tender Joints by Physician Experience Level With Biologics at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of tender joints was calculated by the physician experience level with biologics at study Month 2, Month 4, and Month 6. A total of 28 joints were evaluated. Physician experience is defined as the number of years the treating physician has experience managing rheumatoid arthritis with biologics.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Tender Joints
  0 to 6 years - Month 2 (n=1160) | -5.5 (5.93)
  0 to 6 years - Month 4 (n=1160) | -8.0 (6.54)
  0 to 6 years - Month 6 (n=1160) | -8.9 (6.76)
  6 to 10 years - Month 2 (n=1745) | -5.5 (5.78)
  6 to 10 years - Month 4 (n=1745) | -7.6 (6.51)
  6 to 10 years - Month 6 (n=1745) | -8.6 (6.61)
  >10 years - Month 2 (n=355) | -5.3 (5.66)
  >10 years - Month 4 (n=355) | -7.4 (6.34)
  >10 years - Month 6 (n=355) | -8.0 (6.90)

31. Secondary Outcome: Mean Change From Baseline in the Number of Tender Joints by the Number of Patients Treated by the Physician With Biologics at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of tender joints was calculated by the baseline number of patients the physician treats with biologics at study Month 2, Month 4, and Month 6. A total of 28 joints were evaluated. The number of patients treated with biologics is defined as the number of patients treated by the physician in the last month with biologics for rheumatoid arthritis.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Tender Joints
  1-17 patients in prior month - Month 2 (n=1056) | -5.5 (5.95)
  1-17 patients in prior month - Month 4 (n=1056) | -8.0 (6.33)
  1-17 patients in prior month - Month 6 (n=1056) | -9.2 (6.62)
  18-34 patients in prior month - Month 2 (n=1061) | -5.7 (5.69)
  18-34 patients in prior month - Month 4 (n=1061) | -7.8 (6.59)
  18-34 patients in prior month - Month 6 (n=1061) | -8.6 (6.44)
  >=35 patients in prior month - Month 2 (n=1097) | -5.3 (5.79)
  >=35 patients in prior month - Month 4 (n=1097) | -7.5 (6.54)
  >=35 patients in prior month - Month 6 (n=1097) | -8.2 (6.93)

32. Secondary Outcome: Mean Change From Baseline in the Number of Tender Joints by the the Physician Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the number of tender joints. was calculated by the physician's expectation of treatment outcome at study Month 2, Month 4, and Month 6. A total of 28 joints were evaluated. The physician's expectation of treatment outcomes was assessed at the start of Month 4 at which time physicians were asked to rate their expectations of treatment outcome in each participant as: high disease activity, moderate disease activity, low disease activity, or remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Tender Joints
  High disease activity - Month 2 (n=40) | -7.2 (5.80)
  High disease activity - Month 4 (n=40) | -9.4 (6.32)
  High disease activity - Month 6 (n=40) | -10.4 (6.32)
  Moderate disease activity - Month 2 (n=325) | -5.0 (6.02)
  Moderate disease activity - Month 4 (n=325) | -7.3 (6.83)
  Moderate disease activity - Month 6 (n=325) | -8.3 (6.82)
  Low disease activity - Month 2 (n=1932) | -5.5 (5.86)
  Low disease activity - Month 4 (n=1932) | -7.9 (6.58)
  Low disease activity - Month 6 (n=1932) | -8.9 (6.85)
  Remission - Month 2 (n=966) | -5.6 (5.68)
  Remission - Month 4 (n=966) | -7.5 (6.22)
  Remission - Month 6 (n=966) | -8.3 (6.32)

33. Secondary Outcome: Mean Change From Baseline in Participant Global Assessment of Disease Activity by Concomitant MTX Dose at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant global assessment of disease activity was calculated by concomitant MTX dose (low < 10mg/wk, medium >= 10 to < 15 mg/week, and high >=15 mg/week) at study Month 2, Month 4, and Month 6. The participant global assessment of disease activity was evaluated using a visual analogue scale (VAS; 0mm [best] -100mm [worst]) with increasing scores indicating increased level of disease.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Low MTX Dose - Month 2 (n=142) | -23.1 (24.89)
  Low MTX Dose - Month 4 (n=142) | -29.3 (26.58)
  Low MTX Dose - Month 6 (n=142) | -27.9 (29.33)
  Medium MTX Dose - Month 2 (n=526) | -22.6 (22.99)
  Medium MTX Dose - Month 4 (n=526) | -28.9 (24.93)
  Medium MTX Dose - Month 6 (n=526) | -32.4 (27.85)
  High MTX Dose - Month 2 (n=1995) | -20.3 (25.07)
  High MTX Dose - Month 4 (n=1995) | -26.2 (27.46)
  High MTX Dose - Month 6 (n=1995) | -30.0 (28.68)

34. Secondary Outcome: Mean Change From Baseline in Participant Global Assessment of Disease Activity by Concomitant DMARD Background Treatment at Month 2, Month 4, and Month 6
Description: The participant global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease. DMARD Combination 1 = MTX + hydrochloroquine, chloroquine, chloroquine phosphate; Combination 2 = MTX + leflunomide; Combination 3 = MTX + sulfasalazine; Combination 4 = MTX + hydrochloroquine, chloroquine, chloroquine phosphate + sulfasalazine; Combination 5 = leflunomide only.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  DMARD Combination 1 - Month 2 (n=1681) | -21.2 (24.61)
  DMARD Combination 1 - Month 4 (n=1681) | -27.5 (27.23)
  DMARD Combination 1 - Month 6 (n=1681) | -30.7 (28.48)
  DMARD Combination 2 - Month 2 (n=433) | -19.2 (24.84)
  DMARD Combination 2 - Month 4 (n=433) | -26.4 (27.18)
  DMARD Combination 2 - Month 6 (n=433) | -30.8 (29.14)
  DMARD Combination 3 - Month 2 (n=216) | -19.8 (25.82)
  DMARD Combination 3 - Month 4 (n=216) | -23.8 (28.38)
  DMARD Combination 3 - Month 6 (n=216) | -26.4 (28.74)
  DMARD Combination 4 - Month 2 (n=150) | -23.3 (25.13)
  DMARD Combination 4 -Month 4 (n=150) | -27.2 (24.16)
  DMARD Combination 4 - Month 6 (n=150) | -32.1 (28.95)
  DMARD Combination 5 - Month 2 (n=106) | -21.1 (23.93)
  DMARD Combination 5 - Month 4 (n=106) | -27.3 (24.14)
  DMARD Combination 5 - Month 6 (n=106) | -28.9 (28.75)
  DMARD Combination 6 - Month 2 (n=303) | -21.8 (24.95)
  DMARD Combination 6 - Month 4 (n=303) | -26.5 (28.61)
  DMARD Combination 6 - Month 6 (n=303) | -29.5 (29.29)

35. Secondary Outcome: Mean Change From Baseline in Participant Global Assessment of Disease Activity by Concomitant Corticosteroid Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the participant global assessment of disease activity by participant concomitant corticosteroid use was calculated at study Month 2, Month 4, and Month 6. The participant global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Did Not Receive Corticosteroids - Month 2 (n=1202) | -20.5 (23.98)
  Did Not Receive Corticosteroids - Month 4 (n=1202) | -27.0 (26.90)
  Did Not Receive Corticosteroids - Month 6 (n=1202) | -29.2 (28.68)
  Received Corticosteroids - Month 2 (n=2078) | -21.3 (25.04)
  Received Corticosteroids - Month 4 (n=2078) | -26.4 (27.33)
  Received Corticosteroids - Month 6 (n=2078) | -30.7 (28.42)

36. Secondary Outcome: Mean Change From Baseline in Participant Global Assessment of Disease Activity Score by the Number of DMARD Failures at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the participant global assessment of disease activity score by the number of participant DMARD failures was calculated at study Month 2, Month 4, and Month 6. The participant global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Failed 1 DMARD - Month 2 (n=1129) | -20.9 (23.98)
  Failed 1 DMARD - Month 4 (n=1129) | -27.1 (28.25)
  Failed 1 DMARD - Month 6 (n=1129) | -29.9 (29.42)
  Failed 2 DMARDs - Month 2 (n=1176) | -20.8 (24.56)
  Failed 2 DMARDs - Month 4 (n=1176) | -26.1 (26.67)
  Failed 2 DMARDs - Month 6 (n=1176) | -30.1 (28.58)
  Failed >=3 DMARDs - Month 2 (n=974) | -21.3 (23.73)
  Failed >=3 DMARDs - Month 4 (n=974) | -26.8 (26.52)
  Failed >=3 DMARDs - Month 6 (n=974) | -30.4 (27.43)

37. Secondary Outcome: Mean Change From Baseline in Participant Global Assessment of Disease Activity by Duration of Disease at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the participant global assessment of disease activity by the participant duration of disease was calculated at study Month 2, Month 4, and Month 6. The duration of disease is defined as the time since the diagnosis of rheumatoid arthritis. The participant global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Duration < 2 years - Month 2 (n=899) | -19.4 (25.51)
  Duration < 2 years - Month 4 (n=899) | -25.6 (28.21)
  Duration < 2 years - Month 6 (n=899) | -29.5 (29.45)
  Duration 2 to <5 years - Month 2 (n=764) | -20.9 (24.33)
  Duration 2 to <5 years - Month 4 (n=764) | -25.9 (27.38)
  Duration 2 to <5 years - Month 6 (n=764) | -28.9 (28.26)
  Duration 5 to 10 years - Month 2 (n=692) | -22.2 (24.76)
  Duration 5 to 10 years - Month 4 (n=692) | -27.8 (26.51)
  Duration 5 to 10 years - Month 6 (n=692) | -30.2 (28.36)
  Duration > 10 years - Month 2 (n=924) | -21.8 (23.96)
  Duration > 10 years - Month 4 (n=924) | -27.3 (26.46)
  Duration > 10 years - Month 6 (n=924) | -31.8 (27.91)

38. Secondary Outcome: Mean Change From Baseline in Participant Global Assessment of Disease Activity by Baseline Level of Disease Activity at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the participant global assessment of disease activity by the participant baseline level of disease activity was calculated at study Month 2, Month 4, and Month 6. The participant global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  DAS28 > 3.2 to <=5.1 - Month 2 (n=698) | -16.0 (23.68)
  DAS28 > 3.2 to <=5.1 - Month 4 (n=698) | -20.0 (26.21)
  DAS28 > 3.2 to <=5.1 - Month 6 (n=698) | -22.6 (27.31)
  DAS28 > 5.1 - Month 2 (n=2572) | -22.4 (24.73)
  DAS28 > 5.1 - Month 4 (n=2572) | -28.5 (27.15)
  DAS28 > 5.1 - Month 6 (n=2572) | -32.3 (28.47)

39. Secondary Outcome: Mean Change From Baseline in Participant Global Assessment of Disease Activity by Baseline RF Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the participant global assessment of disease activity by the participant baseline RF level was calculated at study Month 2, Month 4, and Month 6. The participant global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  RF <=22 IU/mL - Month 2 (n=1026) | 18.0 (24.82)
  RF <=22 IU/mL - Month 4 (n=1026) | -24.7 (27.89)
  RF <=22 IU/mL - Month 6 (n=1026) | -27.6 (28.48)
  RF >22 to <=146 IU/mL - Month 2 (n=1081) | -20.7 (24.07)
  RF >22 to <=146 IU/mL - Month 4 (n=1081) | -25.7 (26.77)
  RF >22 to <=146 IU/mL - Month 6 (n=1081) | -28.5 (28.15)
  RF >146 IU/mL - Month 2 (n=1127) | -24.2 (24.81)
  RF >146 IU/mL - Month 4 (n=1127) | -29.6 (26.72)
  RF >146 IU/mL - Month 6 (n=1127) | -34.2 (28.54)

40. Secondary Outcome: Mean Change From Baseline in Participant Global Assessment of Disease Activity by Baseline Anti-CCP Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the participant global assessment of disease activity by the participant baseline serum level of anti-CCP was calculated at study Month 2, Month 4, and Month 6. The participant global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Anti-CCP <=40 U/mL - Month 2 (n=1038) | -17.2 (24.22)
  Anti-CCP <=40 U/mL - Month 4 (n=1038) | -23.3 (27.04)
  Anti-CCP <=40 U/mL - Month 6 (n=1038) | -27.4 (28.21)
  Anti-CCP >40 to <=380 U/mL - Month 2 (n=1112) | -22.6 (25.23)
  Anti-CCP >40 to <=380 U/mL - Month 4 (n=1112) | -28.1 (27.86)
  Anti-CCP >40 to <=380 U/mL - Month 6 (n=1112) | -29.7 (28.88)
  Anti-CCP >380 U/mL - Month 2 (n=1075) | -23.1 (23.99)
  Anti-CCP >380 U/mL - Month 4 (n=1075) | -28.4 (26.44)
  Anti-CCP >380 U/mL - Month 6 (n=1075) | -33.3 (28.26)

41. Secondary Outcome: Mean Change From Baseline in Participant Global Assessment of Disease Activity by Smoking Status at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the participant global assessment of disease activity by participant baseline smoking status was calculated at study Month 2, Month 4, and Month 6. The participant global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease. Pack years smoked is defined as the total number of packs smoked per day multiplied by the number of years the participant smoked.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Non-Smoker - Month 2 (n=1963) | -20.7 (24.43)
  Non-Smoker - Month 4 (n=1963) | -27.3 (26.73)
  Non-Smoker - Month 6 (n=1963) | -31.5 (27.99)
  Smoking history >=20 years - Month 2 (n=324) | -21.1 (25.34)
  Smoking history >=20 years - Month 4 (n=324) | -26.2 (27.96)
  Smoking history >=20 years - Month 6 (n=324) | -29.9 (28.05)
  Smoking history <20 years - Month 2 (n=314) | -24.2 (24.92)
  Smoking history <20 years - Month 4 (n=314) | -28.5 (27.04)
  Smoking history <20 years - Month 6 (n=314) | -31.2 (27.73)
  Currently smokes <0.5 packs/day - Month 2 (n=223) | -17.5 (23.82)
  Currently smokes <0.5 packs/day - Month 4 (n=223) | -24.0 (27.76)
  Currently smokes <0.5 pack/day - Month 6 (n=223) | -26.3 (29.99)
  Currently smokes 0.5-1 pack/day - Month 2 (n=397) | -21.3 (24.57)
  Currently smokes 0.5-1 pack/day - Month 4 (n=397) | -24.7 (27.65)
  Currently smokes 0.5-1 pack/day - Month 6 (n=397) | -26.3 (30.57)
  Currently smokes >1 packs/day - Month 2 (n=59) | -21.9 (29.42)
  Currently smokes >1 packs/day - Month 4 (n=59) | -20.7 (31.65)
  Currently smokes >1 packs/day - Month 6 (n=59) | -22.8 (29.35)
  Pack years <7.5 - Month 2 (n=423) | -21.9 (25.21)
  Pack years <7.5 - Month 4 (n=423) | -26.4 (27.80)
  Pack years <7.5 - Month 6 (n=423) | -29.8 (28.76)
  Pack years 7.5 to 20.5 - Month 2 (n=454) | -21.4 (24.97)
  Pack years 7.5 to 20.5 - Month 4 (n=454) | -27.3 (26.86)
  Pack years 7.5 to 20.5 - Month 6 (n=454) | -28.4 (29.04)
  Pack years >20.5 - Month 2 (n=418) | -20.6 (25.00)
  Pack years >20.5 - Month 4 (n=418) | -23.2 (28.82)
  Pack years >20.5 - Month 6 (n=418) | -26.3 (28.89)

42. Secondary Outcome: Mean Change From Baseline in Participant Global Assessment of Disease Activity by Eligibility for Anti-TNF Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the participant global assessment of disease activity by the participant eligibility for anti-TNF treatment was calculated at study Month 2, Month 4, and Month 6. The participant global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Anti-TNF treatment Ineligible - Month 2 (n=106) | -18.9 (21.65)
  Anti-TNF treatment Ineligible - Month 4 (n=106) | -24.7 (24.02)
  Anti-TNF treatment Ineligible - Month 6 (n=106) | -25.8 (27.59)
  Anti-TNF treatment Eligible - Month 2 (n=3174) | -21.0 (24.75)
  Anti-TNF treatment Eligible - Month 4 (n=3174) | -26.7 (27.27)
  Anti-TNF treatment Eligible - Month 6 (n=3174) | -30.3 (28.54)

43. Secondary Outcome: Mean Change From Baseline in Participant Global Assessment of Disease Activity by Participant Baseline Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the participant global assessment of disease activity by the participant baseline expectation of treatment outcome was evaluated at study Month 2, Month 4, and Month 6. The participant global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease. The participant expectation scale was evaluated by questionnaire for a categorical score of 1 (best) to 5 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  <=1.5 - Month 2 (n=1212) | -23.9 (25.79)
  <=1.5 - Month 4 (n=1212) | -29.5 (28.50)
  <=1.5 - Month 6 (n=1212) | -33.9 (28.65)
  >1.5 to 1.86 - Month 2 (n=1009) | -21.3 (24.59)
  >1.5 to 1.86 - Month 4 (n=1009) | -27.0 (27.03)
  >1.5 to 1.86 - Month 6 (n=1009) | -30.3 (28.79)
  >=1.86 - Month 2 (n=1054) | -17.3 (22.83)
  >=1.86 - Month 4 (n=1054) | -22.8 (25.20)
  >=1.86 - Month 6 (n=1054) | -25.6 (27.53)

44. Secondary Outcome: Mean Change From Baseline in Participant Global Assessment of Disease Activity by Physician Experience Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the participant global assessment of disease activity by the treating physician level of experience was evaluated at study Month 2, Month 4, and Month 6. The participant global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease. Physician experience is defined as the number of years the treating physician has experience managing patients with rheumatoid arthritis.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  <=10 years - Month 2 (n=1305) | -21.0 (24.66)
  <=10 years - Month 4 (n=1305) | -26.2 (26.73)
  <=10 years - Month 6 (n=1305) | -29.6 (28.41)
  >10 to 20 years - Month 2 (n=1105) | -20.8 (24.01)
  >10 to 20 years - Month 4 (n=1105) | -27.5 (26.88)
  >10 to 20 years - Month 6 (n=1105) | -31.1 (28.37)
  >20 years - Month 2 (n=850) | -21.3 (25.30)
  >20 years - Month 4 (n=850) | -26.2 (28.21)
  >20 years - Month 6 (n=850) | -29.8 (28.72)

45. Secondary Outcome: mm [Best]Mean Change From Baseline in Participant Global Assessment of Disease Activity by Physician Experience Level With Biologics at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the participant global assessment of disease activity by physician experience level with biologics was evaluated at study Month 2, Month 4, and Month 6. The participant global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease. Physician experience is defined as the number of years the treating physician has experience managing rheumatoid arthritis with biologics.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  0 to 6 years - Month 2 (n=1160) | -21.2 (24.02)
  0 to 6 years - Month 4 (n=1160) | -26.8 (25.74)
  0 to 6 years - Month 6 (n=1160) | -30.4 (27.68)
  6 to 10 years - Month 2 (n=1745) | -20.9 (24.99)
  6 to 10 years - Month 4 (n=1745) | -26.5 (27.81)
  6 to 10 years - Month 6 (n=1745) | -29.8 (29.06)
  >10 years - Month 2 (n=355) | -20.5 (24.60)
  >10 years - Month 4 (n=355) | -27.3 (28.62)
  >10 years - Month 6 (n=355) | -31.2 (28.22)

46. Secondary Outcome: Mean Change From Baseline in Participant Global Assessment of Disease Activity by the Number of Patients Treated by the Physician With Biologics at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the participant global assessment of disease activity by the number of patients treated with biologics by the treating physician was evaluated at study Month 2, Month 4, and Month 6. The participant global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease. The number of patients treated with biologics is defined as the number of patients with rheumatoid arthritis treated by the physician in the last month with biologic agents.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  1-17 patients in prior month - Month 2 (n=1056) | -21.0 (23.25)
  1-17 patients in prior month - Month 4 (n=1056) | -26.3 (25.27)
  1-17 patients in prior month - Month 6 (n=1056) | -31.4 (27.38)
  18-34 patients in prior month - Month 2 (n=1061) | -20.8 (24.98)
  18-34 patients in prior month - Month 4 (n=1061) | -26.7 (27.63)
  18-34 patients in prior month - Month 6 (n=1061) | -28.8 (28.63)
  >=35 patients in prior month - Month 2 (n=1097) | -21.2 (25.38)
  >=35 patients in prior month - Month 4 (n=1097) | -27.0 (28.19)
  >=35 patients in prior month - Month 6 (n=1097) | -30.3 (29.13)

47. Secondary Outcome: Mean Change From Baseline in Participant Global Assessment of Disease Activity by the the Physician Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the participant global assessment of disease activity by the physician's expectation of treatment outcome was evaluated at study Month 2, Month 4, and Month 6. The participant global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease. The physician's expectation of treatment outcome was assessed at the start of Month 4, when physicians were asked to rate their expectations of treatment outcome as: high disease activity, moderate disease activity, low disease activity, or remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  High disease activity - Month 2 (n=40) | -25.1 (25.56)
  High disease activity - Month 4 (n=40) | -22.4 (24.52)
  High disease activity - Month 6 (n=40) | -30.6 (27.95)
  Moderate disease activity - Month 2 (n=325) | -17.3 (24.53)
  Moderate disease activity - Month 4 (n=325) | -23.4 (27.22)
  Moderate disease activity - Month 6 (n=325) | -28.3 (27.88)
  Low disease activity - Month 2 (n=1932) | -21.4 (24.36)
  Low disease activity - Month 4 (n=1932) | -27.3 (27.08)
  Low disease activity - Month 6 (n=1932) | -31.0 (28.16)
  Remission - Month 2 (n=966) | -21.2 (25.13)
  Remission - Month 4 (n=966) | -26.5 (27.25)
  Remission - Month 6 (n=966) | -28.9 (29.27)

48. Secondary Outcome: Mean Change From Baseline in the Erythrocyte Sedimentation Rate (ESR) by Concomitant MTX Dose at Month 2, Month 4, and Month 6
Description: The change from baseline in participant serum ESR was calculated by concomitant MTX dose (low < 10mg/wk, medium >= 10 to < 15 mg/week, and high >=15 mg/week) at study Month 2, Month 4, and Month 6.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mm/h
  Low MTX Dose - Month 2 (n=142) | -9.4 (14.73)
  Low MTX Dose - Month 4 (n=142) | -9.8 (18.98)
  Low MTX Dose - Month 6 (n=142) | -9.2 (21.99)
  Medium MTX Dose - Month 2 (n=526) | -11.2 (17.91)
  Medium MTX Dose - Month 4 (n=526) | -11.5 (21.29)
  Medium MTX Dose - Month 6 (n=526) | -12.8 (22.52)
  High MTX Dose - Month 2 (n=1995) | -9.2 (17.85)
  High MTX Dose - Month 4 (n=1995) | -10.3 (19.03)
  High MTX Dose - Month 6 (n=1995) | -10.9 (20.43)

49. Secondary Outcome: Mean Change From Baseline in ESR by Concomitant DMARD Background Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum ESR by concomitant DMARD background treatment was calculated at study Month 2, Month 4, and Month 6. DMARD Combination 1 = MTX + hydrochloroquine, chloroquine, chloroquine phosphate; Combination 2 = MTX + leflunomide; Combination 3 = MTX + sulfasalazine; Combination 4 = MTX + hydrochloroquine, chloroquine, chloroquine phosphate + sulfasalazine; Combination 5 = leflunomide only.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mm/h
  DMARD Combination 1 - Month 2 (n=1681) | -9.8 (17.03)
  DMARD Combination 1 - Month 4 (n=1681) | -10.9 (18.94)
  DMARD Combination 1 - Month 6 (n=1681) | -11.6 (20.53)
  DMARD Combination 2 - Month 2 (n=433) | -8.1 (19.27)
  DMARD Combination 2 - Month 4 (n=433) | -9.2 (20.60)
  DMARD Combination 2 - Month 6 (n=433) | -10.9 (22.12)
  DMARD Combination 3 - Month 2 (n=216) | -10.0 (20.15)
  DMARD Combination 3 - Month 4 (n=216) | -9.9 (19.25)
  DMARD Combination 3 - Month 6 (n=216) | -9.8 (22.15)
  DMARD Combination 4 - Month 2 (n=150) | -10.3 (15.74)
  DMARD Combination 4 -Month 4 (n=150) | -14.9 (23.30)
  DMARD Combination 4 - Month 6 (n=150) | -11.9 (21.73)
  DMARD Combination 5 - Month 2 (n=106) | -10.0 (18.88)
  DMARD Combination 5 - Month 4 (n=106) | -8.7 (19.13)
  DMARD Combination 5 - Month 6 (n=106) | -9.0 (20.65)
  DMARD Combination 6 - Month 2 (n=303) | -7.6 (17.87)
  DMARD Combination 6 - Month 4 (n=303) | -8.1 (20.40)
  DMARD Combination 6 - Month 6 (n=303) | -8.3 (21.40)

50. Secondary Outcome: Mean Change From Baseline in ESR by Concomitant Corticosteroid Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in serum ESR by participant concomitant corticosteroid use was calculated at study Month 2, Month 4, and Month 6.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mm/h
  Did Not Receive Corticosteroids - Month 2 (n=1202) | -9.3 (16.83)
  Did Not Receive Corticosteroids - Month 4 (n=1202) | -10.4 (18.58)
  Did Not Receive Corticosteroids - Month 6 (n=1202) | -10.7 (20.59)
  Received Corticosteroids - Month 2 (n=2078) | -9.4 (18.28)
  Received Corticosteroids - Month 4 (n=2078) | -10.1 (20.02)
  Received Corticosteroids - Month 6 (n=2078) | -10.7 (21.36)

51. Secondary Outcome: Mean Change From Baseline in ESR by the Number of DMARD Failures at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum ESR by the number of participant DMARD failures was calculated at study Month 2, Month 4, and Month 6.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mm/h
  Failed 1 DMARD - Month 2 (n=1129) | -10.0 (17.77)
  Failed 1 DMARD - Month 4 (n=1129) | -11.5 (20.15)
  Failed 1 DMARD - Month 6 (n=1129) | -12.0 (21.71)
  Failed 2 DMARDs - Month 2 (n=1176) | -9.0 (18.03)
  Failed 2 DMARDs - Month 4 (n=1176) | -9.6 (19.25)
  Failed 2 DMARDs - Month 6 (n=1176) | -10.3 (20.83)
  Failed >=3 DMARDs - Month 2 (n=974) | -9.1 (17.42)
  Failed >=3 DMARDs - Month 4 (n=974) | -9.5 (18.96)
  Failed >=3 DMARDs - Month 6 (n=974) | -9.9 (20.61)

52. Secondary Outcome: Mean Change From Baseline in ESR by Duration of Disease at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the participant serum ESR by the participant duration of disease was calculated at study Month 2, Month 4, and Month 6. The duration of disease is defined as the time since the diagnosis of rheumatoid arthritis.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mm/h
  Duration < 2 years - Month 2 (n=899) | -8.6 (17.77)
  Duration < 2 years - Month 4 (n=899) | -10.6 (20.08)
  Duration < 2 years - Month 6 (n=899) | -11.2 (21.35)
  Duration 2 to <5 years - Month 2 (n=764) | -9.1 (17.97)
  Duration 2 to <5 years - Month 4 (n=764) | -9.5 (19.60)
  Duration 2 to <5 years - Month 6 (n=764) | -9.4 (20.81)
  Duration 5 to 10 years - Month 2 (n=692) | -9.5 (17.69)
  Duration 5 to 10 years - Month 4 (n=692) | -10.2 (18.85)
  Duration 5 to 10 years - Month 6 (n=692) | -11.4 (21.47)
  Duration > 10 years - Month 2 (n=924) | -10.2 (17.63)
  Duration > 10 years - Month 4 (n=924) | -10.5 (19.37)
  Duration > 10 years - Month 6 (n=924) | -10.9 (20.74)

53. Secondary Outcome: Mean Change From Baseline in ESR by Baseline Level of Disease Activity at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum ESR by the participant baseline level of disease activity was calculated at study Month 2, Month 4, and Month 6. DAS28-ESR > 5.1 = high disease activity, DAS28-ESR < 3.2 to < =5.1 = low disease activity, and DAS28-ESR <2.6 = remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mm/h
  DAS28 > 3.2 to <=5.1 - Month 2 (n=698) | -3.3 (11.24)
  DAS28 > 3.2 to <=5.1 - Month 4 (n=698) | -2.2 (13.03)
  DAS28 > 3.2 to <=5.1 - Month 6 (n=698) | -2.2 (13.83)
  DAS28 > 5.1 - Month 2 (n=2572) | -11.1 (18.76)
  DAS28 > 5.1 - Month 4 (n=2572) | -12.4 (20.36)
  DAS28 > 5.1 - Month 6 (n=2572) | -13.1 (22.09)

54. Secondary Outcome: Mean Change From Baseline in ESR by Baseline RF Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum ESR by the participant baseline RF level was calculated at study Month 2, Month 4, and Month 6.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mm/h
  RF <=22 IU/mL - Month 2 (n=1026) | -8.6 (17.12)
  RF <=22 IU/mL - Month 4 (n=1026) | -9.2 (18.36)
  RF <=22 IU/mL - Month 6 (n=1026) | -9.7 (19.73)
  RF >22 to <=146 IU/mL - Month 2 (n=1081) | -9.7 (17.75)
  RF >22 to <=146 IU/mL - Month 4 (n=1081) | -10.3 (19.18)
  RF >22 to <=146 IU/mL - Month 6 (n=1081) | -10.3 (20.90)
  RF >146 IU/mL - Month 2 (n=1127) | -9.8 (18.35)
  RF >146 IU/mL - Month 4 (n=1127) | -11.1 (20.70)
  RF >146 IU/mL - Month 6 (n=1127) | -12.2 (22.41)

55. Secondary Outcome: Mean Change From Baseline in ESR by Baseline Anti-CCP Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in ESR by the participant baseline serum level of anti-CCP was calculated at study Month 2, Month 4, and Month 6.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mm/h
  Anti-CCP <=40 U/mL - Month 2 (n=1038) | -8.6 (16.79)
  Anti-CCP <=40 U/mL - Month 4 (n=1038) | -8.9 (17.67)
  Anti-CCP <=40 U/mL - Month 6 (n=1038) | -9.8 (20.33)
  Anti-CCP >40 to <=380 U/mL - Month 2 (n=1112) | -9.7 (18.17)
  Anti-CCP >40 to <=380 U/mL - Month 4 (n=1112) | -10.7 (20.44)
  Anti-CCP >40 to <=380 U/mL - Month 6 (n=1112) | -11.0 (20.64)
  Anti-CCP >380 U/mL - Month 2 (n=1075) | -9.7 (18.37)
  Anti-CCP >380 U/mL - Month 4 (n=1075) | -11.1 (20.21)
  Anti-CCP >380 U/mL - Month 6 (n=1075) | -11.4 (22.30)

56. Secondary Outcome: Mean Change From Baseline in ESR by Smoking History at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum ESR by participant baseline smoking status was calculated at study Month 2, Month 4, and Month 6. Pack years smoked is defined as the total number of packs smoked per day multiplied by the number of years the participant smoked.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mm/h
  Non-Smoker - Month 2 (n=1963) | -9.7 (18.40)
  Non-Smoker - Month 4 (n=1963) | -10.8 (20.04)
  Non-Smoker - Month 6 (n=1963) | -11.7 (21.57)
  Smoking history >=20 years - Month 2 (n=324) | -10.3 (18.11)
  Smoking history >=20 years - Month 4 (n=324) | -10.6 (19.52)
  Smoking history >=20 years - Month 6 (n=324) | -9.7 (20.95)
  Smoking history <20 years - Month 2 (n=314) | -8.4 (17.55)
  Smoking history <20 years - Month 4 (n=314) | -10.1 (18.24)
  Smoking history <20 years - Month 6 (n=314) | -9.9 (20.03)
  Currently smokes <0.5 packs/day - Month 2 (n=223) | -9.3 (17.51)
  Currently smokes <0.5 packs/day - Month 4 (n=223) | -9.4 (19.35)
  Currently smokes <0.5 pack/day - Month 6 (n=223) | -10.7 (22.22)
  Currently smokes 0.5-1 pack/day - Month 2 (n=397) | -8.0 (14.88)
  Currently smokes 0.5-1 pack/day - Month 4 (n=397) | -8.6 (18.01)
  Currently smokes 0.5-1 pack/day - Month 6 (n=397) | -8.0 (18.68)
  Currently smokes >1 packs/day - Month 2 (n=59) | -6.3 (12.82)
  Currently smokes >1 packs/day - Month 4 (n=59) | -4.8 (16.93)
  Currently smokes >1 packs/day - Month 6 (n=59) | -6.2 (20.00)
  Pack years <7.5 - Month 2 (n=423) | -9.1 (17.40)
  Pack years <7.5 - Month 4 (n=423) | -9.2 (18.24)
  Pack years <7.5 - Month 6 (n=423) | -10.1 (21.17)
  Pack years 7.5 to 20.5 - Month 2 (n=454) | -9.0 (16.61)
  Pack years 7.5 to 20.5 - Month 4 (n=454) | -9.8 (18.60)
  Pack years 7.5 to 20.5 - Month 6 (n=454) | -10.1 (18.73)
  Pack years >20.5 - Month 2 (n=418) | -8.2 (16.42)
  Pack years >20.5 - Month 4 (n=418) | -9.2 (19.44)
  Pack years >20.5 - Month 6 (n=418) | -7.6 (20.91)

57. Secondary Outcome: Mean Change From Baseline in ESR by Eligibility for Anti-TNF Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum ESR by the participant eligibility for anti-TNF treatment was calculated at study Month 2, Month 4, and Month 6.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mm/h
  Anti-TNF treatment Ineligible - Month 2 (n=106) | -5.6 (10.46)
  Anti-TNF treatment Ineligible - Month 4 (n=106) | -5.0 (10.87)
  Anti-TNF treatment Ineligible - Month 6 (n=106) | -4.7 (11.99)
  Anti-TNF treatment Eligible - Month 2 (n=3174) | -9.5 (17.94)
  Anti-TNF treatment Eligible - Month 4 (n=3174) | -10.4 (19.70)
  Anti-TNF treatment Eligible - Month 6 (n=3174) | -10.9 (21.29)

58. Secondary Outcome: Mean Change From Baseline in ESR by Baseline Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum ESR by the participant baseline expectation of treatment outcome was evaluated at study Month 2, Month 4, and Month 6. The participant expectation scale was evaluated by questionnaire for a categorical score of 1 (best) to 5 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mm/h
  <=1.5 - Month 2 (n=1212) | -10.1 (18.15)
  <=1.5 - Month 4 (n=1212) | -11.2 (19.25)
  <=1.5 - Month 6 (n=1212) | -11.4 (21.53)
  >1.5 to 1.86 - Month 2 (n=1009) | -9.6 (18.27)
  >1.5 to 1.86 - Month 4 (n=1009) | -11.3 (20.44)
  >1.5 to 1.86 - Month 6 (n=1009) | -11.8 (21.58)
  >=1.86 - Month 2 (n=1054) | -8.2 (16.79)
  >=1.86 - Month 4 (n=1054) | -8.0 (18.73)
  >=1.86 - Month 6 (n=1054) | -8.9 (19.96)

59. Secondary Outcome: Mean Change From Baseline in ESR by Physician Experience Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum ESR by the treating physician level of experience was evaluated at study Month 2, Month 4, and Month 6. Physician experience is defined as the number of years the treating physician has experience managing patients with rheumatoid arthritis.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mm/h
  <=10 years - Month 2 (n=1305) | -8.6 (17.45)
  <=10 years - Month 4 (n=1305) | -9.4 (19.02)
  <=10 years - Month 6 (n=1305) | -9.9 (20.85)
  >10 to 20 years - Month 2 (n=1105) | -9.6 (18.39)
  >10 to 20 years - Month 4 (n=1105) | -10.7 (20.44)
  >10 to 20 years - Month 6 (n=1105) | -11.8 (22.27)
  >20 years - Month 2 (n=850) | -10.2 (17.49)
  >20 years - Month 4 (n=850) | -10.9 (19.13)
  >20 years - Month 6 (n=850) | -10.6 (19.95)

60. Secondary Outcome: Mean Change From Baseline in ESR by Physician Experience Level With Biologics at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum ESR by physician experience level with biologics was evaluated at study Month 2, Month 4, and Month 6. Physician experience is defined as the number of years the treating physician has experience managing rheumatoid arthritis with biologics.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mm/h
  0 to 6 years - Month 2 (n=1160) | -8.8 (18.10)
  0 to 6 years - Month 4 (n=1160) | -10.7 (19.43)
  0 to 6 years - Month 6 (n=1160) | -9.9 (21.87)
  6 to 10 years - Month 2 (n=1745) | -9.7 (17.65)
  6 to 10 years - Month 4 (n=1745) | -9.6 (19.76)
  6 to 10 years - Month 6 (n=1745) | -11.0 (20.90)
  >10 years - Month 2 (n=355) | -9.7 (17.44)
  >10 years - Month 4 (n=355) | -11.5 (18.81)
  >10 years - Month 6 (n=355) | -12.0 (19.62)

61. Secondary Outcome: Mean Change From Baseline in ESR by the Number of Patients Treated by the Physician With Biologics at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum ESR by the number of patients treated with biologics by the treating physician was evaluated at study Month 2, Month 4, and Month 6. The number of patients treated with biologics is defined as the number of patients with rheumatoid arthritis treated by the physician in the last month with biologic agents.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mm/h
  1-17 patients in prior month - Month 2 (n=1056) | -8.9 (18.47)
  1-17 patients in prior month - Month 4 (n=1056) | -9.2 (19.18)
  1-17 patients in prior month - Month 6 (n=1056) | -9.5 (20.50)
  18-34 patients in prior month - Month 2 (n=1061) | -9.8 (16.19)
  18-34 patients in prior month - Month 4 (n=1061) | -10.9 (19.55)
  18-34 patients in prior month - Month 6 (n=1061) | -11.5 (21.16)
  >=35 patients in prior month - Month 2 (n=1097) | -9.2 (17.96)
  >=35 patients in prior month - Month 4 (n=1097) | -10.0 (19.33)
  >=35 patients in prior month - Month 6 (n=1097) | -10.9 (21.02)

62. Secondary Outcome: Mean Change From Baseline in ESR by the the Physician Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum ESR by the physician's expectation of treatment outcome was evaluated at study Month 2, Month 4, and Month 6. The physician's expectation of treatment outcome was assessed at the start of Month 4, when physicians were asked to rate their expectations of treatment outcome as: high disease activity, moderate disease activity, low disease activity, or remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mm/h
  High disease activity - Month 2 (n=40) | -16.9 (20.16)
  High disease activity - Month 4 (n=40) | -17.0 (23.02)
  High disease activity - Month 6 (n=40) | -13.0 (26.66)
  Moderate disease activity - Month 2 (n=325) | -8.8 (19.09)
  Moderate disease activity - Month 4 (n=325) | -10.1 (20.39)
  Moderate disease activity - Month 6 (n=325) | -11.6 (21.77)
  Low disease activity - Month 2 (n=1932) | -9.3 (17.54)
  Low disease activity - Month 4 (n=1932) | -10.3 (19.45)
  Low disease activity - Month 6 (n=1932) | -10.5 (20.73)
  Remission - Month 2 (n=966) | -9.4 (17.70)
  Remission - Month 4 (n=966) | -10.0 (19.15)
  Remission - Month 6 (n=966) | -10.9 (21.33)

63. Secondary Outcome: Mean Change From Baseline in C-Reactive Protein (CRP) by Concomitant MTX Dose at Month 2, Month 4, and Month 6
Description: The change from baseline in participant serum CRP was calculated by concomitant MTX dose (low < 10mg/wk, medium >= 10 to < 15 mg/week, and high >=15 mg/week) at study Month 2, Month 4, and Month 6.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mg/L
  Low MTX Dose - Month 2 (n=138) | -6.43 (15.483)
  Low MTX Dose - Month 4 (n=138) | -4.97 (19.260)
  Low MTX Dose - Month 6 (n=138) | -6.61 (17.632)
  Medium MTX Dose - Month 2 (n=519) | -7.14 (17.591)
  Medium MTX Dose - Month 4 (n=519) | -6.54 (20.221)
  Medium MTX Dose - Month 6 (n=519) | -5.93 (23.755)
  High MTX Dose - Month 2 (n=1967) | -5.52 (18.452)
  High MTX Dose - Month 4 (n=1967) | -5.46 (18.921)
  High MTX Dose - Month 6 (n=1967) | -5.76 (19.045)

64. Secondary Outcome: Mean Change From Baseline in CRP by Concomitant DMARD Background Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum CRP by concomitant DMARD background treatment was calculated at study Month 2, Month 4, and Month 6. DMARD Combination 1 = MTX + hydrochloroquine, chloroquine, chloroquine phosphate; Combination 2 = MTX + leflunomide; Combination 3 = MTX + sulfasalazine; Combination 4 = MTX + hydrochloroquine, chloroquine, chloroquine phosphate + sulfasalazine; Combination 5 = leflunomide only.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mg/L
  DMARD Combination 1 - Month 2 (n=1662) | -6.02 (16.365)
  DMARD Combination 1 - Month 4 (n=1662) | -5.74 (18.459)
  DMARD Combination 1 - Month 6 (n=1662) | -5.91 (19.101)
  DMARD Combination 2 - Month 2 (n=424) | -6.14 (16.979)
  DMARD Combination 2 - Month 4 (n=424) | -5.07 (21.648)
  DMARD Combination 2 - Month 6 (n=424) | -6.43 (18.324)
  DMARD Combination 3 - Month 2 (n=211) | -2.56 (22.236)
  DMARD Combination 3 - Month 4 (n=211) | -3.32 (19.341)
  DMARD Combination 3 - Month 6 (n=211) | -2.37 (16.441)
  DMARD Combination 4 - Month 2 (n=147) | -7.57 (22.433)
  DMARD Combination 4 -Month 4 (n=147) | -9.61 (22.126)
  DMARD Combination 4 - Month 6 (n=147) | -9.54 (22.444)
  DMARD Combination 5 - Month 2 (n=104) | -4.42 (28.394)
  DMARD Combination 5 - Month 4 (n=104) | -4.49 (16.258)
  DMARD Combination 5 - Month 6 (n=104) | -3.62 (36.080)
  DMARD Combination 6 - Month 2 (n=301) | -3.90 (16.817)
  DMARD Combination 6 - Month 4 (n=301) | -4.70 (17.356)
  DMARD Combination 6 - Month 6 (n=301) | -4.08 (19.620)

65. Secondary Outcome: Mean Change From Baseline in CRP by Concomitant Corticosteroid Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in serum CRP by participant concomitant corticosteroid use was calculated at study Month 2, Month 4, and Month 6.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mg/L
  Did Not Receive Corticosteroids - Month 2 (n=1187) | -5.14 (15.017)
  Did Not Receive Corticosteroids - Month 4 (n=1187) | -4.90 (15.643)
  Did Not Receive Corticosteroids - Month 6 (n=1187) | -5.00 (18.391)
  Received Corticosteroids - Month 2 (n=2048) | -6.04 (19.355)
  Received Corticosteroids - Month 4 (n=2048) | -5.98 (20.850)
  Received Corticosteroids - Month 6 (n=2048) | -6.20 (20.738)

66. Secondary Outcome: Mean Change From Baseline in CRP by the Number of DMARD Failures at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum CRP by the number of participant DMARD failures was calculated at study Month 2, Month 4, and Month 6.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mg/L
  Failed 1 DMARD - Month 2 (n=1118) | -6.38 (18.525)
  Failed 1 DMARD - Month 4 (n=1118) | -6.23 (20.809)
  Failed 1 DMARD - Month 6 (n=1118) | -6.06 (21.514)
  Failed 2 DMARDs - Month 2 (n=1158) | -5.20 (17.550)
  Failed 2 DMARDs - Month 4 (n=1158) | -4.89 (18.155)
  Failed 2 DMARDs - Month 6 (n=1158) | -5.54 (18.247)
  Failed >=3 DMARDs - Month 2 (n=958) | -5.56 (17.533)
  Failed >=3 DMARDs - Month 4 (n=958) | -5.69 (18.158)
  Failed >=3 DMARDs - Month 6 (n=958) | -5.69 (19.959)

67. Secondary Outcome: Mean Change From Baseline in CRP by Duration of Disease at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the participant serum CRP by the participant duration of disease was calculated at study Month 2, Month 4, and Month 6. The duration of disease is defined as the time since the diagnosis of rheumatoid arthritis.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mg/L
  Duration < 2 years - Month 2 (n=885) | -5.84 (18.067)
  Duration < 2 years - Month 4 (n=885) | -5.40 (21.661)
  Duration < 2 years - Month 6 (n=885) | -6.03 (21.956)
  Duration 2 to <5 years - Month 2 (n=756) | -6.42 (20.069)
  Duration 2 to <5 years - Month 4 (n=756) | -6.23 (19.018)
  Duration 2 to <5 years - Month 6 (n=756) | -6.15 (20.592)
  Duration 5 to 10 years - Month 2 (n=681) | -4.73 (15.933)
  Duration 5 to 10 years - Month 4 (n=681) | -4.49 (18.010)
  Duration 5 to 10 years - Month 6 (n=681) | -5.15 (16.892)
  Duration > 10 years - Month 2 (n=912) | -5.73 (17.183)
  Duration > 10 years - Month 4 (n=912) | -6.05 (17.284)
  Duration > 10 years - Month 6 (n=912) | -5.63 (19.402)

68. Secondary Outcome: Mean Change From Baseline in CRP by Baseline Level of Disease Activity at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum CRP by the participant baseline level of disease activity was calculated at study Month 2, Month 4, and Month 6. DAS28-ESR scores of > 3.2 to <=5.1 indicate moderate disease activity and DAS28-ESR scores of > 5.1 indicate high disease activity.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mg/L
  DAS28 > 3.2 to <=5.1 - Month 2 (n=687) | -3.07 (11.053)
  DAS28 > 3.2 to <=5.1 - Month 4 (n=687) | -1.61 (13.582)
  DAS28 > 3.2 to <=5.1 - Month 6 (n=687) | -1.57 (13.418)
  DAS28 > 5.1 - Month 2 (n=2538) | -6.43 (19.287)
  DAS28 > 5.1 - Month 4 (n=2538) | -6.67 (20.241)
  DAS28 > 5.1 - Month 6 (n=2538) | -6.89 (21.215)

69. Secondary Outcome: Mean Change From Baseline in CRP by Baseline RF Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum CRP by the participant baseline RF level was calculated at study Month 2, Month 4, and Month 6.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mg/L
  RF <=22 IU/mL - Month 2 (n=1025) | -5.18 (16.961)
  RF <=22 IU/mL - Month 4 (n=1025) | -4.63 (18.781)
  RF <=22 IU/mL - Month 6 (n=1025) | -5.19 (18.356)
  RF >22 to <=146 IU/mL - Month 2 (n=1079) | -6.12 (15.703)
  RF >22 to <=146 IU/mL - Month 4 (n=1079) | -5.89 (17.219)
  RF >22 to <=146 IU/mL - Month 6 (n=1079) | -5.46 (21.063)
  RF >146 IU/mL - Month 2 (n=1125) | -5.85 (20.488)
  RF >146 IU/mL - Month 4 (n=1125) | -6.21 (21.056)
  RF >146 IU/mL - Month 6 (n=1125) | -6.59 (20.170)

70. Secondary Outcome: Mean Change From Baseline in CRP by Baseline Anti-CCP Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in CRP by the participant baseline serum level of anti-CCP was calculated at study Month 2, Month 4, and Month 6.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mg/L
  Anti-CCP <=40 U/mL - Month 2 (n=1027) | -5.16 (17.703)
  Anti-CCP <=40 U/mL - Month 4 (n=1027) | -4.79 (19.454)
  Anti-CCP <=40 U/mL - Month 6 (n=1027) | -5.03 (18.512)
  Anti-CCP >40 to <=380 U/mL - Month 2 (n=1101) | -5.95 (17.423)
  Anti-CCP >40 to <=380 U/mL - Month 4 (n=1101) | -5.73 (18.955)
  Anti-CCP >40 to <=380 U/mL - Month 6 (n=1101) | -5.60 (18.699)
  Anti-CCP >380 U/mL - Month 2 (n=1070) | -6.00 (18.651)
  Anti-CCP >380 U/mL - Month 4 (n=1070) | -6.22 (19.067)
  Anti-CCP >380 U/mL - Month 6 (n=1070) | -6.60 (22.345)

71. Secondary Outcome: Mean Change From Baseline in CRP by Smoking Status at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum CRP by participant baseline smoking status was calculated at study Month 2, Month 4, and Month 6. Pack years smoked is defined as the total number of packs smoked per day multiplied by the number of years the participant smoked.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mg/L
  Non-Smoker - Month 2 (n=1941) | -6.00 (18.946)
  Non-Smoker - Month 4 (n=1941) | -5.96 (20.052)
  Non-Smoker - Month 6 (n=1941) | -6.27 (21.278)
  Smoking history >=20 years - Month 2 (n=318) | -5.33 (13.490)
  Smoking history >=20 years - Month 4 (n=318) | -4.42 (18.329)
  Smoking history >=20 years - Month 6 (n=318) | -3.70 (16.922)
  Smoking history <20 years - Month 2 (n=312) | -5.88 (19.794)
  Smoking history <20 years - Month 4 (n=312) | -6.50 (17.869)
  Smoking history <20 years - Month 6 (n=312) | -7.38 (19.301)
  Currently smokes <0.5 packs/day - Month 2 (n=218) | -4.28 (16.141)
  Currently smokes <0.5 packs/day - Month 4 (n=218) | -4.85 (18.384)
  Currently smokes <0.5 pack/day - Month 6 (n=218) | -4.72 (15.013)
  Currently smokes 0.5-1 pack/day - Month 2 (n=388) | -5.61 (13.870)
  Currently smokes 0.5-1 pack/day - Month 4 (n=388) | -4.88 (15.045)
  Currently smokes 0.5-1 pack/day - Month 6 (n=388) | -4.57 (18.217)
  Currently smokes >1 packs/day - Month 2 (n=58) | -3.44 (21.229)
  Currently smokes >1 packs/day - Month 4 (n=58) | -1.86 (23.322)
  Currently smokes >1 packs/day - Month 6 (n=58) | -2.76 (19.927)
  Pack years <7.5 - Month 2 (n=418) | -6.13 (18.761)
  Pack years <7.5 - Month 4 (n=418) | -5.91 (18.169)
  Pack years <7.5 - Month 6 (n=418) | -6.75 (18.752)
  Pack years 7.5 to 20.5 - Month 2 (n=450) | -4.73 (13.845)
  Pack years 7.5 to 20.5 - Month 4 (n=450) | -4.63 (16.089)
  Pack years 7.5 to 20.5 - Month 6 (n=450) | -4.60 (15.440)
  Pack years >20.5 - Month 2 (n=405) | -4.92 (15.558)
  Pack years >20.5 - Month 4 (n=405) | -4.40 (18.166)
  Pack years >20.5 - Month 6 (n=405) | -3.48 (18.229)

72. Secondary Outcome: Mean Change From Baseline in CRP by Eligibility for Anti-TNF Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum CRP by the participant eligibility for anti-TNF treatment was calculated at study Month 2, Month 4, and Month 6.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mg/L
  Anti-TNF treatment Ineligible - Month 2 (n=105) | -2.92 (10.633)
  Anti-TNF treatment Ineligible - Month 4 (n=105) | -2.74 (11.237)
  Anti-TNF treatment Ineligible - Month 6 (n=105) | -3.16 (10.453)
  Anti-TNF treatment Eligible - Month 2 (n=3130) | -5.81 (18.078)
  Anti-TNF treatment Eligible - Month 4 (n=3130) | -5.68 (19.314)
  Anti-TNF treatment Eligible - Month 6 (n=3130) | -5.85 (20.146)

73. Secondary Outcome: Mean Change From Baseline in CRP by Participant Baseline Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum CRP by the participant baseline expectation of treatment outcome was evaluated at study Month 2, Month 4, and Month 6. The participant expectation scale was evaluated by questionnaire for a categorical score of 1 (best) to 5 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mg/L
  <=1.5 - Month 2 (n=1201) | -5.83 (15.963)
  <=1.5 - Month 4 (n=1201) | -5.58 (17.902)
  <=1.5 - Month 6 (n=1201) | -5.83 (17.496)
  >1.5 to 1.86 - Month 2 (n=995) | -6.61 (18.586)
  >1.5 to 1.86 - Month 4 (n=995) | -6.66 (21.059)
  >1.5 to 1.86 - Month 6 (n=995) | -6.47 (22.984)
  >=1.86 - Month 2 (n=1034) | -4.69 (19.286)
  >=1.86 - Month 4 (n=1034) | -4.51 (18.487)
  >=1.86 - Month 6 (n=1034) | -5.00 (19.364)

74. Secondary Outcome: Mean Change From Baseline in CRP by Physician Experience Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum CRP by the treating physician level of experience was evaluated at study Month 2, Month 4, and Month 6. Physician experience is defined as the number of years the treating physician has experience managing patients with rheumatoid arthritis.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mg/L
  <=10 years - Month 2 (n=1284) | -5.17 (17.628)
  <=10 years - Month 4 (n=1284) | -5.29 (17.491)
  <=10 years - Month 6 (n=1284) | -5.77 (20.401)
  >10 to 20 years - Month 2 (n=1094) | -5.60 (19.412)
  >10 to 20 years - Month 4 (n=1094) | -5.58 (20.544)
  >10 to 20 years - Month 6 (n=1094) | -5.65 (20.715)
  >20 years - Month 2 (n=837) | -6.71 (16.262)
  >20 years - Month 4 (n=837) | -6.03 (19.794)
  >20 years - Month 6 (n=837) | -5.96 (18.132)

75. Secondary Outcome: Mean Change From Baseline in CRP by Physician Experience Level With Biologics at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum CRP by physician experience level with biologics was evaluated at study Month 2, Month 4, and Month 6. Physician experience is defined as the number of years the treating physician has experience managing rheumatoid arthritis with biologics.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mg/L
  0 to 6 years - Month 2 (n=1147) | -5.40 (16.834)
  0 to 6 years - Month 4 (n=1147) | -5.53 (18.865)
  0 to 6 years - Month 6 (n=1147) | -6.38 (18.656)
  6 to 10 years - Month 2 (n=1717) | -5.95 (18.516)
  6 to 10 years - Month 4 (n=1717) | -5.59 (19.658)
  6 to 10 years - Month 6 (n=1717) | -5.42 (20.802)
  >10 years - Month 2 (n=351) | -5.58 (18.496)
  >10 years - Month 4 (n=351) | -5.68 (17.691)
  >10 years - Month 6 (n=351) | -5.60 (19.623)

76. Secondary Outcome: Mean Change From Baseline in CRP by the Number of Patients Treated by the Physician With Biologics at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum CRP by the number of patients treated with biologics by the treating physician was evaluated at study Month 2, Month 4, and Month 6. The number of patients treated with biologics is defined as the number of patients with rheumatoid arthritis treated by the physician in the last month with biologic agents.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mg/L
  1-17 patients in prior month - Month 2 (n=1043) | -5.61 (17.530)
  1-17 patients in prior month - Month 4 (n=1043) | -5.51 (19.219)
  1-17 patients in prior month - Month 6 (n=1043) | -6.01 (17.911)
  18-34 patients in prior month - Month 2 (n=1049) | -5.31 (18.054)
  18-34 patients in prior month - Month 4 (n=1049) | -5.24 (20.441)
  18-34 patients in prior month - Month 6 (n=1049) | -5.49 (21.234)
  >=35 patients in prior month - Month 2 (n=1077) | -6.18 (18.134)
  >=35 patients in prior month - Month 4 (n=1077) | -5.92 (17.615)
  >=35 patients in prior month - Month 6 (n=1077) | -5.81 (20.194)

77. Secondary Outcome: Mean Change From Baseline in CRP by the the Physician Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The mean change from baseline in participant serum CRP by the physician's expectation of treatment outcome was evaluated at study Month 2, Month 4, and Month 6. The physician's expectation of treatment outcome was assessed at the start of Month 4, when physicians were asked to rate their expectations of treatment outcome as: high disease activity, moderate disease activity, low disease activity, or remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
mg/L
  High disease activity - Month 2 (n=40) | -12.35 (19.948)
  High disease activity - Month 4 (n=40) | -11.02 (23.210)
  High disease activity - Month 6 (n=40) | -11.41 (20.392)
  Moderate disease activity - Month 2 (n=313) | -6.74 (19.737)
  Moderate disease activity - Month 4 (n=313) | -8.72 (20.915)
  Moderate disease activity - Month 6 (n=313) | -8.97 (22.089)
  Low disease activity - Month 2 (n=1906) | -5.82 (19.413)
  Low disease activity - Month 4 (n=1906) | -5.70 (19.519)
  Low disease activity - Month 6 (n=1906) | -5.86 (20.553)
  Remission - Month 2 (n=959) | -4.80 (13.488)
  Remission - Month 4 (n=959) | -4.13 (17.227)
  Remission - Month 6 (n=959) | -4.32 (17.589)

78. Secondary Outcome: Mean Change From Baseline in the Physician Global Assessment of Disease Activity by Concomitant MTX Dose at Month 2, Month 4, and Month 6
Description: The mean change from baseline in physician global assessment of disease activity was calculated by concomitant MTX dose (low < 10mg/wk, medium >= 10 to < 15 mg/week, and high >=15 mg/week) at study Month 2, Month 4, and Month 6. The physician global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Low MTX Dose - Month 2 (n=142) | -24.6 (19.80)
  Low MTX Dose - Month 4 (n=142) | -32.1 (21.50)
  Low MTX Dose - Month 6 (n=142) | -35.8 (22.02)
  Medium MTX Dose - Month 2 (n=523) | -25.9 (21.29)
  Medium MTX Dose - Month 4 (n=523) | -34.4 (21.19)
  Medium MTX Dose - Month 6 (n=523) | -38.2 (22.63)
  High MTX Dose - Month 2 (n=1987) | -24.1 (20.53)
  High MTX Dose - Month 4 (n=1987) | -32.9 (21.47)
  High MTX Dose - Month 6 (n=1987) | -37.3 (22.93)

79. Secondary Outcome: Mean Change From Baseline in the Physician Global Assessment of Disease Activity by Concomitant DMARD Background Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the physician global assessment of disease by concomitant DMARD background treatment was evaluated at Month 2, Month 4, and Month 6. The physician global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease. DMARD Combination 1 = MTX + hydrochloroquine, chloroquine, chloroquine phosphate; Combination 2 = MTX + leflunomide; Combination 3 = MTX + sulfasalazine; Combination 4 = MTX + hydrochloroquine, chloroquine, chloroquine phosphate + sulfasalazine; Combination 5 = leflunomide only.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  DMARD Combination 1 - Month 2 (n=1674) | -24.7 (20.42)
  DMARD Combination 1 - Month 4 (n=1674) | -33.0 (21.63)
  DMARD Combination 1 - Month 6 (n=1674) | -36.5 (23.22)
  DMARD Combination 2 - Month 2 (n=432) | -23.5 (21.44)
  DMARD Combination 2 - Month 4 (n=432) | -33.5 (21.15)
  DMARD Combination 2 - Month 6 (n=432) | -40.5 (21.00)
  DMARD Combination 3 - Month 2 (n=215) | -23.9 (20.91)
  DMARD Combination 3 - Month 4 (n=215) | -31.8 (21.43)
  DMARD Combination 3 - Month 6 (n=215) | -37.1 (22.84)
  DMARD Combination 4 - Month 2 (n=149) | -25.1 (20.53)
  DMARD Combination 4 -Month 4 (n=149) | -34.5 (20.87)
  DMARD Combination 4 - Month 6 (n=149) | -39.7 (22.46)
  DMARD Combination 5 - Month 2 (n=105) | -26.1 (21.63)
  DMARD Combination 5 - Month 4 (n=105) | -33.5 (21.17)
  DMARD Combination 5 - Month 6 (n=105) | -35.7 (22.58)
  DMARD Combination 6 - Month 2 (n=302) | -25.4 (21.24)
  DMARD Combination 6 - Month 4 (n=302) | -33.3 (22.52)
  DMARD Combination 6 - Month 6 (n=302) | -37.3 (23.02)

80. Secondary Outcome: Mean Change From Baseline in the Physician Global Assessment of Disease Activity by Concomitant Corticosteroid Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the physician global assessment of disease activity by participant concomitant corticosteroid use was calculated at study Month 2, Month 4, and Month 6. The physician global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Did Not Receive Corticosteroids - Month 2 (n=1197) | -23.6 (20.09)
  Did Not Receive Corticosteroids - Month 4 (n=1197) | -32.3 (21.55)
  Did Not Receive Corticosteroids - Month 6 (n=1197) | -35.9 (23.12)
  Received Corticosteroids - Month 2 (n=2069) | -25.0 (21.08)
  Received Corticosteroids - Month 4 (n=2069) | -33.3 (21.66)
  Received Corticosteroids - Month 6 (n=2069) | -37.8 (22.77)

81. Secondary Outcome: Mean Change From Baseline in the Physician Global Assessment of Disease Activity Score by the Number of DMARD Failures at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the physician global assessment of disease activity score by the number of participant DMARD failures was calculated at study Month 2, Month 4, and Month 6. The physician global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Failed 1 DMARD - Month 2 (n=1124) | -24.7 (20.96)
  Failed 1 DMARD - Month 4 (n=1124) | -32.8 (22.34)
  Failed 1 DMARD - Month 6 (n=1124) | -36.1 (23.85)
  Failed 2 DMARDs - Month 2 (n=1171) | -24.5 (21.20)
  Failed 2 DMARDs - Month 4 (n=1171) | -32.8 (20.79)
  Failed 2 DMARDs - Month 6 (n=1171) | -37.7 (21.69)
  Failed >=3 DMARDs - Month 2 (n=970) | -24.2 (19.89)
  Failed >=3 DMARDs - Month 4 (n=970) | -33.2 (21.91)
  Failed >=3 DMARDs - Month 6 (n=970) | -37.6 (23.24)

82. Secondary Outcome: Mean Change From Baseline in the Physician Global Assessment of Disease Activity by Duration of Disease at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the physician global assessment of disease activity by the participant duration of disease was calculated at study Month 2, Month 4, and Month 6. The duration of disease is defined as the time since the diagnosis of rheumatoid arthritis. The physician global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Duration < 2 years - Month 2 (n=895) | -23.5 (21.06)
  Duration < 2 years - Month 4 (n=895) | -31.7 (22.44)
  Duration < 2 years - Month 6 (n=895) | -35.3 (23.98)
  Duration 2 to <5 years - Month 2 (n=761) | -25.0 (20.76)
  Duration 2 to <5 years - Month 4 (n=761) | -33.4 (21.79)
  Duration 2 to <5 years - Month 6 (n=761) | -37.5 (22.13)
  Duration 5 to 10 years - Month 2 (n=688) | -23.6 (2128)
  Duration 5 to 10 years - Month 4 (n=688) | -32.4 (21.00)
  Duration 5 to 10 years - Month 6 (n=688) | -36.7 (22.90)
  Duration > 10 years - Month 2 (n=921) | -25.7 (19.92)
  Duration > 10 years - Month 4 (n=921) | -34.2 (21.10)
  Duration > 10 years - Month 6 (n=921) | -38.7 (22.39)

83. Secondary Outcome: Mean Change From Baseline in the Physician Global Assessment of Disease Activity by Baseline Level of Disease Activity at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the physician global assessment of disease activity by the participant baseline level of disease activity was calculated at study Month 2, Month 4, and Month 6. The participant global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  DAS28 > 3.2 to <=5.1 - Month 2 (n=696) | -21.3 (19.24)
  DAS28 > 3.2 to <=5.1 - Month 4 (n=696) | -27.4 (20.01)
  DAS28 > 3.2 to <=5.1 - Month 6 (n=696) | -30.5 (20.35)
  DAS28 > 5.1 - Month 2 (n=2560) | -25.4 (21.00)
  DAS28 > 5.1 - Month 4 (n=2560) | -34.4 (21.81)
  DAS28 > 5.1 - Month 6 (n=2560) | -38.9 (23.24)

84. Secondary Outcome: Mean Change From Baseline in the Physician Global Assessment of Disease Activity by Baseline RF Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the physician global assessment of disease activity by the participant baseline RF level was calculated at study Month 2, Month 4, and Month 6. The physician global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  RF <=22 IU/mL - Month 2 (n=1023) | -21.9 (20.57)
  RF <=22 IU/mL - Month 4 (n=1023) | -29.9 (21.63)
  RF <=22 IU/mL - Month 6 (n=1023) | -34.2 (22.90)
  RF >22 to <=146 IU/mL - Month 2 (n=1077) | -23.9 (20.35)
  RF >22 to <=146 IU/mL - Month 4 (n=1077) | -32.4 (21.51)
  RF >22 to <=146 IU/mL - Month 6 (n=1077) | -36.5 (22.72)
  RF >146 IU/mL - Month 2 (n=1120) | -27.5 (20.91)
  RF >146 IU/mL - Month 4 (n=1120) | -36.3 (21.17)
  RF >146 IU/mL - Month 6 (n=1120) | -40.5 (22.58)

85. Secondary Outcome: Mean Change From Baseline in the Physician Global Assessment of Disease Activity by Baseline Anti-CCP Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the physician global assessment of disease activity by the participant baseline serum level of anti-CCP was calculated at study Month 2, Month 4, and Month 6. The physician global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: The efficacy evaluable population comprised all participants with a baseline DAS28-ESR or at least one post-baseline measurement of DAS28-ESR. n values represent the number of participants at baseline.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Anti-CCP <=40 U/mL - Month 2 (n=1035) | -21.6 (20.82)
  Anti-CCP <=40 U/mL - Month 4 (n=1035) | -30.4 (22.23)
  Anti-CCP <=40 U/mL - Month 6 (n=1035) | -34.6 (23.64)
  Anti-CCP >40 to <=380 U/mL - Month 2 (n=1105) | -24.6 (20.60)
  Anti-CCP >40 to <=380 U/mL - Month 4 (n=1105) | -33.0 (21.29)
  Anti-CCP >40 to <=380 U/mL - Month 6 (n=1105) | -36.7 (22.92)
  Anti-CCP >380 U/mL - Month 2 (n=1071) | -27.1 (20.62)
  Anti-CCP >380 U/mL - Month 4 (n=1071) | -35.2 (21.23)
  Anti-CCP >380 U/mL - Month 6 (n=1071) | -40.2 (21.96)

86. Secondary Outcome: Mean Change From Baseline in the Physician Global Assessment of Disease Activity by Smoking Status at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the physician global assessment of disease activity by participant baseline smoking status was calculated at study Month 2, Month 4, and Month 6. The physician global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease. Pack years smoked is defined as the total number of packs smoked per day multiplied by the number of years the participant smoked.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Non-Smoker - Month 2 (n=1954) | -25.0 (20.86)
  Non-Smoker - Month 4 (n=1954) | -33.9 (21.26)
  Non-Smoker - Month 6 (n=1954) | -38.3 (22.38)
  Smoking history >=20 years - Month 2 (n=323) | -26.5 (19.97)
  Smoking history >=20 years - Month 4 (n=323) | -34.3 (21.45)
  Smoking history >=20 years - Month 6 (n=323) | -38.7 (21.91)
  Smoking history <20 years - Month 2 (n=313) | -25.3 (20.78)
  Smoking history <20 years - Month 4 (n=313) | -33.1 (21.79)
  Smoking history <20 years - Month 6 (n=313) | -37.1 (24.62)
  Currently smokes <0.5 packs/day - Month 2 (n=222) | -22.0 (19.85)
  Currently smokes <0.5 packs/day - Month 4 (n=222) | -31.0 (22.71)
  Currently smokes <0.5 pack/day - Month 6 (n=222) | -34.8 (24.11)
  Currently smokes 0.5-1 pack/day - Month 2 (n=395) | -21.6 (20.33)
  Currently smokes 0.5-1 pack/day - Month 4 (n=395) | -28.6 (22.11)
  Currently smokes 0.5-1 pack/day - Month 6 (n=395) | -31.6 (23.62)
  Currently smokes >1 packs/day - Month 2 (n=59) | -22.7 (24.16)
  Currently smokes >1 packs/day - Month 4 (n=59) | -28.9 (22.61)
  Currently smokes >1 packs/day - Month 6 (n=59) | -34.2 (21.29)
  Pack years <7.5 - Month 2 (n=422) | -24.8 (20.94)
  Pack years <7.5 - Month 4 (n=422) | -32.8 (22.77)
  Pack years <7.5 - Month 6 (n=422) | -36.7 (24.61)
  Pack years 7.5 to 20.5 - Month 2 (n=451) | -23.2 (19.99)
  Pack years 7.5 to 20.5 - Month 4 (n=451) | -31.5 (20.84)
  Pack years 7.5 to 20.5 - Month 6 (n=451) | -34.8 (23.22)
  Pack years >20.5 - Month 2 (n=417) | -23.7 (20.75)
  Pack years >20.5 - Month 4 (n=417) | -30.3 (22.73)
  Pack years >20.5 - Month 6 (n=417) | -34.6 (22.86)

87. Secondary Outcome: Mean Change From Baseline in the Physician Global Assessment of Disease Activity by Eligibility for Anti-TNF Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the physician global assessment of disease activity by the participant eligibility for anti-TNF treatment was calculated at study Month 2, Month 4, and Month 6. The physician global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Anti-TNF treatment Ineligible - Month 2 (n=105) | -22.0 (18.89)
  Anti-TNF treatment Ineligible - Month 4 (n=105) | -27.9 (19.21)
  Anti-TNF treatment Ineligible - Month 6 (n=105) | -31.6 (20.66)
  Anti-TNF treatment Eligible - Month 2 (n=3161) | -24.6 (20.79)
  Anti-TNF treatment Eligible - Month 4 (n=3161) | -33.1 (21.68)
  Anti-TNF treatment Eligible - Month 6 (n=3161) | -37.3 (22.96)

88. Secondary Outcome: Mean Change From Baseline in the Physician Global Assessment of Disease Activity by Participant Baseline Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the physician global assessment of disease activity by the participant baseline expectation of treatment outcome was evaluated at study Month 2, Month 4, and Month 6. The physician global assessment of disease activity was evaluated using a VAS (0mm [best] -100mm [worst]) with increasing scores indicating increased level of disease. The participant expectation scale was evaluated by questionnaire for a categorical score of 1 (best) to 5 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  <=1.5 - Month 2 (n=1208) | -26.4 (21.50)
  <=1.5 - Month 4 (n=1208) | -34.7 (22.21)
  <=1.5 - Month 6 (n=1208) | -39.2 (23.01)
  >1.5 to 1.86 - Month 2 (n=1005) | -25.2 (20.46)
  >1.5 to 1.86 - Month 4 (n=1005) | -34.3 (21.06)
  >1.5 to 1.86 - Month 6 (n=1005) | -38.0 (22.25)
  >=1.86 - Month 2 (n=1049) | -21.6 (19.79)
  >=1.86 - Month 4 (n=1049) | -29.6 (21.11)
  >=1.86 - Month 6 (n=1049) | -33.8 (23.13)

89. Secondary Outcome: Mean Change From Baseline in the Physician Global Assessment of Disease Activity by Physician Experience Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the physician global assessment of disease activity by the treating physician level of experience was evaluated at study Month 2, Month 4, and Month 6. The participant global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease. Physician experience is defined as the number of years the treating physician has experience managing patients with rheumatoid arthritis.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  <=10 years - Month 2 (n=1305) | -23.7 (21.25)
  <=10 years - Month 4 (n=1305) | -33.2 (21.86)
  <=10 years - Month 6 (n=1305) | -37.0 (23.43)
  >10 to 20 years - Month 2 (n=1101) | -25.6 (20.53)
  >10 to 20 years - Month 4 (n=1101) | -33.6 (21.50)
  >10 to 20 years - Month 6 (n=1101) | -38.8 (22.62)
  >20 years - Month 2 (n=846) | -24.5 (20.05)
  >20 years - Month 4 (n=846) | -31.9 (21.41)
  >20 years - Month 6 (n=846) | -35.1 (22.25)

90. Secondary Outcome: Mean Change From Baseline in the Physician Global Assessment of Disease Activity by Physician Experience Level With Biologics at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the physician global assessment of disease activity by physician experience level with biologics was evaluated at study Month 2, Month 4, and Month 6. The physician global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease. Physician experience is defined as the number of years the treating physician has experience managing rheumatoid arthritis with biologics.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  0 to 6 years - Month 2 (n=1159) | -23.5 (20.84)
  0 to 6 years - Month 4 (n=1159) | -32.5 (21.94)
  0 to 6 years - Month 6 (n=1159) | -37.3 (23.13)
  6 to 10 years - Month 2 (n=1740) | -24.9 (20.80)
  6 to 10 years - Month 4 (n=1740) | -33.2 (21.50)
  6 to 10 years - Month 6 (n=1740) | -37.1 (22.86)
  >10 years - Month 2 (n=353) | -26.4 (19.63)
  >10 years - Month 4 (n=353) | -33.3 (21.24)
  >10 years - Month 6 (n=353) | -36.6 (22.29)

91. Secondary Outcome: Mean Change From Baseline in the Physician Global Assessment of Disease Activity by the Number of Patients Treated by the Physician With Biologics at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the physician global assessment of disease activity by the number of patients treated with biologics by the treating physician was evaluated at study Month 2, Month 4, and Month 6. The physician global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease. The number of patients treated with biologics is defined as the number of patients with rheumatoid arthritis treated by the physician in the last month with biologic agents.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Units on a Scale
  1-17 patients in prior month - Month 2 (n=1053) | -23.1 (19.37)
  1-17 patients in prior month - Month 4 (n=1053) | -32.4 (20.04)
  1-17 patients in prior month - Month 6 (n=1053) | -38.3 (21.95)
  18-34 patients in prior month - Month 2 (n=1060) | -25.5 (21.04)
  18-34 patients in prior month - Month 4 (n=1060) | -33.7 (21.96)
  18-34 patients in prior month - Month 6 (n=1060) | -37.0 (23.00)
  >=35 patients in prior month - Month 2 (n=1095) | -25.0 (21.38)
  >=35 patients in prior month - Month 4 (n=1095) | -32.7 (22.79)
  >=35 patients in prior month - Month 6 (n=1095) | -36.0 (23.67)

92. Secondary Outcome: Mean Change From Baseline in the Physician Global Assessment of Disease Activity by the the Physician Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the physician global assessment of disease activity by the baseline physician expectation of treatment outcome was evaluated at study Month 2, Month 4, and Month 6. The physician global assessment of disease activity was evaluated using a VAS (0mm [best] - 100mm [worst]) with increasing scores indicating increased level of disease. The physician's expectation of treatment outcome was assessed at the start of Month 4, when physicians were asked to rate their expectations of treatment outcome as: high disease activity, moderate disease activity, low disease activity, or remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Units on a Scale
  High disease activity - Month 2 (n=39) | -28.5 (18.27)
  High disease activity - Month 4 (n=39) | -37.3 (24.56)
  High disease activity - Month 6 (n=39) | -38.9 (28.37)
  Moderate disease activity - Month 2 (n=325) | -24.1 (20.53)
  Moderate disease activity - Month 4 (n=325) | -32.6 (22.50)
  Moderate disease activity - Month 6 (n=325) | -37.4 (23.94)
  Low disease activity - Month 2 (n=1927) | -24.8 (20.72)
  Low disease activity - Month 4 (n=1927) | -33.6 (21.18)
  Low disease activity - Month 6 (n=1927) | -38.0 (22.40)
  Remission - Month 2 (n=966) | -24.0 (20.84)
  Remission - Month 4 (n=966) | -31.6 (21.96)
  Remission - Month 6 (n=966) | -35.1 (23.21)

93. Secondary Outcome: Mean Change From Baseline in DAS28-ESR Score by Concomitant MTX Dose at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the DAS28-ESR was calculated by concomitant MTX dose (low < 10mg/wk, medium >= 10 to < 15 mg/week, and high >=15 mg/week) at study Month 2, Month 4, and Month 6. The DAS28-ESR measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the ESR. The DAS28-ESR is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-ESR > 5.1 = high disease activity, DAS28-ESR < 3.2 = low disease activity, and DAS28-ESR <2.6 = remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Low MTX Dose - Month 2 (n=142) | -1.40 (1.060)
  Low MTX Dose - Month 4 (n=142) | -1.97 (1.271)
  Low MTX Dose - Month 6 (n=142) | -2.23 (1.358)
  Medium MTX Dose - Month 2 (n=526) | -1.43 (1.037)
  Medium MTX Dose - Month 4 (n=526) | -2.01 (1.252)
  Medium MTX Dose - Month 6 (n=526) | -2.35 (1.400)
  High MTX Dose - Month 2 (n=1995) | -1.42 (1.131)
  High MTX Dose - Month 4 (n=1995) | -2.00 (1.275)
  High MTX Dose - Month 6 (n=1995) | -2.29 (1.376)

94. Secondary Outcome: Mean Change From Baseline in DAS28-ESR Score by Concomitant DMARD Background Treatment at Month 2, Month 4, and Month 6
Description: The DAS28-ESR measures disease burden using patient global health (self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the ESR. The DAS28-ESR is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-ESR > 5.1 = high disease activity, DAS28-ESR < 3.2 = low disease activity, and DAS28-ESR <2.6 = remission. DMARD Combination 1 = MTX + hydrochloroquine, chloroquine, chloroquine phosphate; Combination 2 = MTX + leflunomide; Combination 3 = MTX+sulfasalazine; Combination 4 = MTX + hydrochloroquine, chloroquine, chloroquine phosphate + sulfasalazine; Combination 5 = leflunomide.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  DMARD Combination 1 - Month 2 (n=1681) | -1.44 (1.092)
  DMARD Combination 1 - Month 4 (n=1681) | -2.03 (1.279)
  DMARD Combination 1 - Month 6 (n=1681) | -2.32 (1.386)
  DMARD Combination 2 - Month 2 (n=433) | -1.35 (1.163)
  DMARD Combination 2 - Month 4 (n=433) | -1.94 (1.274)
  DMARD Combination 2 - Month 6 (n=433) | -2.32 (1.329)
  DMARD Combination 3 - Month 2 (n=216) | -1.42 (1.208)
  DMARD Combination 3 - Month 4 (n=216) | -1.85 (1.280)
  DMARD Combination 3 - Month 6 (n=216) | -2.10 (1.441)
  DMARD Combination 4 - Month 2 (n=150) | -1.39 (1.059)
  DMARD Combination 4 -Month 4 (n=150) | -2.12 (1.334)
  DMARD Combination 4 - Month 6 (n=150) | -2.46 (1.493)
  DMARD Combination 5 - Month 2 (n=106) | -1.46 (1.099)
  DMARD Combination 5 - Month 4 (n=106) | -2.09 (1.148)
  DMARD Combination 5 - Month 6 (n=106) | -2.18 (1.329)
  DMARD Combination 6 - Month 2 (n=303) | -1.40 (1.098)
  DMARD Combination 6 - Month 4 (n=303) | -1.90 (1.288)
  DMARD Combination 6 - Month 6 (n=303) | -2.13 (1.352)

95. Secondary Outcome: Mean Change From Baseline in DAS28-ESR by Concomitant Corticosteroid Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the DAS28-ESR by participant concomitant corticosteroid use was calculated at study Month 2, Month 4, and Month 6. The DAS28-ESR measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the ESR. The DAS28-ESR is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-ESR > 5.1 = high disease activity, DAS28-ESR <3.2 = low disease activity, and DAS28-ESR <2.6 = remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Did Not Receive Corticosteroids - Month 2 (n=1202) | -1.41 (1.079)
  Did Not Receive Corticosteroids - Month 4 (n=1202) | -2.00 (1.233)
  Did Not Receive Corticosteroids - Month 6 (n=1202) | -2.30 (1.380)
  Received Corticosteroids - Month 2 (n=2078) | -1.41 (1.123)
  Received Corticosteroids - Month 4 (n=2078) | -1.95 (1.291)
  Received Corticosteroids - Month 6 (n=2078) | -2.24 (1.376)

96. Secondary Outcome: Mean Change From Baseline in DAS28-ESR Score by the Number of DMARD Failures at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the DAS28-ESR score by the number of participant DMARD failures was calculated at study Month 2, Month 4, and Month 6. The DAS28-ESR measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the ESR. The DAS28-ESR is expressed on a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-ESR > 5.1 = high disease activity, DAS28-ESR < 3.2 = low disease activity, and DAS28-ESR <2.6 = remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Failed 1 DMARD - Month 2 (n=1129) | -1.47 (1.142)
  Failed 1 DMARD - Month 4 (n=1129) | -2.05 (1.361)
  Failed 1 DMARD - Month 6 (n=1129) | -2.32 (1.471)
  Failed 2 DMARDs - Month 2 (n=1176) | -1.41 (1.117)
  Failed 2 DMARDs - Month 4 (n=1176) | -1.93 (1.254)
  Failed 2 DMARDs - Month 6 (n=1176) | -2.26 (1.347)
  Failed >=3 DMARDs - Month 2 (n=974) | -1.35 (1.050)
  Failed >=3 DMARDs - Month 4 (n=974) | -1.92 (1.175)
  Failed >=3 DMARDs - Month 6 (n=974) | -2.20 (1.301)

97. Secondary Outcome: Mean Change From Baseline in DAS28-ESR Score by Duration of Disease at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the DAS28-ESR score by the participant duration of disease was calculated at study Month 2, Month 4, and Month 6. The duration of disease is defined as the time since the diagnosis of rheumatoid arthritis. The DAS28-ESR measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the ESR. The DAS28-ESR is expressed on a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-ESR >5.1 = high disease activity, DAS28-ESR <3.2 = low disease activity, and DAS28-ESR <2.6 = remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Duration < 2 years - Month 2 (n=899) | -1.39 (1.172)
  Duration < 2 years - Month 4 (n=899) | -1.97 (1.380)
  Duration < 2 years - Month 6 (n=899) | -2.25 (1.453)
  Duration 2 to <5 years - Month 2 (n=764) | -1.43 (1.100)
  Duration 2 to <5 years - Month 4 (n=764) | -1.97 (1.214)
  Duration 2 to <5 years - Month 6 (n=764) | -2.23 (1.361)
  Duration 5 to 10 years - Month 2 (n=692) | -1.40 (1.069)
  Duration 5 to 10 years - Month 4 (n=692) | -1.97 (1.204)
  Duration 5 to 10 years - Month 6 (n=692) | -2.25 (1.385)
  Duration > 10 years - Month 2 (n=924) | -1.44 (1.076)
  Duration > 10 years - Month 4 (n=924) | -1.97 (1.256)
  Duration > 10 years - Month 6 (n=924) | -2.30 (1.311)

98. Secondary Outcome: Mean Change From Baseline in DAS28-ESR Score by Baseline Level of Disease Activity at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the DAS28-ESR score by the participant baseline level of disease activity was calculated at study Month 2, Month 4, and Month 6. The DAS28-ESR measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the ESR with increasing scores indicating increased level of disease burden. The DAS28-ESR is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). DAS28-ESR > 5.1 = high disease activity, DAS28-ESR < 3.2 to < =5.1 = low disease activity, and DAS28-ESR <2.6 = remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  DAS28 > 3.2 to <=5.1 - Month 2 (n=698) | -1.10 (1.001)
  DAS28 > 3.2 to <=5.1 - Month 4 (n=698) | -1.43 (1.085)
  DAS28 > 3.2 to <=5.1 - Month 6 (n=698) | -1.61 (1.184)
  DAS28 > 5.1 - Month 2 (n=2572) | -1.50 (1.111)
  DAS28 > 5.1 - Month 4 (n=2572) | -2.12 (1.272)
  DAS28 > 5.1 - Month 6 (n=2572) | -2.45 (1.368)

99. Secondary Outcome: Mean Change From Baseline in DAS28-ESR Score by Baseline RF Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the DAS28-ESR by the participant baseline RF level was calculated at study Month 2, Month 4, and Month 6. The DAS28-ESR measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the ESR. Increasing scores indicate increased burden of disease. The DAS28-ESR is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). DAS28-ESR > 5.1 = high disease activity, DAS28-ESR < 3.2 = low disease activity, and DAS28-ESR <2.6 = remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  RF <=22 IU/mL - Month 2 (n=1026) | -1.34 (1.140)
  RF <=22 IU/mL - Month 4 (n=1026) | -1.90 (1.284)
  RF <=22 IU/mL - Month 6 (n=1026) | -2.19 (1.427)
  RF >22 to <=146 IU/mL - Month 2 (n=1081) | -1.41 (1.077)
  RF >22 to <=146 IU/mL - Month 4 (n=1081) | -1.95 (1.249)
  RF >22 to <=146 IU/mL - Month 6 (n=1081) | -2.21 (1.362)
  RF >146 IU/mL - Month 2 (n=1127) | -1.49 (1.106)
  RF >146 IU/mL - Month 4 (n=1127) | -2.06 (1.282)
  RF >146 IU/mL - Month 6 (n=1127) | -2.38 (1.347)

100. Secondary Outcome: Mean Change From Baseline in DAS28-ESR Score by Baseline Anti-CCP Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the DAS28-ESR score by the participant baseline serum level of anti-CCP was calculated at study Month 2, Month 4, and Month 6. The DAS28-ESR measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the ESR. Increasing scores indicate increased burden of disease. The DAS28-ESR is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). DAS28-ESR > 5.1 = high disease activity, DAS28-ESR < 3.2 = low disease activity, and DAS28-ESR <2.6 = remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Anti-CCP <=40 U/mL - Month 2 (n=1038) | -1.30 (1.120)
  Anti-CCP <=40 U/mL - Month 4 (n=1038) | -1.85 (1.277)
  Anti-CCP <=40 U/mL - Month 6 (n=1038) | -2.17 (1.424)
  Anti-CCP >40 to <=380 U/mL - Month 2 (n=1112) | -1.46 (1.071)
  Anti-CCP >40 to <=380 U/mL - Month 4 (n=1112) | -2.04 (1.274)
  Anti-CCP >40 to <=380 U/mL - Month 6 (n=1112) | -2.27 (1.371)
  Anti-CCP >380 U/mL - Month 2 (n=1075) | -1.48 (1.127)
  Anti-CCP >380 U/mL - Month 4 (n=1075) | -2.01 (1.261)
  Anti-CCP >380 U/mL - Month 6 (n=1075) | -2.35 (1.343)

101. Secondary Outcome: Mean Change From Baseline in DAS28-ESR Score by Smoking Status at Month 2, Month 4, and Month 6
Description: The DAS28-ESR measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the ESR. The DAS28-ESR is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-ESR > 5.1 = high disease activity, DAS28-ESR < 3.2 = low disease activity, and DAS28-ESR <2.6 = remission. Pack years smoked is defined as the total number of packs smoked per day multiplied by the number of years the participant smoked.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Non-Smoker - Month 2 (n=1963) | -1.44 (1.111)
  Non-Smoker - Month 4 (n=1963) | -2.04 (1.260)
  Non-Smoker - Month 6 (n=1963) | -2.36 (1.341)
  Smoking history >=20 years - Month 2 (n=324) | -1.44 (1.096)
  Smoking history >=20 years - Month 4 (n=324) | -1.88 (1.227)
  Smoking history >=20 years - Month 6 (n=324) | -2.23 (1.355)
  Smoking history <20 years - Month 2 (n=314) | -1.47 (1.18)
  Smoking history <20 years - Month 4 (n=314) | -1.99 (1.312)
  Smoking history <20 years - Month 6 (n=314) | -2.28 (1.399)
  Currently smokes <0.5 packs/day - Month 2 (n=223) | -1.26 (1.111)
  Currently smokes <0.5 packs/day - Month 4 (n=223) | -1.87 (1.309)
  Currently smokes <0.5 pack/day - Month 6 (n=223) | -2.17 (1.522)
  Currently smokes 0.5-1 pack/day - Month 2 (n=397) | -1.30 (1.032)
  Currently smokes 0.5-1 pack/day - Month 4 (n=397) | -1.76 (1.234)
  Currently smokes 0.5-1 pack/day - Month 6 (n=397) | -1.90 (1.376)
  Currently smokes >1 packs/day - Month 2 (n=59) | -1.31 (1.369)
  Currently smokes >1 packs/day - Month 4 (n=59) | -1.57 (1.465)
  Currently smokes >1 packs/day - Month 6 (n=59) | -1.77 (1.521)
  Pack years <7.5 - Month 2 (n=423) | -1.42 (1.158)
  Pack years <7.5 - Month 4 (n=423) | -1.94 (1.316)
  Pack years <7.5 - Month 6 (n=423) | -2.24 (1.463)
  Pack years 7.5 to 20.5 - Month 2 (n=454) | -1.41 (1.049)
  Pack years 7.5 to 20.5 - Month 4 (n=454) | -1.94 (1.247)
  Pack years 7.5 to 20.5 - Month 6 (n=454) | -2.16 (1.386)
  Pack years >20.5 - Month 2 (n=418) | -1.29 (1.071)
  Pack years >20.5 - Month 4 (n=418) | -1.69 (1.227)
  Pack years >20.5 - Month 6 (n=418) | -1.93 (1.380)

102. Secondary Outcome: Mean Change From Baseline in DAS28-ESR Score by Eligibility for Anti-TNF Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the DAS28-ESR score by the participant eligibility for anti-TNF treatment was calculated at study Month 2, Month 4, and Month 6. The DAS28-ESR measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the ESR. The DAS28-ESR is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-ESR > 5.1 = high disease activity, DAS28-ESR < 3.2 = low disease activity, and DAS28-ESR <2.6 = remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Anti-TNF treatment Ineligible - Month 2 (n=106) | -1.29 (0.881)
  Anti-TNF treatment Ineligible - Month 4 (n=106) | -1.87 (1.051)
  Anti-TNF treatment Ineligible - Month 6 (n=106) | -1.86 (1.117)
  Anti-TNF treatment Eligible - Month 2 (n=3174) | -1.42 (1.114)
  Anti-TNF treatment Eligible - Month 4 (n=3174) | -1.97 (1.277)
  Anti-TNF treatment Eligible - Month 6 (n=3174) | -2.27 (1.383)

103. Secondary Outcome: Mean Change From Baseline in DAS28-ESR Score by Participant Baseline Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the DAS28-ESR score by the participant baseline expectation of treatment outcome was evaluated at study Month 2, Month 4, and Month 6. The DAS28-ESR measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the ESR. The DAS28-ESR is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-ESR > 5.1 = high disease activity, DAS28-ESR < 3.2 = low disease activity, and DAS28-ESR <2.6 = remission. The participant expectation scale was evaluated by questionnaire for a categorical score of 1 (best) to 5 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  <=1.5 - Month 2 (n=1212) | -1.56 (1.132)
  <=1.5 - Month 4 (n=1212) | -2.11 (1.283)
  <=1.5 - Month 6 (n=1212) | -2.43 (1.377)
  >1.5 to 1.86 - Month 2 (n=1009) | -1.40 (1.094)
  >1.5 to 1.86 - Month 4 (n=1009) | -2.01 (1.288)
  >1.5 to 1.86 - Month 6 (n=1009) | -2.28 (1.386)
  >=1.86 - Month 2 (n=1054) | -1.25 (1.063)
  >=1.86 - Month 4 (n=1054) | -1.75 (1.208)
  >=1.86 - Month 6 (n=1054) | -2.04 (1.344)

104. Secondary Outcome: Mean Change From Baseline in DAS28-ESR Score by Physician Experience Level at Month 2, Month 4, and Month 6
Description: The DAS28-ESR measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the ESR. The DAS28-ESR is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-ESR > 5.1 = high disease activity, DAS28-ESR < 3.2 = low disease activity, and DAS28-ESR <2.6 = remission. Physician experience is defined as the number of years the treating physician has experience managing patients with rheumatoid arthritis.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  <=10 years - Month 2 (n=1305) | -1.35 (1.073)
  <=10 years - Month 4 (n=1305) | -1.93 (1.240)
  <=10 years - Month 6 (n=1305) | -2.20 (1.342)
  >10 to 20 years - Month 2 (n=1105) | -1.46 (1.126)
  >10 to 20 years - Month 4 (n=1105) | -2.03 (1.313)
  >10 to 20 years - Month 6 (n=1105) | -2.38 (1.423)
  >20 years - Month 2 (n=850) | -1.45 (1.127)
  >20 years - Month 4 (n=850) | -1.95 (1.261)
  >20 years - Month 6 (n=850) | -2.22 (1.359)

105. Secondary Outcome: Mean Change From Baseline in DAS28-ESR Score by Physician Experience Level With Biologics at Month 2, Month 4, and Month 6
Description: The DAS28-ESR measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the ESR. The DAS28-ESR is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-ESR > 5.1 = high disease activity, DAS28-ESR < 3.2 = low disease activity, and DAS28-ESR <2.6 = remission. Physician experience is defined as the number of years the treating physician has experience managing rheumatoid arthritis with biologics.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  0 to 6 years - Month 2 (n=1160) | -1.36 (1.063)
  0 to 6 years - Month 4 (n=1160) | -1.94 (1.237)
  0 to 6 years - Month 6 (n=1160) | -2.22 (1.359)
  6 to 10 years - Month 2 (n=1745) | -1.44 (1.124)
  6 to 10 years - Month 4 (n=1745) | -1.97 (1.293)
  6 to 10 years - Month 6 (n=1745) | -2.28 (1.385)
  >10 years - Month 2 (n=355) | -1.46 (1.151)
  >10 years - Month 4 (n=355) | -2.05 (1.269)
  >10 years - Month 6 (n=355) | -2.33 (1.389)

106. Secondary Outcome: Mean Change From Baseline in DAS28-ESR Score by the Number of Patients Treated by the Physician With Biologics at Month 2, Month 4, and Month 6
Description: The DAS28-ESR measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the ESR. The DAS28-ESR is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-ESR > 5.1 = high disease activity, DAS28-ESR < 3.2 = low disease activity, and DAS28-ESR <2.6 = remission. The number of patients treated with biologics is defined as the number of patients with rheumatoid arthritis treated by the physician in the last month with biologic agents.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  1-17 patients in prior month - Month 2 (n=1056) | -1.34 (1.034)
  1-17 patients in prior month - Month 4 (n=1056) | -1.89 (1.154)
  1-17 patients in prior month - Month 6 (n=1056) | -2.26 (1.269)
  18-34 patients in prior month - Month 2 (n=1061) | -1.46 (1.095)
  18-34 patients in prior month - Month 4 (n=1061) | -2.01 (1.291)
  18-34 patients in prior month - Month 6 (n=1061) | -2.26 (1.392)
  >=35 patients in prior month - Month 2 (n=1097) | -1.44 (1.177)
  >=35 patients in prior month - Month 4 (n=1097) | -2.00 (1.350)
  >=35 patients in prior month - Month 6 (n=1097) | -2.27 (1.449)

107. Secondary Outcome: Mean Change From Baseline in DAS28-ESR by the the Physician Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The DAS28-ESR measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the ESR. The DAS28-ESR is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-ESR > 5.1 = high disease activity, DAS28-ESR < 3.2 = low disease activity, and DAS28-ESR <2.6 = remission. The physician's expectation of treatment outcome was assessed at the start of Month 4, when physicians were asked to rate their expectations of treatment outcome as: high disease activity, moderate disease activity, low disease activity, or remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  High disease activity - Month 2 (n=40) | -1.84 (1.388)
  High disease activity - Month 4 (n=40) | -2.28 (1.359)
  High disease activity - Month 6 (n=40) | -2.54 (1.638)
  Moderate disease activity - Month 2 (n=325) | -1.24 (1.067)
  Moderate disease activity - Month 4 (n=325) | -1.72 (1.160)
  Moderate disease activity - Month 6 (n=325) | -2.06 (1.339)
  Low disease activity - Month 2 (n=1932) | -1.37 (1.070)
  Low disease activity - Month 4 (n=1932) | -1.95 (1.252)
  Low disease activity - Month 6 (n=1932) | -2.24 (1.361)
  Remission - Month 2 (n=966) | -1.54 (1.161)
  Remission - Month 4 (n=966) | -2.09 (1.322)
  Remission - Month 6 (n=966) | -2.37 (1.400)

108. Secondary Outcome: Mean Change From Baseline in DAS28-CRP Score by Concomitant MTX Dose at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the DAS28-CRP was calculated by concomitant MTX dose (low < 10mg/wk, medium >= 10 to < 15 mg/week, and high >=15 mg/week) at study Month 2, Month 4, and Month 6. The DAS28-CRP measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the CRP. The DAS28-CRP is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-CRP> 5.1 = high disease activity, DAS28-CRP < 3.2 = low disease activity, and DAS28-CRP <2.6 = remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Low MTX Dose - Month 2 (n=138) | -1.34 (1.014)
  Low MTX Dose - Month 4 (n=138) | -1.87 (1.184)
  Low MTX Dose - Month 6 (n=138) | -2.18 (1.266)
  Medium MTX Dose - Month 2 (n=519) | -1.38 (1.011)
  Medium MTX Dose - Month 4 (n=519) | -1.94 (1.178)
  Medium MTX Dose - Month 6 (n=519) | -2.23 (1.339)
  High MTX Dose - Month 2 (n=1967) | -1.34 (1.067)
  High MTX Dose - Month 4 (n=1967) | -1.87 (1.215)
  High MTX Dose - Month 6 (n=1967) | -2.16 (1.286)

109. Secondary Outcome: Mean Change From Baseline in DAS28-CRP Score by Concomitant DMARD Background Treatment at Month 2, Month 4, and Month 6
Description: The DAS28-CRP measures disease burden using patient global health (patient self-assessment), tender joint-counts & swollen joint-counts (up to 28), and the CRP. The DAS28-CRP is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-CRP >5.1 =high disease activity, DAS28-CRP <3.2=low disease activity, and DAS28-CRP <2.6=remission. DMARD Combination 1 = MTX + hydrochloroquine, chloroquine, chloroquine phosphate; Combination 2 = MTX + leflunomide; Combination 3 = MTX + sulfasalazine; Combination 4 = MTX + hydrochloroquine, chloroquine, chloroquine phosphate + sulfasalazine; Combination 5 =leflunomide.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  DMARD Combination 1 - Month 2 (n=1662) | -1.36 (1.032)
  DMARD Combination 1 - Month 4 (n=1662) | -1.90 (1.216)
  DMARD Combination 1 - Month 6 (n=1662) | -2.18 (1.305)
  DMARD Combination 2 - Month 2 (n=424) | -1.32 (1.123)
  DMARD Combination 2 - Month 4 (n=424) | -1.86 (1.252)
  DMARD Combination 2 - Month 6 (n=424) | -2.21 (1.254)
  DMARD Combination 3 - Month 2 (n=211) | -1.31 (1.168)
  DMARD Combination 3 - Month 4 (n=211) | -1.76 (1.203)
  DMARD Combination 3 - Month 6 (n=211) | -1.94 (1.308)
  DMARD Combination 4 - Month 2 (n=147) | -1.33 (1.022)
  DMARD Combination 4 -Month 4 (n=147) | -1.92 (1.153)
  DMARD Combination 4 - Month 6 (n=147) | -2.33 (1.361)
  DMARD Combination 5 - Month 2 (n=104) | -1.39 (1.019)
  DMARD Combination 5 - Month 4 (n=104) | -1.95 (1.127)
  DMARD Combination 5 - Month 6 (n=104) | -2.10 (1.303)
  DMARD Combination 6 - Month 2 (n=301) | -1.35 (1.029)
  DMARD Combination 6 - Month 4 (n=301) | -1.86 (1.216)
  DMARD Combination 6 - Month 6 (n=301) | -2.06 (1.279)

110. Secondary Outcome: Mean Change From Baseline in DAS28-CRP by Concomitant Corticosteroid Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the DAS28-CRP by participant concomitant corticosteroid use was calculated at study Month 2, Month 4, and Month 6. The DAS28-CRP measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the CRP. The DAS28-CRP is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-CRP> 5.1 = high disease activity, DAS28-CRP < 3.2 = low disease activity, and DAS28-CRP <2.6 = remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Did Not Receive Corticosteroids - Month 2 (n=1187) | -1.34 (1.013)
  Did Not Receive Corticosteroids - Month 4 (n=1187) | -1.86 (1.152)
  Did Not Receive Corticosteroids - Month 6 (n=1187) | -2.16 (1.289)
  Received Corticosteroids - Month 2 (n=2048) | -1.35 (1.072)
  Received Corticosteroids - Month 4 (n=2048) | -1.86 (1.237)
  Received Corticosteroids - Month 6 (n=2048) | -2.14 (1.297)

111. Secondary Outcome: Mean Change From Baseline in DAS28-CRP Score by the Number of DMARD Failures at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the DAS28-CRP score by the number of participant DMARD failures was calculated at study Month 2, Month 4, and Month 6. The DAS28-CRP measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the CRP. The DAS28-CRP is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-CRP> 5.1 = high disease activity, DAS28-CRP < 3.2 = low disease activity, and DAS28-CRP <2.6 = remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Failed 1 DMARD - Month 2 (n=1118) | -1.39 (1.082)
  Failed 1 DMARD - Month 4 (n=1118) | -1.91 (1.288)
  Failed 1 DMARD - Month 6 (n=1118) | -2.19 (1.366)
  Failed 2 DMARDs - Month 2 (n=1158) | -1.35 (1.064)
  Failed 2 DMARDs - Month 4 (n=1158) | -1.83 (1.186)
  Failed 2 DMARDs - Month 6 (n=1158) | -2.13 (1.271)
  Failed >=3 DMARDs - Month 2 (n=958) | -1.30 (0.993)
  Failed >=3 DMARDs - Month 4 (n=958) | -1.84 (1.128)
  Failed >=3 DMARDs - Month 6 (n=958) | -2.12 (1.234)

112. Secondary Outcome: Mean Change From Baseline in DAS28-CRP Score by Duration of Disease at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the DAS28-CRP score by the participant duration of disease was calculated at study Month 2, Month 4, and Month 6. The duration of disease is defined as the time since the diagnosis of rheumatoid arthritis. The DAS28-CRP measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the CRP. The DAS28-CRP is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-CRP> 5.1 = high disease activity, DAS28-CRP < 3.2 = low disease activity, and DAS28-CRP <2.6 = remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Duration < 2 years - Month 2 (n=885) | -1.31 (1.113)
  Duration < 2 years - Month 4 (n=885) | -1.82 (1.296)
  Duration < 2 years - Month 6 (n=885) | -2.10 (1.353)
  Duration 2 to <5 years - Month 2 (n=756) | -1.38 (1.042)
  Duration 2 to <5 years - Month 4 (n=756) | -1.90 (1.169)
  Duration 2 to <5 years - Month 6 (n=756) | -2.16 (1.278)
  Duration 5 to 10 years - Month 2 (n=681) | -1.33 (1.022)
  Duration 5 to 10 years - Month 4 (n=681) | -1.87 (1.148)
  Duration 5 to 10 years - Month 6 (n=681) | -2.12 (1.298)
  Duration > 10 years - Month 2 (n=912) | -1.37 (1.016)
  Duration > 10 years - Month 4 (n=912) | -1.87 (1.188)
  Duration > 10 years - Month 6 (n=912) | -2.20 (1.243)

113. Secondary Outcome: Mean Change From Baseline in DAS28-CRP Score by Baseline Level of Disease Activity at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the DAS28-CRP score by the participant baseline level of disease activity was calculated at study Month 2, Month 4, and Month 6. The DAS28-CRP measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the CRP with increasing scores indicating increased burden of disease. The DAS28-CRP is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). DAS28-CRP > 5.1 = high disease activity, DAS28-CRP < 3.2 to < =5.1 = low disease activity, and DAS28-CRP <2.6 = remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  DAS28 > 3.2 to <=5.1 - Month 2 (n=687) | -1.06 (0.931)
  DAS28 > 3.2 to <=5.1 - Month 4 (n=687) | -1.37 (1.025)
  DAS28 > 3.2 to <=5.1 - Month 6 (n=687) | -1.55 (1.088)
  DAS28 > 5.1 - Month 2 (n=2538) | -1.43 (1.063)
  DAS28 > 5.1 - Month 4 (n=2538) | -2.00 (1.216)
  DAS28 > 5.1 - Month 6 (n=2538) | -2.31 (1.296)

114. Secondary Outcome: Mean Change From Baseline in DAS28-CRP Score by Baseline RF Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the DAS28-CRP by the participant baseline RF level was calculated at study Month 2, Month 4, and Month 6. The DAS28-CRP measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the CRP. The DAS28-CRP is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-CRP> 5.1 = high disease activity, DAS28-CRP < 3.2 = low disease activity, and DAS28-CRP <2.6 = remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  RF <=22 IU/mL - Month 2 (n=1025) | -1.23 (1.057)
  RF <=22 IU/mL - Month 4 (n=1025) | -1.75 (1.200)
  RF <=22 IU/mL - Month 6 (n=1025) | -2.02 (1.294)
  RF >22 to <=146 IU/mL - Month 2 (n=1079) | -1.34 (1.017)
  RF >22 to <=146 IU/mL - Month 4 (n=1079) | -1.85 (1.170)
  RF >22 to <=146 IU/mL - Month 6 (n=1079) | -2.12 (1.280)
  RF >146 IU/mL - Month 2 (n=1125) | -1.45 (1.067)
  RF >146 IU/mL - Month 4 (n=1125) | -1.98 (1.238)
  RF >146 IU/mL - Month 6 (n=1125) | -2.29 (1.295)

115. Secondary Outcome: Mean Change From Baseline in DAS28-CRP Score by Baseline Anti-CCP Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the DAS28-CRP score by the participant baseline serum level of anti-CCP was calculated at study Month 2, Month 4, and Month 6. The DAS28-CRP measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the CRP. The DAS28-CRP is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-CRP> 5.1 = high disease activity, DAS28-CRP < 3.2 = low disease activity, and DAS28-CRP <2.6 = remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Anti-CCP <=40 U/mL - Month 2 (n=1027) | -1.22 (1.048)
  Anti-CCP <=40 U/mL - Month 4 (n=1027) | -1.73 (1.200)
  Anti-CCP <=40 U/mL - Month 6 (n=1027) | -2.02 (1.285)
  Anti-CCP >40 to <=380 U/mL - Month 2 (n=1101) | -1.38 (1.022)
  Anti-CCP >40 to <=380 U/mL - Month 4 (n=1101) | -1.92 (1.208)
  Anti-CCP >40 to <=380 U/mL - Month 6 (n=1101) | -2.16 (1.301)
  Anti-CCP >380 U/mL - Month 2 (n=1070) | -1.43 (1.072)
  Anti-CCP >380 U/mL - Month 4 (n=1070) | -1.92 (1.204)
  Anti-CCP >380 U/mL - Month 6 (n=1070) | -2.26 (1.284)

116. Secondary Outcome: Mean Change From Baseline in DAS28-CRP Score by Smoking Status at Month 2, Month 4, and Month 6
Description: The DAS28-CRP measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the CRP. The DAS28-CRP is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-CRP> 5.1 = high disease activity, DAS28-CRP < 3.2 = low disease activity, and DAS28-CRP <2.6 = remission. Pack years smoked is defined as the total number of packs smoked per day multiplied by the number of years the participant smoked.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Non-Smoker - Month 2 (n=1941) | -1.38 (1.054)
  Non-Smoker - Month 4 (n=1941) | -1.94 (1.195)
  Non-Smoker - Month 6 (n=1941) | -2.26 (1.257)
  Smoking history >=20 years - Month 2 (n=318) | -1.36 (1.036)
  Smoking history >=20 years - Month 4 (n=318) | -1.74 (1.190)
  Smoking history >=20 years - Month 6 (n=318) | -2.11 (1.309)
  Smoking history <20 years - Month 2 (n=312) | -1.41 (1.068)
  Smoking history <20 years - Month 4 (n=312) | -1.88 (1.266)
  Smoking history <20 years - Month 6 (n=312) | -2.15 (1.325)
  Currently smokes <0.5 packs/day - Month 2 (n=218) | -1.15 (1.037)
  Currently smokes <0.5 packs/day - Month 4 (n=218) | -1.76 (1.241)
  Currently smokes <0.5 pack/day - Month 6 (n=218) | -2.04 (1.364)
  Currently smokes 0.5-1 pack/day - Month 2 (n=388) | -1.22 (0.984)
  Currently smokes 0.5-1 pack/day - Month 4 (n=388) | -1.63 (1.155)
  Currently smokes 0.5-1 pack/day - Month 6 (n=388) | -1.77 (1.289)
  Currently smokes >1 packs/day - Month 2 (n=58) | -1.33 (1.246)
  Currently smokes >1 packs/day - Month 4 (n=58) | -1.55 (1.248)
  Currently smokes >1 packs/day - Month 6 (n=58) | -1.63 (1.386)
  Pack years <7.5 - Month 2 (n=418) | -1.34 (1.088)
  Pack years <7.5 - Month 4 (n=418) | -1.82 (1.239)
  Pack years <7.5 - Month 6 (n=418) | -2.12 (1.346)
  Pack years 7.5 to 20.5 - Month 2 (n=450) | -1.32 (1.021)
  Pack years 7.5 to 20.5 - Month 4 (n=450) | -1.83 (1.195)
  Pack years 7.5 to 20.5 - Month 6 (n=450) | -2.03 (1.319)
  Pack years >20.5 - Month 2 (n=405) | -1.22 (0.989)
  Pack years >20.5 - Month 4 (n=405) | -1.57 (1.148)
  Pack years >20.5 - Month 6 (n=405) | -1.81 (1.294)

117. Secondary Outcome: Mean Change From Baseline in DAS28-CRP Score by Eligibility for Anti-TNF Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the DAS28-CRP score by the participant eligibility for anti-TNF treatment was calculated at study Month 2, Month 4, and Month 6. The DAS28-CRP measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the CRP. The DAS28-CRP is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-CRP> 5.1 = high disease activity, DAS28-CRP < 3.2 = low disease activity, and DAS28-CRP <2.6 = remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Anti-TNF treatment Ineligible - Month 2 (n=105) | -1.17 (0.867)
  Anti-TNF treatment Ineligible - Month 4 (n=105) | -1.75 (0.982)
  Anti-TNF treatment Ineligible - Month 6 (n=105) | -1.81 (1.086)
  Anti-TNF treatment Eligible - Month 2 (n=3130) | -1.35 (1.056)
  Anti-TNF treatment Eligible - Month 4 (n=3130) | -1.87 (1.213)
  Anti-TNF treatment Eligible - Month 6 (n=3130) | -2.16 (1.299)

118. Secondary Outcome: Mean Change From Baseline in DAS28-CRP Score by Participant Baseline Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the DAS28-CRP score by the participant baseline expectation of treatment outcome was evaluated at study Month 2, Month 4, and Month 6. The DAS28-CRP measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the CRP. The DAS28-CRP is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-CRP> 5.1 = high disease activity, DAS28-CRP < 3.2 = low disease activity, and DAS28-CRP <2.6 = remission. The participant expectation scale was evaluated by questionnaire for a categorical score of 1 (best) to 5 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  <=1.5 - Month 2 (n=1201) | -1.48 (1.081)
  <=1.5 - Month 4 (n=1201) | -1.97 (1.225)
  <=1.5 - Month 6 (n=1201) | -2.31 (1.285)
  >1.5 to 1.86 - Month 2 (n=995) | -1.35 (1.031)
  >1.5 to 1.86 - Month 4 (n=995) | -1.92 (1.212)
  >1.5 to 1.86 - Month 6 (n=995) | -2.16 (1.294)
  >=1.86 - Month 2 (n=1034) | -1.19 (1.006)
  >=1.86 - Month 4 (n=1034) | -1.67 (1.153)
  >=1.86 - Month 6 (n=1034) | -1.94 (1.278)

119. Secondary Outcome: Mean Change From Baseline in DAS28-CRP Score by Physician Experience Level at Month 2, Month 4, and Month 6
Description: The DAS28-CRP measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the CRP. The DAS28-CRP is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-CRP> 5.1 = high disease activity, DAS28-CRP < 3.2 = low disease activity, and DAS28-CRP <2.6 = remission. Physician experience is defined as the number of years the treating physician has experience managing patients with rheumatoid arthritis.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  <=10 years - Month 2 (n=1284) | -1.30 (1.026)
  <=10 years - Month 4 (n=1284) | -1.83 (1.171)
  <=10 years - Month 6 (n=1284) | -2.12 (1.274)
  >10 to 20 years - Month 2 (n=1094) | -1.39 (1.051)
  >10 to 20 years - Month 4 (n=1094) | -1.93 (1.242)
  >10 to 20 years - Month 6 (n=1094) | -2.23 (1.305)
  >20 years - Month 2 (n=837) | -1.36 (1.082)
  >20 years - Month 4 (n=837) | -1.83 (1.208)
  >20 years - Month 6 (n=837) | -2.09 (1.301)

120. Secondary Outcome: Mean Change From Baseline in DAS28-CRP Score by Physician Experience Level With Biologics at Month 2, Month 4, and Month 6
Description: The DAS28-CRP measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the CRP. The DAS28-CRP is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-CRP> 5.1 = high disease activity, DAS28-CRP < 3.2 = low disease activity, and DAS28-CRP <2.6 = remission. Physician experience is defined as the number of years the treating physician has experience managing rheumatoid arthritis with biologics.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  0 to 6 years - Month 2 (n=1147) | -1.31 (1.028)
  0 to 6 years - Month 4 (n=1147) | -1.83 (1.179)
  0 to 6 years - Month 6 (n=1147) | -2.16 (1.281)
  6 to 10 years - Month 2 (n=1717) | -1.37 (1.047)
  6 to 10 years - Month 4 (n=1717) | -1.87 (1.220)
  6 to 10 years - Month 6 (n=1717) | -2.14 (1.292)
  >10 years - Month 2 (n=351) | -1.40 (1.126)
  >10 years - Month 4 (n=351) | -1.93 (1.225)
  >10 years - Month 6 (n=351) | -2.16 (1.337)

121. Secondary Outcome: Mean Change From Baseline in DAS28-CRP Score by the Number of Patients Treated by the Physician With Biologics at Month 2, Month 4, and Month 6
Description: The DAS28-CRP measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the CRP. The DAS28-CRP is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-CRP> 5.1 = high disease activity, DAS28-CRP < 3.2 = low disease activity, and DAS28-CRP <2.6 = remission. The number of patients treated with biologics is defined as the number of patients with rheumatoid arthritis treated by the physician in the last month with biologic agents.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Units on a Scale
  1-17 patients in prior month - Month 2 (n=1043) | -1.31 (1.001)
  1-17 patients in prior month - Month 4 (n=1043) | -1.81 (1.111)
  1-17 patients in prior month - Month 6 (n=1043) | -2.21 (1.228)
  18-34 patients in prior month - Month 2 (n=1049) | -1.36 (1.040)
  18-34 patients in prior month - Month 4 (n=1049) | -1.88 (1.228)
  18-34 patients in prior month - Month 6 (n=1049) | -2.13 (1.297)
  >=35 patients in prior month - Month 2 (n=1077) | -1.38 (1.100)
  >=35 patients in prior month - Month 4 (n=1077) | -1.90 (1.269)
  >=35 patients in prior month - Month 6 (n=1077) | -2.11 (1.339)

122. Secondary Outcome: Mean Change From Baseline in DAS28-CRP by the the Physician Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The DAS28-CRP measures disease burden using patient global health (patient self-assessment), tender joint-counts and swollen joint-counts (up to 28), and the CRP. The DAS28-CRP is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst). Increasing scores indicate increased burden of disease with DAS28-CRP> 5.1 = high disease activity, DAS28-CRP < 3.2 = low disease activity, and DAS28-CRP <2.6 = remission. The physician's expectation of treatment outcome was assessed at the start of Month 4, when physicians were asked to rate their expectations of treatment outcome as: high disease activity, moderate disease activity, low disease activity, or remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  High disease activity - Month 2 (n=40) | -1.68 (1.084)
  High disease activity - Month 4 (n=40) | -2.10 (1.190)
  High disease activity - Month 6 (n=40) | -2.57 (1.485)
  Moderate disease activity - Month 2 (n=313) | -1.19 (0.992)
  Moderate disease activity - Month 4 (n=313) | -1.67 (1.104)
  Moderate disease activity - Month 6 (n=313) | -1.96 (1.265)
  Low disease activity - Month 2 (n=1906) | -1.32 (1.037)
  Low disease activity - Month 4 (n=1906) | -1.85 (1.207)
  Low disease activity - Month 6 (n=1906) | -2.14 (1.300)
  Remission - Month 2 (n=959) | -1.44 (1.083)
  Remission - Month 4 (n=959) | -1.94 (1.224)
  Remission - Month 6 (n=959) | -2.20 (1.271)

123. Secondary Outcome: Mean Change From Baseline in the Simplified Disease Activity Index (SDAI) Score by Concomitant MTX Dose at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the SDAI was calculated by concomitant MTX dose (low < 10mg/wk, medium >= 10 to < 15 mg/week, and high >=15 mg/week) at study Month 2, Month 4, and Month 6. The SDAI is the numerical sum of five outcome parameters: tender and swollen joint count (based on a 28-joint assessment), patient and physician global assessment of disease activity (VAS 0cm [best] - 10cm [worst]) and level of C-reactive protein (mg/dL, normal <1 mg/dL) with increasing scores indicating increased level of disease. The SDAI is expressed as a score on a scale with the minimum score=0 (best) to maximum score=86 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Low MTX Dose - Month 2 (n=138) | -15.55 (11.605)
  Low MTX Dose - Month 4 (n=138) | -20.69 (13.346)
  Low MTX Dose - Month 6 (n=138) | -23.81 (14.063)
  Medium MTX Dose - Month 2 (n=516) | -15.74 (11.579)
  Medium MTX Dose - Month 4 (n=516) | -21.38 (12.872)
  Medium MTX Dose - Month 6 (n=516) | -24.01 (13.992)
  High MTX Dose - Month 2 (n=1959) | -14.99 (11.920)
  High MTX Dose - Month 4 (n=1959) | -20.52 (13.061)
  High MTX Dose - Month 6 (n=1959) | -23.00 (13.743)

124. Secondary Outcome: Mean Change From Baseline in SDAI Score by Concomitant DMARD Background Treatment at Month 2, Month 4, and Month 6
Description: The SDAI is the numerical sum of 5 outcome parameters: tender and swollen joint count (28-joint assessment), patient and physician global assessment of disease activity (VAS 0cm [best] - 10 cm [worst]) and level of C-reactive protein (mg/dL, normal <1 mg/dL) with increasing scores indicating increased level of disease. The SDAI is expressed as a score on a scale with the minimum score=0 (best) to maximum score=86 (worst). DMARD Combination 1 = MTX + hydrochloroquine, chloroquine, chloroquine phosphate; Combination 2 = MTX + leflunomide; Combination 3 = MTX + sulfasalazine; Combination 4 = MTX + hydrochloroquine, chloroquine, chloroquine phosphate + sulfasalazine; Combination 5 = leflunomide.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  DMARD Combination 1 - Month 2 (n=1655) | -15.22 (11.434)
  DMARD Combination 1 - Month 4 (n=1655) | -20.59 (12.977)
  DMARD Combination 1 - Month 6 (n=1655) | -23.07 (13.766)
  DMARD Combination 2 - Month 2 (n=423) | -15.16 (12.811)
  DMARD Combination 2 - Month 4 (n=423) | -21.02 (13.780)
  DMARD Combination 2 - Month 6 (n=423) | -24.31 (13.540)
  DMARD Combination 3 - Month 2 (n=210) | -14.64 (13.206)
  DMARD Combination 3 - Month 4 (n=210) | -19.84 (13.763)
  DMARD Combination 3 - Month 6 (n=210) | -21.41 (14.685)
  DMARD Combination 4 - Month 2 (n=146) | -14.86 (11.590)
  DMARD Combination 4 -Month 4 (n=146) | -21.52 (12.601)
  DMARD Combination 4 - Month 6 (n=146) | -24.45 (14.879)
  DMARD Combination 5 - Month 2 (n=103) | -15.63 (11.838)
  DMARD Combination 5 - Month 4 (n=103) | -20.71 (11.925)
  DMARD Combination 5 - Month 6 (n=103) | -21.67 (13.876)
  DMARD Combination 6 - Month 2 (n=300) | -14.11 (11.443)
  DMARD Combination 6 - Month 4 (n=300) | -19.70 (12.639)
  DMARD Combination 6 - Month 6 (n=300) | -21.41 (13.670)

125. Secondary Outcome: Mean Change From Baseline in SDAI by Concomitant Corticosteroid Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the SDAI by participant concomitant corticosteroid use was calculated at study Month 2, Month 4, and Month 6. The SDAI is the numerical sum of five outcome parameters: tender and swollen joint count (based on a 28-joint assessment), patient and physician global assessment of disease activity (VAS 0 cm [best] - 10 cm [worst]) and level of C-reactive protein (mg/dL, normal <1 mg/dL) with increasing scores indicating increased level of disease. The SDAI is expressed as a score on a scale with the minimum score=0 (best) to maximum score=86 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Did Not Receive Corticosteroids - Month 2 (n=1182) | -14.86 (11.130)
  Did Not Receive Corticosteroids - Month 4 (n=1182) | -20.20 (12.452)
  Did Not Receive Corticosteroids - Month 6 (n=1182) | -22.50 (13.513)
  Received Corticosteroids - Month 2 (n=2039) | -15.12 (12.102)
  Received Corticosteroids - Month 4 (n=2039) | -20.54 (13.367)
  Received Corticosteroids - Month 6 (n=2039) | -23.12 (13.962)

126. Secondary Outcome: Mean Change From Baseline in SDAI by the Number of DMARD Failures at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the SDAI by the number of participant DMARD failures was calculated at study Month 2, Month 4, and Month 6. The SDAI is the numerical sum of five outcome parameters: tender and swollen joint count (based on a 28-joint assessment), patient and physician global assessment of disease activity (VAS 0cm [best] - 10 cm [worst]) and level of C-reactive protein (mg/dL, normal <1 mg/dL) with increasing scores indicating increased level of disease. The SDAI is expressed as a score on a scale with the minimum score=0 (best) to maximum score=86 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Failed 1 DMARD - Month 2 (n=1113) | -15.69 (11.955)
  Failed 1 DMARD - Month 4 (n=1113) | -20.82 (13.873)
  Failed 1 DMARD - Month 6 (n=1113) | -23.31 (14.472)
  Failed 2 DMARDs - Month 2 (n=1153) | -14.97 (11.902)
  Failed 2 DMARDs - Month 4 (n=1153) | -20.26 (12.712)
  Failed 2 DMARDs - Month 6 (n=1153) | -22.74 (13.451)
  Failed >=3 DMARDs - Month 2 (n=954) | -14.33 (11.303)
  Failed >=3 DMARDs - Month 4 (n=954) | -20.12 (12.421)
  Failed >=3 DMARDs - Month 6 (n=954) | -22.60 (13.430)

127. Secondary Outcome: Mean Change From Baseline in SDAI by Duration of Disease at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the SDAI by the participant duration of disease was calculated at study Month 2, Month 4, and Month 6. The duration of disease is defined as the time since the diagnosis of rheumatoid arthritis. The SDAI is the numerical sum of five outcome parameters: tender and swollen joint count (based on a 28-joint assessment), patient and physician global assessment of disease activity (VAS 0cm [best] - 10 cm [worst]) and level of C-reactive protein (mg/dL, normal <1 mg/dL) with increasing scores indicating increased level of disease. The SDAI is expressed as a score on a scale with the minimum score=0 (best) to maximum score=86 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Duration < 2 years - Month 2 (n=881) | -14.62 (12.465)
  Duration < 2 years - Month 4 (n=881) | -19.74 (13.904)
  Duration < 2 years - Month 6 (n=881) | -22.04 (14.136)
  Duration 2 to <5 years - Month 2 (n=753) | -15.37 (11.745)
  Duration 2 to <5 years - Month 4 (n=753) | -20.84 (12.672)
  Duration 2 to <5 years - Month 6 (n=753) | -23.12 (13.619)
  Duration 5 to 10 years - Month 2 (n=677) | -14.75 (11.368)
  Duration 5 to 10 years - Month 4 (n=677) | -20.50 (12.587)
  Duration 5 to 10 years - Month 6 (n=677) | -22.63 (13.893)
  Duration > 10 years - Month 2 (n=909) | -15.35 (11.331)
  Duration > 10 years - Month 4 (n=909) | -20.65 (12.804)
  Duration > 10 years - Month 6 (n=909) | -23.71 (13.516)

128. Secondary Outcome: Mean Change From Baseline in SDAI by Baseline Level of Disease Activity at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the SDAI by the participant baseline level of disease activity was calculated at study Month 2, Month 4, and Month 6. The SDAI is the numerical sum of five outcome parameters: tender and swollen joint count (based on a 28-joint assessment), patient and physician global assessment of disease activity (VAS 0cm [best] - 10 cm [worst]) and level of C-reactive protein (mg/dL, normal <1 mg/dL) with increasing scores indicating increased level of disease with increasing scores indicating increased burden of disease. DAS28-ESR > 5.1 = high disease activity, DAS28-ESR < 3.2 to < =5.1 = low disease activity, and DAS28-ESR <2.6 = remission. The SDAI is expressed as a score on a scale with the minimum score=0 (best) to maximum score=86 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  DAS28 > 3.2 to <=5.1 - Month 2 (n=685) | -9.34 (8.351)
  DAS28 > 3.2 to <=5.1 - Month 4 (n=685) | -12.20 (8.638)
  DAS28 > 3.2 to <=5.1 - Month 6 (n=685) | -13.42 (8.997)
  DAS28 > 5.1 - Month 2 (n=2526) | -16.61 (12.035)
  DAS28 > 5.1 - Month 4 (n=2526) | -22.66 (13.121)
  DAS28 > 5.1 - Month 6 (n=2526) | -25.48 (13.745)

129. Secondary Outcome: Mean Change From Baseline in SDAI by Baseline RF Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the SDAI by the participant baseline RF level was calculated at study Month 2, Month 4, and Month 6. The SDAI is the numerical sum of 5 outcome parameters: tender and swollen joint count (28-joint assessment), patient and physician global assessment of disease activity (VAS 0cm [best] - 10 cm [worst]) and level of C-reactive protein (mg/dL, normal <1 mg/dL) with increasing scores indicating increased level of disease. The SDAI is expressed as a score on a scale with the minimum score=0 (best) to maximum score=86 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  RF <=22 IU/mL - Month 2 (n=1022) | -13.31 (11.369)
  RF <=22 IU/mL - Month 4 (n=1022) | -18.68 (12.690)
  RF <=22 IU/mL - Month 6 (n=1022) | -21.03 (13.335)
  RF >22 to <=146 IU/mL - Month 2 (n=1075) | -14.73 (11.288)
  RF >22 to <=146 IU/mL - Month 4 (n=1075) | -19.89 (12.479)
  RF >22 to <=146 IU/mL - Month 6 (n=1075) | -22.09 (13.315)
  RF >146 IU/mL - Month 2 (n=1118) | -16.88 (12.288)
  RF >146 IU/mL - Month 4 (n=1118) | -22.53 (13.618)
  RF >146 IU/mL - Month 6 (n=1118) | -25.38 (14.328)

130. Secondary Outcome: Mean Change From Baseline in SDAI by Baseline Anti-CCP Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the SDAI by the participant baseline serum level of anti-CCP was calculated at study Month 2, Month 4, and Month 6. The SDAI is the numerical sum of 5 outcome parameters: tender and swollen joint count (28-joint assessment), patient and physician global assessment of disease activity (VAS 0cm [best] - 10 cm [worst]) and level of C-reactive protein (mg/dL, normal <1 mg/dL) with increasing scores indicating increased level of disease. The SDAI is expressed as a score on a scale with the minimum score=0 (best) to maximum score=86 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Anti-CCP <=40 U/mL - Month 2 (n=1024) | -13.40 (11.370)
  Anti-CCP <=40 U/mL - Month 4 (n=1024) | -18.92 (12.860)
  Anti-CCP <=40 U/mL - Month 6 (n=1024) | -21.41 (13.526)
  Anti-CCP >40 to <=380 U/mL - Month 2 (n=1094) | -15.39 (11.601)
  Anti-CCP >40 to <=380 U/mL - Month 4 (n=1094) | -21.01 (12.787)
  Anti-CCP >40 to <=380 U/mL - Month 6 (n=1094) | -22.89 (13.718)
  Anti-CCP >380 U/mL - Month 2 (n=1066) | -16.23 (12.156)
  Anti-CCP >380 U/mL - Month 4 (n=1066) | -21.23 (13.436)
  Anti-CCP >380 U/mL - Month 6 (n=1066) | -24.38 (14.046)

131. Secondary Outcome: Mean Change From Baseline in SDAI by Smoking Status at Month 2, Month 4, and Month 6
Description: The SDAI is the numerical sum of 5 outcome parameters: tender and swollen joint count (28-joint assessment), patient and physician global assessment of disease activity (VAS 0cm [best] - 10 cm [worst]) and level of C-reactive protein (mg/dL, normal <1 mg/dL) with increasing scores indicating increased level of disease. Pack years smoked is defined as the total number of packs smoked per day multiplied by the number of years the participant smoked. The SDAI is expressed as a score on a scale with the minimum score=0 (best) to maximum score=86 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Non-Smoker - Month 2 (n=1932) | -15.64 (11.959)
  Non-Smoker - Month 4 (n=1932) | -21.45 (13.082)
  Non-Smoker - Month 6 (n=1932) | -24.25 (13.565)
  Smoking history >=20 years - Month 2 (n=317) | -15.10 (11.260)
  Smoking history >=20 years - Month 4 (n=317) | -19.34 (13.177)
  Smoking history >=20 years - Month 6 (n=317) | -22.54 (14.104)
  Smoking history <20 years - Month 2 (n=311) | -15.16 (11.477)
  Smoking history <20 years - Month 4 (n=311) | -19.81 (12.777)
  Smoking history <20 years - Month 6 (n=311) | -22.09 (13.648)
  Currently smokes <0.5 packs/day - Month 2 (n=217) | -13.29 (11.523)
  Currently smokes <0.5 packs/day - Month 4 (n=217) | -19.75 (12.965)
  Currently smokes <0.5 pack/day - Month 6 (n=217) | -21.63 (13.986)
  Currently smokes 0.5-1 pack/day - Month 2 (n=386) | -12.85 (10.766)
  Currently smokes 0.5-1 pack/day - Month 4 (n=386) | -17.31 (12.300)
  Currently smokes 0.5-1 pack/day - Month 6 (n=386) | -18.53 (13.500)
  Currently smokes >1 packs/day - Month 2 (n=58) | -14.23 (14.048)
  Currently smokes >1 packs/day - Month 4 (n=58) | -17.48 (13.194)
  Currently smokes >1 packs/day - Month 6 (n=58) | -17.91 (14.453)
  Pack years <7.5 - Month 2 (n=417) | -15.03 (11.772)
  Pack years <7.5 - Month 4 (n=417) | -20.22 (13.138)
  Pack years <7.5 - Month 6 (n=417) | -22.30 (14.299)
  Pack years 7.5 to 20.5 - Month 2 (n=447) | -14.06 (11.024)
  Pack years 7.5 to 20.5 - Month 4 (n=447) | -19.43 (12.462)
  Pack years 7.5 to 20.5 - Month 6 (n=447) | -20.97 (13.912)
  Pack years >20.5 - Month 2 (n=404) | -13.27 (10.943)
  Pack years >20.5 - Month 4 (n=404) | -17.00 (12.278)
  Pack years >20.5 - Month 6 (n=404) | -19.27 (13.313)

132. Secondary Outcome: Mean Change From Baseline in SDAI by Eligibility for Anti-TNF Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the SDAI by the participant eligibility for anti-TNF treatment was calculated at study Month 2, Month 4, and Month 6. The SDAI is the numerical sum of 5 outcome parameters: tender and swollen joint count (28-joint assessment), patient and physician global assessment of disease activity (VAS 0cm [best] - 10 cm [worst]) and level of C-reactive protein (mg/dL, normal <1 mg/dL) with increasing scores indicating increased level of disease. The SDAI is expressed as a score on a scale with the minimum score=0 (best) to maximum score=86 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Anti-TNF treatment Ineligible - Month 2 (n=104) | -12.10 (9.033)
  Anti-TNF treatment Ineligible - Month 4 (n=104) | -17.08 (10.679)
  Anti-TNF treatment Ineligible - Month 6 (n=104) | -17.50 (11.278)
  Anti-TNF treatment Eligible- Month 2 (n=3117) | -15.12 (11.823)
  Anti-TNF treatment Eligible - Month 4 (n=3117) | -20.52 (13.094)
  Anti-TNF treatment Eligible - Month 6 (n=3117) | -23.07 (13.841)

133. Secondary Outcome: Mean Change From Baseline in SDAI by Participant Baseline Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the SDAI by the participant baseline expectation of treatment outcome was evaluated at study Month 2, Month 4, and Month 6. The SDAI is the numerical sum of 5 outcome parameters: tender and swollen joint count (28-joint assessment), patient and physician global assessment of disease activity (VAS 0cm [best] - 10 cm [worst]) and level of C-reactive protein (mg/dL, normal <1 mg/dL) with increasing scores indicating increased level of disease. The SDAI is expressed as a score on a scale with the minimum score=0 (best) to maximum score=86 (worst). The participant expectation scale was evaluated by questionnaire for a categorical score of 1 (best) to 5 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  <=1.5 - Month 2 (n=1197) | -16.51 (12.063)
  <=1.5 - Month 4 (n=1197) | -21.74 (13.182)
  <=1.5 - Month 6 (n=1197) | -24.42 (13.894)
  >1.5 to 1.86 - Month 2 (n=991) | -15.24 (11.600)
  >1.5 to 1.86 - Month 4 (n=991) | -21.04 (13.244)
  >1.5 to 1.86 - Month 6 (n=991) | -23.20 (13.816)
  >=1.86 - Month 2 (n=1029) | -13.09 (11.276)
  >=1.86 - Month 4 (n=1029) | -18.24 (12.411)
  >=1.86 - Month 6 (n=1029) | -20.76 (13.431)

134. Secondary Outcome: Mean Change From Baseline in SDAI by Physician Experience Level at Month 2, Month 4, and Month 6
Description: The SDAI is the numerical sum of 5 outcome parameters: tender and swollen joint count (28-joint assessment), patient and physician global assessment of disease activity (VAS 0cm [best] - 10 cm [worst]) and level of C-reactive protein (mg/dL, normal <1 mg/dL) with increasing scores indicating increased level of disease. The SDAI is expressed as a score on a scale with the minimum score=0 (best) to maximum score=86 (worst). Physician experience is defined as the number of years the treating physician has experience managing patients with rheumatoid arthritis.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  <=10 years - Month 2 (n=1284) | -14.49 (11.734)
  <=10 years - Month 4 (n=1284) | -20.20 (12.818)
  <=10 years - Month 6 (n=1284) | -22.60 (13.587)
  >10 to 20 years - Month 2 (n=1090) | -15.62 (11.857)
  >10 to 20 years - Month 4 (n=1090) | -20.95 (13.465)
  >10 to 20 years - Month 6 (n=1090) | -23.71 (13.926)
  >20 years - Month 2 (n=833) | -15.10 (11.571)
  >20 years - Month 4 (n=833) | -20.13 (12.810)
  >20 years - Month 6 (n=833) | -22.32 (13.857)

135. Secondary Outcome: Mean Change From Baseline in SDAI by Physician Experience Level With Biologics at Month 2, Month 4, and Month 6
Description: The SDAI is the numerical sum of 5 outcome parameters: tender and swollen joint count (28-joint assessment), patient and physician global assessment of disease activity (VAS 0cm [best] - 10 cm [worst]) and level of C-reactive protein (mg/dL, normal <1 mg/dL) with increasing scores indicating increased level of disease. The SDAI is expressed as a score on a scale with the minimum score=0 (best) to maximum score=86 (worst). Physician experience is defined as the number of years the treating physician has experience managing rheumatoid arthritis with biologics.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  0 to 6 years - Month 2 (n=1146) | -14.71 (11.851)
  0 to 6 years - Month 4 (n=1146) | -20.41 (13.109)
  0 to 6 years - Month 6 (n=1146) | -23.43 (13.784)
  6 to 10 years - Month 2 (n=1712) | -15.25 (11.694)
  6 to 10 years - Month 4 (n=1712) | -20.50 (13.078)
  6 to 10 years - Month 6 (n=1712) | -22.75 (13.831)
  >10 years - Month 2 (n=349) | -14.99 (11.616)
  >10 years - Month 4 (n=349) | -20.17 (12.644)
  >10 years - Month 6 (n=349) | -21.93 (13.491)

136. Secondary Outcome: Mean Change From Baseline in SDAI by the Number of Patients Treated by the Physician With Biologics at Month 2, Month 4, and Month 6
Description: The SDAI is the numerical sum of 5 outcome parameters: tender and swollen joint count (28-joint assessment), patient and physician global assessment of disease activity (VAS 0cm [best] - 10 cm [worst]) and level of C-reactive protein (mg/dL, normal <1 mg/dL) with increasing scores indicating increased level of disease. The SDAI is expressed as a score on a scale with the minimum score=0 (best) to maximum score=86 (worst). The number of patients treated with biologics is defined as the number of patients with rheumatoid arthritis treated by the physician in the last month with biologic agents.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  1-17 patients in prior month - Month 2 (n=1040) | -14.80 (11.566)
  1-17 patients in prior month - Month 4 (n=1040) | -20.65 (12.437)
  1-17 patients in prior month - Month 6 (n=1040) | -24.32 (13.447)
  18-34 patients in prior month - Month 2 (n=1048) | -15.32 (11.736)
  18-34 patients in prior month - Month 4 (n=1048) | -20.51 (13.421)
  18-34 patients in prior month - Month 6 (n=1048) | -22.65 (13.603)
  >=35 patients in prior month - Month 2 (n=1075) | -15.05 (11.797)
  >=35 patients in prior month - Month 4 (n=1075) | -20.19 (13.201)
  >=35 patients in prior month - Month 6 (n=1075) | -21.88 (14.015)

137. Secondary Outcome: Mean Change From Baseline in SDAI by the the Physician Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The SDAI is the numerical sum of 5 outcome parameters: tender and swollen joint count (28-joint assessment), patient and physician global assessment of disease activity (VAS 0cm [best] - 10 cm [worst]) and level of C-reactive protein (mg/dL, normal <1 mg/dL) with increasing scores indicating increased level of disease. The SDAI is expressed as a score on a scale with the minimum score=0 (best) to maximum score=86 (worst). The physician's expectation of treatment outcome was assessed at the start of Month 4, when physicians were asked to rate their expectations of treatment outcome as: high disease activity, moderate disease activity, low disease activity, or remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  High disease activity - Month 2 (n=39) | -19.26 (11.686)
  High disease activity - Month 4 (n=39) | -23.66 (11.626)
  High disease activity - Month 6 (n=39) | -27.55 (13.633)
  Moderate disease activity - Month 2 (n=313) | -14.78 (11.904)
  Moderate disease activity - Month 4 (n=313) | -20.39 (12.757)
  Moderate disease activity - Month 6 (n=313) | -23.22 (14.029)
  Low disease activity - Month 2 (n=1901) | -14.93 (11.812)
  Low disease activity - Month 4 (n=1901) | -20.65 (13.258)
  Low disease activity - Month 6 (n=1901) | -23.33 (13.892)
  Remission - Month 2 (n=959) | -15.16 (11.560)
  Remission - Month 4 (n=959) | -19.91 (12.675)
  Remission - Month 6 (n=959) | -21.79 (13.418)

138. Secondary Outcome: Number of Participants Who Achieved DAS28-ESR EULAR Response
Description: EULAR response was assessed at the end of Month 2, Month 4, and Month 6 by the Disease Activity Score using the 28 tender and swollen joint count calculated with erythrocyte sedimentation rate values (DAS28-ESR). A good response would was defined as a decrease >1.2 units and a final DAS28-ESR < 3.2 units, while a moderate response was defined as a decrease > 1.2 units and final DAS28-ESR >= 3.2 units, OR a decrease of 0.6 to 1.2.
Time Frame: Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Number; unit: Participants
Groups:
- GLM50-SC: In Part 1 of the trial, participants received subcutaneous golimumab 50 mg once monthly.
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Participants
  Study Month 2 | 2127
  Study Month 4 | 2522
  Study Month 6 | 2692

139. Secondary Outcome: Number of Participants Who Achieved DAS28-CRP EULAR Response
Description: DAS28-CRP EULAR response is defined as a good or moderate response that results in a DAS28-CRP >=0.6.
Time Frame: Month 2, Month 4, Month 6
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Participants
  Study Month 2 | 2199
  Study Month 4 | 2530
  Study Month 6 | 2667

140. Secondary Outcome: Number of Participants Achieving Low Disease Activity and Remission at Month 2, Month 4, and Month 6
Description: The number of participants achieving low disease activity or remission was calculated by the DAS28-ESR, DAS28-CRP, and SDAI at study Month 2, Month 4, and Month 6. Low disease activity by DAS28-ESR was defined as >= 2.6 to 3.2, and remission was defined as a DAS28-ESR <2.6. Low disease activity by DAS28-CRP was defined as DAS28-CRP >=2.6 to 3.2, and remission was defined as DAS28-CRP >2.6. Low disease activity by SDAI was defined as SDAI >5.0 to <=20, and remission was defined as SDAI <=5.0.
Time Frame: Month 2, Month 4, Month 6
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Participants
  Low Disease Activity by DAS28-ESR - Month 2 | 545
  Low Disease Activity by DAS28-ESR - Month 4 | 923
  Low Disease Activity by DAS28-ESR - Month 6 | 1228
  Low Disease Activity by DAS28-CRP - Month 2 | 805
  Low Disease Activity by DAS28-CRP - Month 4 | 1268
  Low Disease Activity by DAS28-CRP - Month 6 | 1624
  Low Disease Activity by SDAI - Month 2 | 671
  Low Disease Activity by SDAI - Month 4 | 1205
  Low Disease Activity by SDAI - Month 6 | 1585
  Remission by DAS28-ESR - Month 2 | 251
  Remission by DAS28-ESR - Month 4 | 527
  Remission by DAS28-ESR - Month 6 | 784
  Remission by DAS28-CRP - Month 2 | 380
  Remission by DAS28-CRP - Month 4 | 765
  Remission by DAS28-CRP - Month 6 | 1065
  Remission by SDAI - Month 2 | 88
  Remission by SDAI - Month 4 | 285
  Remission by SDAI - Month 6 | 464

141. Secondary Outcome: Mean Change From Baseline in the Disability Index of the Health Assessment Questionnaire (HAQ-DI) by Concomitant MTX Dose at Month 2, Month 4, and Month 6
Description: The mean change from baseline the disability index of the HAQ was calculated by concomitant MTX dose (low < 10mg/wk, medium >= 10 to < 15 mg/week, and high >=15 mg/week) at study Month 2, Month 4, and Month 6. The HAQ-DI assesses 8 categories of daily activity including dressing, arising, eating, walking, hygiene, reach, grip, and common activities with a score 0 (best) to 3 (worst)with 0=able to do, 1=with some difficulty, 2=with much difficulty, and 3=unable to do for a combined total score of 0 (best) to 32 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Low MTX Dose - Month 2 (n=142) | -0.35 (0.521)
  Low MTX Dose - Month 4 (n=142) | -0.50 (0.547)
  Low MTX Dose - Month 6 (n=142) | -0.58 (0.631)
  Medium MTX Dose - Month 2 (n=526) | -0.41 (0.533)
  Medium MTX Dose - Month 4 (n=526) | -0.54 (0.598)
  Medium MTX Dose - Month 6 (n=526) | -0.61 (0.651)
  High MTX Dose - Month 2 (n=1993) | -0.37 (0.528)
  High MTX Dose - Month 4 (n=1993) | -0.50 (0.613)
  High MTX Dose - Month 6 (n=1993) | -0.56 (0.649)

142. Secondary Outcome: Mean Change From Baseline in HAQ-DI by Concomitant DMARD Background Treatment at Month 2, Month 4, and Month 6
Description: The HAQ-DI assesses 8 categories of daily activity including dressing, arising, eating, walking, hygiene, reach, grip, and common activities with a score 0 (best) to 3 (worst) with 0=able to do, 1=with some difficulty, 2=with much difficulty, and 3=unable to do for a combined total score of 0 (best) to 32 (worst). DMARD Combination 1 = MTX + hydrochloroquine, chloroquine, chloroquine phosphate; Combination 2 = MTX + leflunomide; Combination 3 = MTX + sulfasalazine; Combination 4 = MTX + hydrochloroquine, chloroquine, chloroquine phosphate + sulfasalazine; Combination 5 = leflunomide.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  DMARD Combination 1 - Month 2 (n=1679) | -0.37 (0.521)
  DMARD Combination 1 - Month 4 (n=1679) | -0.50 (0.607)
  DMARD Combination 1 - Month 6 (n=1679) | -0.56 (0.651)
  DMARD Combination 2 - Month 2 (n=433) | -0.40 (0.574)
  DMARD Combination 2 - Month 4 (n=433) | -0.55 (0.633)
  DMARD Combination 2 - Month 6 (n=433) | -0.62 (0.671)
  DMARD Combination 3 - Month 2 (n=216) | -0.34 (0.531)
  DMARD Combination 3 - Month 4 (n=216) | -0.43 (0.624)
  DMARD Combination 3 - Month 6 (n=216) | -0.53 (0.588)
  DMARD Combination 4 - Month 2 (n=150) | -0.36 (0.490)
  DMARD Combination 4 -Month 4 (n=150) | -0.45 (0.523)
  DMARD Combination 4 - Month 6 (n=150) | -0.55 (0.627)
  DMARD Combination 5 - Month 2 (n=106) | -0.38 (0.501)
  DMARD Combination 5 - Month 4 (n=106) | -0.67 (0.599)
  DMARD Combination 5 - Month 6 (n=106) | -0.63 (0.709)
  DMARD Combination 6 - Month 2 (n=303) | -0.33 (0.490)
  DMARD Combination 6 - Month 4 (n=303) | -0.43 (0.540)
  DMARD Combination 6 - Month 6 (n=303) | -0.47 (0.579)

143. Secondary Outcome: Mean Change From Baseline in HAQ-DI by Concomitant Corticosteroid Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the HAQ-DI by participant concomitant corticosteroid use was calculated at study Month 2, Month 4, and Month 6. The HAQ-DI assesses 8 categories of daily activity including dressing, arising, eating, walking, hygiene, reach, grip, and common activities with a score 0 (best) to 3 (worst) with 0=able to do, 1=with some difficulty, 2=with much difficulty, and 3=unable to do for a combined total score of 0 (best) to 32 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Did Not Receive Corticosteroids - Month 2 (n=1201) | -0.32 (0.476)
  Did Not Receive Corticosteroids - Month 4 (n=1201) | -0.47 (0.582)
  Did Not Receive Corticosteroids - Month 6 (n=1201) | -0.51 (0.612)
  Received Corticosteroids - Month 2 (n=2076) | -0.39 (0.542)
  Received Corticosteroids - Month 4 (n=2076) | -0.51 (0.604)
  Received Corticosteroids - Month 6 (n=2076) | -0.58 (0.653)

144. Secondary Outcome: Mean Change From Baseline in HAQ-DI by the Number of DMARD Failures at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the HAQ-DI by the number of participant DMARD failures was calculated at study Month 2, Month 4, and Month 6. The HAQ-DI assesses 8 categories of daily activity including dressing, arising, eating, walking, hygiene, reach, grip, and common activities with a score 0 (best) to 3 (worst) with 0=able to do, 1=with some difficulty, 2=with much difficulty, and 3=unable to do for a combined total score of 0 (best) to 32 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Failed 1 DMARD - Month 2 (n=1128) | -0.39 (0.545)
  Failed 1 DMARD - Month 4 (n=1128) | -0.54 (0.630)
  Failed 1 DMARD - Month 6 (n=1128) | -0.60 (0.679)
  Failed 2 DMARDs - Month 2 (n=1175) | -0.37 (0.533)
  Failed 2 DMARDs - Month 4 (n=1175) | -0.48 (0.605)
  Failed 2 DMARDs - Month 6 (n=1175) | -0.55 (0.644)
  Failed >=3 DMARDs - Month 2 (n=973) | -0.33 (0.470)
  Failed >=3 DMARDs - Month 4 (n=973) | -0.46 (0.541)
  Failed >=3 DMARDs - Month 6 (n=973) | -0.51 (0.580)

145. Secondary Outcome: Mean Change From Baseline in HAQ-DI by Duration of Disease at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the HAQ-DI by the participant duration of disease was calculated at study Month 2, Month 4, and Month 6. The duration of disease is defined as the time since the diagnosis of rheumatoid arthritis. The HAQ-DI assesses 8 categories of daily activity including dressing, arising, eating, walking, hygiene, reach, grip, and common activities with a score 0 (best) to 3 (worst) with 0=able to do, 1=with some difficulty, 2=with much difficulty, and 3=unable to do for a combined total score of 0 (best) to 32 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Duration < 2 years - Month 2 (n=897) | -0.36 (0.547)
  Duration < 2 years - Month 4 (n=897) | -0.50 (0.619)
  Duration < 2 years - Month 6 (n=897) | -0.57 (0.669)
  Duration 2 to <5 years - Month 2 (n=763) | -0.38 (0.532)
  Duration 2 to <5 years - Month 4 (n=763) | -0.49 (0.621)
  Duration 2 to <5 years - Month 6 (n=763) | -0.56 (0.662)
  Duration 5 to 10 years - Month 2 (n=692) | -0.40 (0.531)
  Duration 5 to 10 years - Month 4 (n=692) | -0.54 (0.602)
  Duration 5 to 10 years - Month 6 (n=692) | -0.58 (0.642)
  Duration > 10 years - Month 2 (n=924) | -0.33 (0.470)
  Duration > 10 years - Month 4 (n=924) | -0.45 (0.545)
  Duration > 10 years - Month 6 (n=924) | -0.52 (0.582)

146. Secondary Outcome: Mean Change From Baseline in HAQ-DI by Baseline Level of Disease Activity at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the HAQ-DI by the participant baseline level of disease activity was calculated at study Month 2, Month 4, and Month 6. The HAQ-DI assesses 8 categories of daily activity including dressing, arising, eating, walking, hygiene, reach, grip, and common activities with a score 0 (best) to 3 (worst) with 0=able to do, 1=with some difficulty, 2=with much difficulty, and 3=unable to do for a combined total score of 0 (best) to 32 (worst). DAS28-ESR > 5.1 = high disease activity, DAS28-ESR < 3.2 to < =5.1 = low disease activity, and DAS28-ESR <2.6 = remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  DAS28 > 3.2 to <=5.1 - Month 2 (n=697) | -0.25 (0.430)
  DAS28 > 3.2 to <=5.1 - Month 4 (n=697) | -0.33 (0.512)
  DAS28 > 3.2 to <=5.1 - Month 6 (n=697) | -0.37 (0.525)
  DAS28 > 5.1 - Month 2 (n=2570) | -0.40 (0.537)
  DAS28 > 5.1 - Month 4 (n=2570) | -0.54 (0.609)
  DAS28 > 5.1 - Month 6 (n=2570) | -0.61 (0.658)

147. Secondary Outcome: Mean Change From Baseline in HAQ-DI by Baseline RF Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the HAQ-DI by the participant baseline RF level was calculated at study Month 2, Month 4, and Month 6. The HAQ-DI assesses 8 categories of daily activity including dressing, arising, eating, walking, hygiene, reach, grip, and common activities with a score 0 (best) to 3 (worst) with 0=able to do, 1=with some difficulty, 2=with much difficulty, and 3=unable to do for a combined total score of 0 (best) to 32 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  RF <=22 IU/mL - Month 2 (n=1025) | -0.28 (0.486)
  RF <=22 IU/mL - Month 4 (n=1025) | -0.41 (0.580)
  RF <=22 IU/mL - Month 6 (n=1025) | -0.45 (0.599)
  RF >22 to <=146 IU/mL - Month 2 (n=1080) | -0.36 (0.496)
  RF >22 to <=146 IU/mL - Month 4 (n=1080) | -0.48 (0.563)
  RF >22 to <=146 IU/mL - Month 6 (n=1080) | -0.52 (0.602)
  RF >146 IU/mL - Month 2 (n=1126) | -0.46 (0.559)
  RF >146 IU/mL - Month 4 (n=1126) | -0.60 (0.630)
  RF >146 IU/mL - Month 6 (n=1126) | -0.70 (0.686)

148. Secondary Outcome: Mean Change From Baseline in HAQ-DI by Baseline Anti-CCP Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the HAQ-DI by the participant baseline serum level of anti-CCP was calculated at study Month 2, Month 4, and Month 6. The HAQ-DI assesses 8 categories of daily activity including dressing, arising, eating, walking, hygiene, reach, grip, and common activities with a score 0 (best) to 3 (worst) with 0=able to do, 1=with some difficulty, 2=with much difficulty, and 3=unable to do for a combined total score of 0 (best) to 32 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Anti-CCP <=40 U/mL - Month 2 (n=1036) | -0.28 (0.475)
  Anti-CCP <=40 U/mL - Month 4 (n=1036) | -0.41 (0.567)
  Anti-CCP <=40 U/mL - Month 6 (n=1036) | -0.45 (0.587)
  Anti-CCP >40 to <=380 U/mL - Month 2 (n=1112) | -0.40 (0.527)
  Anti-CCP >40 to <=380 U/mL - Month 4 (n=1112) | -0.52 (0.607)
  Anti-CCP >40 to <=380 U/mL - Month 6 (n=1112) | -0.58 (0.641)
  Anti-CCP >380 U/mL - Month 2 (n=1074) | -0.43 (0.535)
  Anti-CCP >380 U/mL - Month 4 (n=1074) | -0.55 (0.604)
  Anti-CCP >380 U/mL - Month 6 (n=1074) | -0.63 (0.666)

149. Secondary Outcome: Mean Change From Baseline in HAQ-DI by Smoking Status at Month 2, Month 4, and Month 6
Description: The HAQ-DI assesses 8 categories of daily activity including dressing, arising, eating, walking, hygiene, reach, grip, and common activities with a score 0 (best) to 3 (worst) with 0=able to do, 1=with some difficulty, 2=with much difficulty, and 3=unable to do for a combined total score of 0 (best) to 32 (worst). Pack years smoked is defined as the total number of packs smoked per day multiplied by the number of years the participant smoked.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Non-Smoker - Month 2 (n=1960) | -0.38 (0.540)
  Non-Smoker - Month 4 (n=1960) | -0.52 (0.615)
  Non-Smoker - Month 6 (n=1960) | -0.59 (0.652)
  Smoking history >=20 years - Month 2 (n=324) | -0.35 (0.462)
  Smoking history >=20 years - Month 4 (n=324) | -0.49 (0.552)
  Smoking history >=20 years - Month 6 (n=324) | -0.52 (0.600)
  Smoking history <20 years - Month 2 (n=314) | -0.43 (0.505)
  Smoking history <20 years - Month 4 (n=314) | -0.51 (0.572)
  Smoking history <20 years - Month 6 (n=314) | -0.57 (0.625)
  Currently smokes <0.5 packs/day - Month 2 (n=223) | -0.30 (0.480)
  Currently smokes <0.5 packs/day - Month 4 (n=223) | -0.44 (0.562)
  Currently smokes <0.5 pack/day - Month 6 (n=223) | -0.52 (0.628)
  Currently smokes 0.5-1 pack/day - Month 2 (n=397) | -0.32 (0.490)
  Currently smokes 0.5-1 pack/day - Month 4 (n=397) | -0.42 (0.571)
  Currently smokes 0.5-1 pack/day - Month 6 (n=397) | -0.45 (0.616)
  Currently smokes >1 packs/day - Month 2 (n=59) | -0.37 (0.517)
  Currently smokes >1 packs/day - Month 4 (n=59) | -0.34 (0.539)
  Currently smokes >1 packs/day - Month 6 (n=59) | -0.42 (0.584)
  Pack years <7.5 - Month 2 (n=423) | -0.38 (0.513)
  Pack years <7.5 - Month 4 (n=423) | -0.49 (0.580)
  Pack years <7.5 - Month 6 (n=423) | -0.58 (0.642)
  Pack years 7.5 to 20.5 - Month 2 (n=454) | -0.37 (0.494)
  Pack years 7.5 to 20.5 - Month 4 (n=454) | -0.48 (0.567)
  Pack years 7.5 to 20.5 - Month 6 (n=454) | -0.52 (0.622)
  Pack years >20.5 - Month 2 (n=418) | -0.31 (0.455)
  Pack years >20.5 - Month 4 (n=418) | -0.40 (0.547)
  Pack years >20.5 - Month 6 (n=418) | -0.42 (0.572)

150. Secondary Outcome: Mean Change From Baseline in HAQ-DI by Eligibility for Anti-TNF Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the HAQ-DI by the participant eligibility for anti-TNF treatment was calculated at study Month 2, Month 4, and Month 6. The HAQ-DI assesses 8 categories of daily activity including dressing, arising, eating, walking, hygiene, reach, grip, and common activities with a score 0 (best) to 3 (worst) with 0=able to do, 1=with some difficulty, 2=with much difficulty, and 3=unable to do for a combined total score of 0 (best) to 32 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Anti-TNF treatment Ineligible - Month 2 (n=106) | -0.27 (0.406)
  Anti-TNF treatment Ineligible - Month 4 (n=106) | -0.44 (0.565)
  Anti-TNF treatment Ineligible - Month 6 (n=106) | -0.47 (0.576)
  Anti-TNF treatment Eligible- Month 2 (n=3171) | -0.37 (0.523)
  Anti-TNF treatment Eligible - Month 4 (n=3171) | -0.50 (0.597)
  EligAnti-TNF treatment Eligible - Month 6 (n=3171) | -0.56 (0.641)

151. Secondary Outcome: Mean Change From Baseline in HAQ-DI by Participant Baseline Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the HAQ-DI by the participant baseline expectation of treatment outcome was evaluated at study Month 2, Month 4, and Month 6. The HAQ-DI assesses 8 categories of daily activity including dressing, arising, eating, walking, hygiene, reach, grip, and common activities with a score 0 (best) to 3 (worst) with 0=able to do, 1=with some difficulty, 2=with much difficulty, and 3=unable to do for a combined total score of 0 (best) to 32 (worst). The participant expectation scale was evaluated by questionnaire for a categorical score of 1 (best) to 5 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  <=1.5 - Month 2 (n=1211) | -0.46 (0.557)
  <=1.5 - Month 4 (n=1211) | -0.59 (0.634)
  <=1.5 - Month 6 (n=1211) | -0.65 (0.691)
  >1.5 to 1.86 - Month 2 (n=1009) | -0.34 (0.488)
  >1.5 to 1.86 - Month 4 (n=1009) | -0.48 (0.580)
  >1.5 to 1.86 - Month 6 (n=1009) | -0.55 (0.610)
  >=1.86 - Month 2 (n=1053) | -0.29 (0.490)
  >=1.86 - Month 4 (n=1053) | -0.39 (0.549)
  >=1.86 - Month 6 (n=1053) | -0.44 (0.583)

152. Secondary Outcome: Mean Change From Baseline in HAQ-DI by Physician Experience Level at Month 2, Month 4, and Month 6
Description: The HAQ-DI assesses 8 categories of daily activity including dressing, arising, eating, walking, hygiene, reach, grip, and common activities with a score 0 (best) to 3 (worst) with 0=able to do, 1=with some difficulty, 2=with much difficulty, and 3=unable to do for a combined total score of 0 (best) to 32 (worst). Physician experience is defined as the number of years the treating physician has experience managing patients with rheumatoid arthritis.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  <=10 years - Month 2 (n=1304) | -0.37 (0.515)
  <=10 years - Month 4 (n=1304) | -0.48 (0.573)
  <=10 years - Month 6 (n=1304) | -0.55 (0.627)
  >10 to 20 years - Month 2 (n=1104) | -0.35 (0.511)
  >10 to 20 years - Month 4 (n=1104) | -0.48 (0.611)
  >10 to 20 years - Month 6 (n=1104) | -0.54 (0.644)
  >20 years - Month 2 (n=850) | -0.39 (0.535)
  >20 years - Month 4 (n=850) | -0.53 (0.607)
  >20 years - Month 6 (n=850) | -0.59 (0.650)

153. Secondary Outcome: Mean Change From Baseline in HAQ-DI by Physician Experience Level With Biologics at Month 2, Month 4, and Month 6
Description: The HAQ-DI assesses 8 categories of daily activity including dressing, arising, eating, walking, hygiene, reach, grip, and common activities with a score 0 (best) to 3 (worst) with 0=able to do, 1=with some difficulty, 2=with much difficulty, and 3=unable to do for a combined total score of 0 (best) to 32 (worst). Physician experience is defined as the number of years the treating physician has experience managing rheumatoid arthritis with biologics.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  0 to 6 years - Month 2 (n=1160) | -0.39 (0.533)
  0 to 6 years - Month 4 (n=1160) | -0.51 (0.596)
  0 to 6 years - Month 6 (n=1160) | -0.60 (0.631)
  6 to 10 years - Month 2 (n=1744) | -0.35 (0.511)
  6 to 10 years - Month 4 (n=1744) | -0.49 (0.593)
  6 to 10 years - Month 6 (n=1744) | -0.53 (0.650)
  >10 years - Month 2 (n=354) | -0.37 (0.512)
  >10 years - Month 4 (n=354) | -0.48 (0.602)
  >10 years - Month 6 (n=354) | -0.54 (0.607)

154. Secondary Outcome: Mean Change From Baseline in HAQ-DI by the Number of Patients Treated by the Physician With Biologics at Month 2, Month 4, and Month 6
Description: The HAQ-DI assesses 8 categories of daily activity including dressing, arising, eating, walking, hygiene, reach, grip, and common activities with a scores ranging from 0 (best) to 3 (best) with 0=able to do, 1=with some difficulty, 2=with much difficulty, and 3=unable to do for a combined total score of 0 (best) to 32 (worst). The number of patients treated with biologics is defined as the number of patients with rheumatoid arthritis treated by the physician in the last month with biologic agents.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Units on a Scale
  1-17 patients in prior month - Month 2 (n=1055) | -0.39 (0.529)
  1-17 patients in prior month - Month 4 (n=1055) | -0.51 (0.594)
  1-17 patients in prior month - Month 6 (n=1055) | -0.59 (0.625)
  18-34 patients in prior month - Month 2 (n=1060) | -0.35 (0.501)
  18-34 patients in prior month - Month 4 (n=1060) | -0.48 (0.580)
  18-34 patients in prior month - Month 6 (n=1060) | -0.53 (0.627)
  >=35 patients in prior month - Month 2 (n=1097) | -0.36 (0.529)
  >=35 patients in prior month - Month 4 (n=1097) | -0.50 (0.609)
  >=35 patients in prior month - Month 6 (n=1097) | -0.55 (0.664)

155. Secondary Outcome: Mean Change From Baseline in HAQ-DI by the the Physician Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The HAQ-DI assesses 8 categories of daily activity including dressing, arising, eating, walking, hygiene, reach, grip, and common activities with a score 0 (best) to 3 (worst) with 0=able to do, 1=with some difficulty, 2=with much difficulty, and 3=unable to do for a combined total score of 0 (best) to 32 (worst). The physician's expectation of treatment outcome was assessed at the start of Month 4, when physicians were asked to rate their expectations of treatment outcome as: high disease activity, moderate disease activity, low disease activity, or remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Units on a Scale
  High disease activity - Month 2 (n=40) | -0.36 (0.563)
  High disease activity - Month 4 (n=40) | -0.49 (0.536)
  High disease activity - Month 6 (n=40) | -0.54 (0.593)
  Moderate disease activity - Month 2 (n=325) | -0.29 (0.482)
  Moderate disease activity - Month 4 (n=325) | -0.43 (0.529)
  Moderate disease activity - Month 6 (n=325) | -0.49 (0.575)
  Low disease activity - Month 2 (n=1930) | -0.38 (0.526)
  Low disease activity - Month 4 (n=1930) | -0.51 (0.610)
  Low disease activity - Month 6 (n=1930) | -0.57 (0.642)
  Remission - Month 2 (n=966) | -0.38 (0.515)
  Remission - Month 4 (n=966) | -0.49 (0.587)
  Remission - Month 6 (n=966) | -0.54 (0.653)

156. Secondary Outcome: Number of Participants Who Achieved Minimal or Absence of Functional Impairment
Description: The number of participants that achieved minimal or absence of functional impairment as assessed by the HAQ at study Month 2, Month 4, and Month 6 was calculated. Minimal or absence of functional impairment was defined as a HAQ score of <=0.5. The HAQ evaluates participants on a scale of 0 to 3, with 0=with no difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do.
Time Frame: Month 2, Month 4, Month 6
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Participants
  Study Month 2 | 865
  Study Month 4 | 1087
  Study Month 6 | 1226

157. Secondary Outcome: Mean Change From Baseline in the EuroQOL (EQ-5D) Quality-of-Life Questionnaire by Concomitant MTX Dose at Month 2, Month 4, and Month 6
Description: Concomitant MTX dose was defined as low < 10mg/wk, medium >= 10 to < 15 mg/week, and and high >=15 mg/week. The EQ-5D assesses the 5 domains of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant is asked to indicate their health state by ticking the box against the most appropriate statement in each of the 5 dimensions. The digits (1 [best] to 3 [worst]; with 0= no problems, 1 = some problems, 2 = some problems, and 3= severe problems) for the 5 dimensions can be combined in a 5-digit number describing the participant's health state. The numerals 1 to 3 have no arithmetic properties and should not be used as a cardinal score.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Low MTX Dose - Month 2 (n=142) | 0.20 (0.331)
  Low MTX Dose - Month 4 (n=142) | 0.25 (0.318)
  Low MTX Dose - Month 6 (n=142) | 0.26 (0.312)
  Medium MTX Dose - Month 2 (n=526) | 0.20 (0.325)
  Medium MTX Dose - Month 4 (n=526) | 0.24 (0.338)
  Medium MTX Dose - Month 6 (n=526) | 0.27 (0.332)
  High MTX Dose - Month 2 (n=1985) | 0.20 (0.311)
  High MTX Dose - Month 4 (n=1985) | 0.23 (0.336)
  High MTX Dose - Month 6 (n=1985) | 0.26 (0.346)

158. Secondary Outcome: Mean Change From Baseline in EQ-5D by Concomitant DMARD Background Treatment at Month 2, Month 4, and Month 6
Description: The EQ-5D assesses the 5 domains of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant is asked to indicate their health state by ticking the box against the most appropriate statement in each of the 5 dimensions. The digits (1 [best] to 3 [worst]; with 0= no problems, 1 = some problems, 2 = some problems, and 3= severe problems) for the 5 dimensions can be combined in a 5-digit number describing the participant's health state. The numerals 1 to 3 have no arithmetic properties and should not be used as a cardinal score. DMARD Combination 1=MTX + hydrochloroquine, chloroquine, chloroquine phosphate; Combination 2=MTX + leflunomide; Combination 3=MTX +sulfasalazine; Combination 4=MTX + hydrochloroquine, chloroquine, chloroquine phosphate+sulfasalazine; Combination 5=leflunomide.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  DMARD Combination 1 - Month 2 (n=1672) | 0.21 (0.313)
  DMARD Combination 1 - Month 4 (n=1672) | 0.24 (0.336)
  DMARD Combination 1 - Month 6 (n=1672) | 0.26 (0.341)
  DMARD Combination 2 - Month 2 (n=432) | 0.19 (0.316)
  DMARD Combination 2 - Month 4 (n=432) | 0.23 (0.337)
  DMARD Combination 2 - Month 6 (n=432) | 0.27 (0.346)
  DMARD Combination 3 - Month 2 (n=216) | 0.16 (0.343)
  DMARD Combination 3 - Month 4 (n=216) | 0.18 (0.355)
  DMARD Combination 3 - Month 6 (n=216) | 0.21 (0.325)
  DMARD Combination 4 - Month 2 (n=150) | 0.25 (0.307)
  DMARD Combination 4 -Month 4 (n=150) | 0.24 (0.316)
  DMARD Combination 4 - Month 6 (n=150) | 0.26 (0.349)
  DMARD Combination 5 - Month 2 (n=105) | 0.22 (0.273)
  DMARD Combination 5 - Month 4 (n=105) | 0.28 (0.302)
  DMARD Combination 5 - Month 6 (n=105) | 0.29 (0.374)
  DMARD Combination 6 - Month 2 (n=303) | 0.17 (0.284)
  DMARD Combination 6 - Month 4 (n=303) | 0.21 (0.306)
  DMARD Combination 6 - Month 6 (n=303) | 0.19 (.341)

159. Secondary Outcome: Mean Change From Baseline in EQ-5D by Concomitant Corticosteroid Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the EQ-5D by participant concomitant corticosteroid use was calculated at study Month 2, Month 4, and Month 6. The EQ-5D assesses the 5 domains of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant is asked to indicate their health state by ticking the box against the most appropriate statement in each of the 5 dimensions. The digits (1 [best] to 3 [worst]; with 0= no problems, 1 = some problems, 2 = some problems, and 3= severe problems) for the 5 dimensions can be combined in a 5-digit number describing the participant's health state. The numerals 1 to 3 have no arithmetic properties and should not be used as a cardinal score.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Did Not Receive Corticosteroids - Month 2 (n=1199) | 0.17 (0.291)
  Did Not Receive Corticosteroids - Month 4 (n=1199) | 0.21 (0.306)
  Did Not Receive Corticosteroids - Month 6 (n=1199) | 0.22 (0.329)
  Received Corticosteroids - Month 2 (n=2069) | 0.21 (0.322)
  Received Corticosteroids - Month 4 (n=2069) | 0.24 (0.343)
  Received Corticosteroids - Month 6 (n=2069) | 0.27 (0.348)

160. Secondary Outcome: Mean Change From Baseline in EQ-5D by the Number of DMARD Failures at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the EQ-5D by the number of participant DMARD failures was calculated at study Month 2, Month 4, and Month 6. The EQ-5D assesses the 5 domains of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant is asked to indicate their health state by ticking the box against the most appropriate statement in each of the 5 dimensions. The digits (1 [best] to 3 [worst]; with 0= no problems, 1 = some problems, 2 = some problems, and 3= severe problems) for the 5 dimensions can be combined in a 5-digit number describing the participant's health state. The numerals 1 to 3 have no arithmetic properties and should not be used as a cardinal score.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Failed 1 DMARD - Month 2 (n=1124) | 0.21 (0.324)
  Failed 1 DMARD - Month 4 (n=1124) | 0.24 (0.338)
  Failed 1 DMARD - Month 6 (n=1124) | 0.27 (0.347)
  Failed 2 DMARDs - Month 2 (n=1173) | 0.19 (0.312)
  Failed 2 DMARDs - Month 4 (n=1173) | 0.22 (0.329)
  Failed 2 DMARDs - Month 6 (n=1173) | 0.24 (0.346)
  Failed >=3 DMARDs - Month 2 (n=970) | 0.19 (0.298)
  Failed >=3 DMARDs - Month 4 (n=970) | 0.22 (0.323)
  Failed >=3 DMARDs - Month 6 (n=970) | 0.24 (0.331)

161. Secondary Outcome: Mean Change From Baseline in EQ-5D by Duration of Disease at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the EQ-5D by the participant duration of disease was calculated at study Month 2, Month 4, and Month 6. The duration of disease is defined as the time since the diagnosis of rheumatoid arthritis. The EQ-5D assesses the 5 domains of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant is asked to indicate their health state by ticking the box against the most appropriate statement in each of the 5 dimensions. The digits (1 [best] to 3 [worst]; with 0= no problems, 1 = some problems, 2 = some problems, and 3= severe problems) for the 5 dimensions can be combined in a 5-digit number describing the participant's health state. The numerals 1 to 3 have no arithmetic properties and should not be used as a cardinal score.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Duration < 2 years - Month 2 (n=893) | 0.18 (0.315)
  Duration < 2 years - Month 4 (n=893) | 0.21 (0.339)
  Duration < 2 years - Month 6 (n=893) | 0.24 (0.342)
  Duration 2 to <5 years - Month 2 (n=760) | 0.21 (0.311)
  Duration 2 to <5 years - Month 4 (n=760) | 0.23 (0.319)
  Duration 2 to <5 years - Month 6 (n=760) | 0.24 (0.339)
  Duration 5 to 10 years - Month 2 (n=691) | 0.22 (0.315)
  Duration 5 to 10 years - Month 4 (n=691) | 0.24 (0.341)
  Duration 5 to 10 years - Month 6 (n=691) | 0.26 (0.357)
  Duration > 10 years - Month 2 (n=923) | 0.19 (0.307)
  Duration > 10 years - Month 4 (n=923) | 0.23 (0.323)
  Duration > 10 years - Month 6 (n=923) | 0.25 (0.334)

162. Secondary Outcome: Mean Change From Baseline in EQ-5D by Baseline Level of Disease Activity at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the EQ-5D by the participant baseline level of disease activity was calculated at study Month 2, Month 4, and Month 6. The EQ-5D assesses the 5 domains of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant is asked to indicate their health state by ticking the box against the most appropriate statement in each of the 5 dimensions. The digits (1 [best] to 3 [worst]; with 0= no problems, 1 = some problems, 2 = some problems, and 3= severe problems) for the 5 dimensions can be combined in a 5-digit number describing the participant's health state. The numerals 1 to 3 have no arithmetic properties and should not be used as a cardinal score. DAS28-ESR > 5.1 = high disease activity, DAS28-ESR < 3.2 to < =5.1 = low disease activity, and DAS28-ESR <2.6 = remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  DAS28 > 3.2 to <=5.1 - Month 2 (n=695) | 0.10 (0.232)
  DAS28 > 3.2 to <=5.1 - Month 4 (n=695) | 0.12 (0.253)
  DAS28 > 3.2 to <=5.1 - Month 6 (n=695) | 0.13 (0.267)
  DAS28 > 5.1 - Month 2 (n=2563) | 0.22 (0.325)
  DAS28 > 5.1 - Month 4 (n=2563) | 0.26 (0.343)
  DAS28 > 5.1 - Month 6 (n=2563) | 0.28 (0.353)

163. Secondary Outcome: Mean Change From Baseline in EQ-5D by Baseline RF Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the EQ-5D by the participant baseline RF level was calculated at study Month 2, Month 4, and Month 6. The EQ-5D assesses the 5 domains of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant is asked to indicate their health state by ticking the box against the most appropriate statement in each of the 5 dimensions. The digits (1 [best] to 3 [worst]; with 0= no problems, 1 = some problems, 2 = some problems, and 3= severe problems) for the 5 dimensions can be combined in a 5-digit number describing the participant's health state. The numerals 1 to 3 have no arithmetic properties and should not be used as a cardinal score.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  RF <=22 IU/mL - Month 2 (n=1020) | 0.16 (0.296)
  RF <=22 IU/mL - Month 4 (n=1020) | 0.19 (0.322)
  RF <=22 IU/mL - Month 6 (n=1020) | 0.21 (0.314)
  RF >22 to <=146 IU/mL - Month 2 (n=1079) | 0.19 (0.305)
  RF >22 to <=146 IU/mL - Month 4 (n=1079) | 0.22 (0.324)
  RF >22 to <=146 IU/mL - Month 6 (n=1079) | 0.23 (0.339)
  RF >146 IU/mL - Month 2 (n=1123) | 0.25 (0.328)
  RF >146 IU/mL - Month 4 (n=1123) | 0.27 (0.338)
  RF >146 IU/mL - Month 6 (n=1123) | 0.30 (0.365)

164. Secondary Outcome: Mean Change From Baseline in EQ-5D by Baseline Anti-CCP Level at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the EQ-5D by the participant baseline serum level of anti-CCP was calculated at study Month 2, Month 4, and Month 6. The EQ-5D assesses the 5 domains of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant is asked to indicate their health state by ticking the box against the most appropriate statement in each of the 5 dimensions. The digits (1 [best] to 3 [worst]; with 0= no problems, 1 = some problems, 2 = some problems, and 3= severe problems) for the 5 dimensions can be combined in a 5-digit number describing the participant's health state. The numerals 1 to 3 have no arithmetic properties and should not be used as a cardinal score.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Anti-CCP <=40 U/mL - Month 2 (n=1033) | 0.15 (0.297)
  Anti-CCP <=40 U/mL - Month 4 (n=1033) | 0.19 (0.324)
  Anti-CCP <=40 U/mL - Month 6 (n=1033) | 0.21 (0.319)
  Anti-CCP >40 to <=380 U/mL - Month 2 (n=1109) | 0.21 (0.313)
  Anti-CCP >40 to <=380 U/mL - Month 4 (n=1109) | 0.24 (0.328)
  Anti-CCP >40 to <=380 U/mL - Month 6 (n=1109) | 0.25 (0.343)
  Anti-CCP >380 U/mL - Month 2 (n=1071) | 0.23 (0.321)
  Anti-CCP >380 U/mL - Month 4 (n=1071) | 0.25 (0.336)
  Anti-CCP >380 U/mL - Month 6 (n=1071) | 0.28 (0.28)

165. Secondary Outcome: Mean Change From Baseline in EQ-5D by Smoking Status at Month 2, Month 4, and Month 6
Description: The EQ-5D assesses the 5 domains of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant is asked to indicate their health state by ticking the box against the most appropriate statement in each of the 5 dimensions. The digits (1 [best] to 3 [worst]; with 0= no problems, 1 = some problems, 2 = some problems, and 3= severe problems) for the 5 dimensions can be combined in a 5-digit number describing the participant's health state. The numerals 1 to 3 have no arithmetic properties and should not be used as a cardinal score. Pack years smoked is defined as the total number of packs smoked per day multiplied by the number of years the participant smoked.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Non-Smoker - Month 2 (n=1957) | 0.21 (0.319)
  Non-Smoker - Month 4 (n=1957) | 0.24 (0.334)
  Non-Smoker - Month 6 (n=1957) | 0.27 (0.339)
  Smoking history >=20 years - Month 2 (n=322) | 0.18 (0.300)
  Smoking history >=20 years - Month 4 (n=322) | 0.20 (0.304)
  Smoking history >=20 years - Month 6 (n=322) | 0.21 (0.324)
  Smoking history <20 years - Month 2 (n=312) | 0.19 (0.315)
  Smoking history <20 years - Month 4 (n=312) | 0.22 (0.334)
  Smoking history <20 years - Month 6 (n=312) | 0.24 (0.351)
  Currently smokes <0.5 packs/day - Month 2 (n=223) | 0.16 (0.301)
  Currently smokes <0.5 packs/day - Month 4 (n=223) | 0.20 (0.338)
  Currently smokes <0.5 pack/day - Month 6 (n=223) | 0.24 (0.344)
  Currently smokes 0.5-1 pack/day - Month 2 (n=395) | 0.20 (0.296)
  Currently smokes 0.5-1 pack/day - Month 4 (n=395) | 0.20 (0.327)
  Currently smokes 0.5-1 pack/day - Month 6 (n=395) | 0.21 (0.363)
  Currently smokes >1 packs/day - Month 2 (n=59) | 0.14 (0.269)
  Currently smokes >1 packs/day - Month 4 (n=59) | 0.15 (0.292)
  Currently smokes >1 packs/day - Month 6 (n=59) | 0.19 (0.325)
  Pack years <7.5 - Month 2 (n=421) | 0.21 (0.314)
  Pack years <7.5 - Month 4 (n=421) | 0.22 (0.333)
  Pack years <7.5 - Month 6 (n=421) | 0.26 (0.357)
  Pack years 7.5 to 20.5 - Month 2 (n=453) | 0.17 (0.284)
  Pack years 7.5 to 20.5 - Month 4 (n=453) | 0.20 (0.310)
  Pack years 7.5 to 20.5 - Month 6 (n=453) | 0.335 (0.19)
  Pack years >20.5 - Month 2 (n=415) | 0.17 (0.301)
  Pack years >20.5 - Month 4 (n=415) | 0.19 (0.325)
  Pack years >20.5 - Month 6 (n=415) | 0.19 (0.342)

166. Secondary Outcome: Mean Change From Baseline in EQ-5D by Eligibility for Anti-TNF Treatment at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the EQ-5D by the participant eligibility for anti-TNF treatment was calculated at study Month 2, Month 4, and Month 6. The EQ-5D assesses the 5 domains of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant is asked to indicate their health state by ticking the box against the most appropriate statement in each of the 5 dimensions. The digits (1 [best] to 3 [worst]; with 0= no problems, 1 = some problems, 2 = some problems, and 3= severe problems) for the 5 dimensions can be combined in a 5-digit number describing the participant's health state. The numerals 1 to 3 have no arithmetic properties and should not be used as a cardinal score.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  Anti-TNF treatment Ineligible - Month 2 (n=106) | 0.15 (0.298)
  Anti-TNF treatment Ineligible - Month 4 (n=106) | 0.18 (0.305)
  Anti-TNF treatment Ineligible - Month 6 (n=106) | 0.19 (0.305)
  Anti-TNF treatment Eligible - Month 2 (n=3162) | 0.20 (0.312)
  Anti-TNF treatment Eligible - Month 4 (n=3162) | 0.23 (0.331)
  Anti-TNF treatment Eligible - Month 6 (n=3162) | 0.25 (0.343)

167. Secondary Outcome: Mean Change From Baseline in EQ-5D by Participant Baseline Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The mean change from baseline in the EQ-5D by the participant baseline expectation of treatment outcome was evaluated at study Month 2, Month 4, and Month 6. The EQ-5D assesses the 5 domains of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant is asked to indicate their health state by ticking the box against the most appropriate statement in each of the 5 dimensions. The digits (1 [best] to 3 [worst]; with 0= no problems, 1 = some problems, 2 = some problems, and 3= severe problems) for the 5 dimensions can be combined in a 5-digit number describing the participant's health state. The numerals 1 to 3 have no arithmetic properties and should not be used as a cardinal score. The participant expectation scale was evaluated by questionnaire for a categorical score of 1 (best) to 5 (worst).
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  <=1.5 - Month 2 (n=1208) | 0.22 (0.323)
  <=1.5 - Month 4 (n=1208) | 0.26 (0.337)
  <=1.5 - Month 6 (n=1208) | 0.28 (0.349)
  >1.5 to 1.86 - Month 2 (n=1006) | 0.20 (0.304)
  >1.5 to 1.86 - Month 4 (n=1006) | 0.23 (0.319)
  >1.5 to 1.86 - Month 6 (n=1006) | 0.25 (0.331)
  >=1.86 - Month 2 (n=1050) | 0.17 (0.304)
  >=1.86 - Month 4 (n=1050) | 0.19 (0.329)
  >=1.86 - Month 6 (n=1050) | 0.21 (0.341)

168. Secondary Outcome: Mean Change From Baseline in EQ-5D by Physician Experience Level at Month 2, Month 4, and Month 6
Description: The EQ-5D assesses the 5 domains of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant is asked to indicate their health state by ticking the box against the most appropriate statement in each of the 5 dimensions. The digits (1 [best] to 3 [worst]; with 0= no problems, 1 = some problems, 2 = some problems, and 3= severe problems) for the 5 dimensions can be combined in a 5-digit number describing the participant's health state. The numerals 1 to 3 have no arithmetic properties and should not be used as a cardinal score. Physician experience is defined as the number of years the treating physician has experience managing patients with rheumatoid arthritis.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  <=10 years - Month 2 (n=1300) | 0.20 (0.311)
  <=10 years - Month 4 (n=1300) | 0.23 (0.335)
  <=10 years - Month 6 (n=1300) | 0.25 (0.352)
  >10 to 20 years - Month 2 (n=1103) | 0.18 (0.316)
  >10 to 20 years - Month 4 (n=1103) | 0.22 (0.331)
  >10 to 20 years - Month 6 (n=1103) | 0.24 (0.340)
  >20 years - Month 2 (n=847) | 0.21 (0.309)
  >20 years - Month 4 (n=847) | 0.25 (0.322)
  >20 years - Month 6 (n=847) | 0.26 (0.330)

169. Secondary Outcome: Mean Change From Baseline in EQ-5D by Physician Experience Level With Biologics at Month 2, Month 4, and Month 6
Description: The EQ-5D assesses the 5 domains of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant is asked to indicate their health state by ticking the box against the most appropriate statement in each of the 5 dimensions. The digits (1 [best] to 3 [worst]; with 0= no problems, 1 = some problems, 2 = some problems, and 3= severe problems) for the 5 dimensions can be combined in a 5-digit number describing the participant's health state. The numerals 1 to 3 have no arithmetic properties and should not be used as a cardinal score. Physician experience is defined as the number of years the treating physician has experience managing rheumatoid arthritis with biologics.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Score on a Scale
  0 to 6 years - Month 2 (n=1154) | 0.21 (0.319)
  0 to 6 years - Month 4 (n=1154) | 0.24 (0.347)
  0 to 6 years - Month 6 (n=1154) | 0.26 (0.356)
  6 to 10 years - Month 2 (n=1743) | 0.19 (0.310)
  6 to 10 years - Month 4 (n=1743) | 0.23 (0.324)
  6 to 10 years - Month 6 (n=1743) | 0.24 (0.338)
  >10 years - Month 2 (n=353) | 0.18 (0.300)
  >10 years - Month 4 (n=353) | 0.21 (0.309)
  >10 years - Month 6 (n=353) | 0.24 (0.318)

170. Secondary Outcome: Mean Change From Baseline in EQ-5D by the Number of Patients Treated by the Physician With Biologics at Month 2, Month 4, and Month 6
Description: The EQ-5D assesses the 5 domains of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant is asked to indicate their health state by ticking the box against the most appropriate statement in each of the 5 dimensions. The digits (1 [best] to 3 [worst]; with 0= no problems, 1 = some problems, 2 = some problems, and 3= severe problems) for the 5 dimensions can be combined in a 5-digit number describing the participant's health state. The numerals 1 to 3 have no arithmetic properties and should not be used as a cardinal score. The number of patients treated with biologics is defined as the number of patients with rheumatoid arthritis treated by the physician in the last month with biologic agents.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Units on a Scale
  1-17 patients in prior month - Month 2 (n=1052) | 0.21 (0.307)
  1-17 patients in prior month - Month 4 (n=1052) | 0.24 (0.326)
  1-17 patients in prior month - Month 6 (n=1052) | 0.26 (0.339)
  18-34 patients in prior month - Month 2 (n=1059) | 0.18 (0.312)
  18-34 patients in prior month - Month 4 (n=1059) | 0.21 (0.327)
  18-34 patients in prior month - Month 6 (n=1059) | 0.24 (0.338)
  >=35 patients in prior month - Month 2 (n=1093) | 0.20 (0.319)
  >=35 patients in prior month - Month 4 (n=1093) | 0.24 (0.340)
  >=35 patients in prior month - Month 6 (n=1093) | 0.25 (0.350)

171. Secondary Outcome: Mean Change From Baseline in EQ-5D by the the Physician Expectation of Treatment Outcome at Month 2, Month 4, and Month 6
Description: The EQ-5D assesses the 5 domains of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant indicates their health state by ticking the box against the most appropriate statement. The digits (1 [best] to 3 [worst]; with 0= no problems, 1 = some problems, 2 = some problems, and 3= severe problems) for the 5 dimensions can be combined in a 5-digit number describing the participant's health state. The numerals 1 to 3 have no arithmetic properties and should not be used as a cardinal score. The physician's expectation of treatment outcome was assessed at the start of Month 4, when physicians were asked to rate their expectations of treatment outcome as: high disease activity, moderate disease activity, low disease activity, or remission.
Time Frame: Baseline, Month 2, Month 4, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Units on a Scale
  High disease activity - Month 2 (n=38) | 0.24 (0.315)
  High disease activity - Month 4 (n=38) | 0.20 (0.355)
  High disease activity - Month 6 (n=38) | 0.20 (0.352)
  Moderate disease activity - Month 2 (n=325) | 0.18 (0.298)
  Moderate disease activity - Month 4 (n=325) | 0.23 (0.320)
  Moderate disease activity - Month 6 (n=325) | 0.25 (0.320)
  Low disease activity - Month 2 (n=1926) | 0.20 (0.323)
  Low disease activity - Month 4 (n=1926) | 0.23 (0.335)
  Low disease activity - Month 6 (n=1926) | 0.25 (0.349)
  Remission - Month 2 (n=964) | 0.19 (0.295)
  Remission - Month 4 (n=964) | 0.22 (0.323)
  Remission - Month 6 (n=964) | 0.23 (0.335)

172. Secondary Outcome: Number of Participants With a Participant Acceptable Symptom State (PASS) at Month 4, Month 6, and Month 8
Description: The number of participants achieving PASS was evaluated at study Month 2, Month 4, and Month 6 was calculated. PASS is participant self-evaluation tool that uses a VAS 0mm (best) - 100mm (worst), with a score <=31 representing an acceptable PASS.
Time Frame: Month 2, Month 4, Month 6
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | GLM50-SC
Number analyzed (Participants) | 3280
Participants
  Study Month 2 | 1578
  Study Month 4 | 1889
  Study Month 6 | 2164

173. Secondary Outcome: Mean Area Under the DAS28-ESR Curve From Study Month 6 to Month 12
Description: The DAS28-ESR is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, ESR, and participant assessment of disease activity measure on a visual analogue scale. The DAS28-ESR has numeric thresholds that define high disease activity (> 5.1), low disease activity (< 3.2) and remission (< 2.6). Minimum score=0 (best) to maximum score=10 (worst). The DAS28-ESR area under the curve can be calculated from the DAS28-ESR score versus time curve to provide an assessment of changes in disease activity over time.
  The area under the DAS28-ESR score versus time curve was computed using the trapezoidal rule and using raw DAS28-ESR score values at Part-2 Baseline, end of Month 12, and at least 2 intermediate time points. The DAS28-ESR area under the curve was then averaged over the total duration (months) and expressed as units on a scale.
Time Frame: End of Month 6, End of Month 12
Population: 8 participants (3 poor quality data, 4 without a post-baseline DAS28-ESR, and 1 did not take Part 2 medication) and 7 participants (5 poor data quality, 1 without a DAS28-ESR at baseline, 1 without post-baseline DAS28-ESR) were excluded from the efficacy evaluable population for the IV-GLM 2mg/kg + SC GLM 50 mg and SC-GLM50 arms, respectively.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- IV-GLM 2 mg/kg + SC GLM 50 mg: Participants received IV-GLM at a dose of 2 mg/kg at the start of Month 7, start of Month 8, and start of Month 10 if remission was not achieved at any of these IV administration visits. If remission was achieved, participants were switched to subcutaneous golimumab
  at a dose of 50 mg once monthly.
- SC-GLM50: Participants received SC GLM at a dose of 50 mg once monthly.
Arm/Group | IV-GLM 2 mg/kg + SC GLM 50 mg | SC-GLM50
Number analyzed (Participants) | 242 | 248
Units on a Scale | 3.67 (0.992) | 3.67 (0.924)

174. Secondary Outcome: Percentage of Participants Achieving Remission
Description: Remission was defined as achievement of a DAS28-ESR < 2.6.
Time Frame: Start of Month 8, Start of Month 9, Start of Month 10, Start of Month 11, End of Month 12
Population: as for outcome 173
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- IV-GLM 2 mg/kg + SC GLM 50 mg: Participants received IV GLM at a dose of 2 mg/kg until remission is achieved at which time they were switched to SC GLM at a dose of 50 mg once monthly.
Arm/Group | IV-GLM 2 mg/kg + SC GLM 50 mg | SC-GLM50
Number analyzed (Participants) | 242 | 248
Percentage of Participants
  Start of Month 8 | 19.8 [15.3 to 25.4] | 13.7 [10.0 to 18.7]
  Start of Month 9 | 28.2 [23.0 to 34.4] | 20.1 [15.7 to 25.]
  Start of Month 10 | 34.2 [28.6 to 40.6] | 29.5 [24. to 35.6]
  Start of Month 11 | 40.3 [34.3 to 46.8] | 39.3 [33.5 to 45.7]
  End of Month 12 | 44.3 [38.2 to 50.9] | 45.1 [39.1 to 51.5]

ADVERSE EVENTS:
Groups:
- Golimumab 50 mg Subcutaneous (GLM50-SC): Participants received GLM50-SC once monthly for a period of 6 months.
- Intravenous GLM (IV-GLM) 2 mg/kg + SC GLM 50 mg: Participants received IV-GLM at a dose of 2 mg/kg at the start of Month 7, start of Month 8, and start of Month 10 if remission was not achieved at any of these IV administration visits. If remission was achieved, participants were switched subcutaneous golimumab
  at a dose of 50 mg once monthly.
- SC-GLM50: Participants received subcutaneous golimumab at a dose of 50 mg once monthly for a period of 6 months in Part 2 of the study.
Arm/Group | Golimumab 50 mg Subcutaneous (GLM50-SC) | Intravenous GLM (IV-GLM) 2 mg/kg + SC GLM 50 mg | SC-GLM50
Serious Adverse Events (participants affected / at risk) | 203/3357 | 17/245 | 7/255
Other Adverse Events (participants affected / at risk) | 0/3357 | 28/245 | 24/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Golimumab 50 mg Subcutaneous (GLM50-SC) (N=3357) | Intravenous GLM (IV-GLM) 2 mg/kg + SC GLM 50 mg (N=245) | SC-GLM50 (N=255)
Pneumonia (Infections and infestations) | 9 (10) | 2 (2) | 1 (1)
Arthritis bacterial (Infections and infestations) | 5 (5) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 5 (5) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 4 (5) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Peritonsillar abcess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Rotavirus infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Abcess oral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Groin abcess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Herpes zoster oticus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Listeria sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ludwig angina (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lymph node tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Syphillis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 9 (9) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar spine stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Polychondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 5 (5) | 2 (2) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Ankle fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Diffuse large B-cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Appendix disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis atrophic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal varicies hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestine obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibriliation (Cardiac disorders) | 3 (4) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0) | 0 (0)
Calcinosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiases (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal amyloidosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arterial bypass operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Arthrodesis (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Lymphadenectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 3 (3) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Endometrial hypertrophy (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Open angle glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Conductive deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Golimumab 50 mg Subcutaneous (GLM50-SC) (N=3357) | Intravenous GLM (IV-GLM) 2 mg/kg + SC GLM 50 mg (N=245) | SC-GLM50 (N=255)
Nasopharyngitis (Infections and infestations) | 0 (0) | 13 (15) | 18 (19)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 15 (17) | 6 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator is granted the right to use the results of all work under this study including but not limited to, the results of tests and any raw data and statistical data generated for investigator's own teaching, research, and publication purposes only. Investigator/Institution agrees, on behalf of itself and its employees, officers, trustees, and agents, not to cause said results to be knowingly used for any commercial purpose whatsoever except as authorized by the sponsor in writing.